CLINICAL TRIAL: NCT00048568
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study and Open-Label Study to Evaluate the Efficacy and Safety of Abatacept in Combination Therapy With Methotrexate Versus Methotrexate Alone in Subjects With Active Rheumatoid Arthritis and Inadequate Response to Methotrexate
Brief Title: A Phase III Study of Abatacept (BMS-188667) in Patients With Active Rheumatoid Arthritis and Inadequate Response to Methotrexate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-102
Record Dates: First submitted 2002-11-02; First posted 2002-11-13 (Estimated); Results first posted 2011-12-05 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Abatacept + Methotrexate (Experimental): Short Term: Abatacept was dosed by weight with participants weighing < 60 kg received abatacept 500 mg; participants ≥ 60 kg and ≤ 100 kg received abatacept 750 mg; and participants > 100 kg received abatacept 1 g. Participants continued treatment with methotrexate (MTX) either orally or parenterally at a minimum dose of 15 mg.
  Interventions: Drug: Abatacept; Drug: Methotrexate
- Placebo + Methotrexate (Active Comparator): Short Term: Participants received a placebo solution intravenously and methotrexate at the dose employed prior to study enrollment and a minimum of 15 mg.
  Interventions: Drug: Methotrexate; Drug: Placebo
- Abatacept + Methotrexate Open Label (Experimental): Open Label: Abatacept was dosed intravenously by weight at 10 mg/kg in the OL period under tiered dosing such that participants weighing < 60 kg received abatacept 500 mg; participants ≥ 60 kg and ≤ 100 kg received abatacept 750 mg; and participants > 100 kg received abatacept 1 g. MTX was continued at the dose used in the DB period.
  Interventions: Drug: Abatacept; Drug: Methotrexate

INTERVENTIONS:
Drug: Abatacept — Intravenous (IV) Solution, - Weight Titered (500 mg < 60 kg); (750 mg 60-100 kg), )1 gram > 100 kg), Day 1, Day 15, Day 29; every 28 days thereafter, 1 year
  Other Names: BMS-188667
  Arms: Abatacept + Methotrexate; Abatacept + Methotrexate Open Label
Drug: Methotrexate — Tablets, Oral, >= 15 mg, weekly, 1 year
  Other Names: MTX
Drug: Placebo — IV solution, Intravenous, D5W, Day 1, Day 15, Day 29; every 28 days thereafter, 1 year
  Arms: Placebo + Methotrexate

SUMMARY:
Short Term: The purpose of this clinical research study is to learn if abatacept (BMS-188667) in combination with methotrexate is better than methotrexate alone in participants that have active rheumatoid arthritis and are not responding to methotrexate. The safety of this treatment will also be studied.

Long Term Extension: The purpose of this amendment is to provide participants who have completed the initial 12-month double-blind treatment period the opportunity to receive open label treatment with active drug treatment until abatacept is approved in the local country or until clinical development has been discontinued.

ELIGIBILITY:
* Rheumatoid Arthritis (RA) for greater than 1 year from the time of initial diagnosis of RA.
* Participants must have been taking methotrexate for at least 3 months with at least a weekly dose of 15 mg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250 (Actual)
Dates: Start 2002-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (48):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Huntsville, Alabama
  - Local Institution, Mobile, Alabama
  - Local Institution, Phoenix, Arizona
  - Local Institution, Scottsdale, Arizona
  - Local Institution, Corona, California
  - Local Institution, Irvine, California
  - Local Institution, La Jolla, California
  - Local Institution, Long Beach, California
  - Local Institution, Rancho Mirage, California
  - Local Institution, Aurora, Colorado
  - Local Institution, Colorado Springs, Colorado
  - Local Institution, Denver, Colorado
  - Local Institution, Hamden, Connecticut
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Gainsville, Florida
  - Local Institution, Palm Harbor, Florida
  - Local Institution, Sarasota, Florida
  - Local Institution, St. Petersburg, Florida
  - Local Institution, Chicago, Illinois
  - Local Institution, Rockford, Illinois
  - Local Institution, Wichita, Kansas
  - Local Institution, Coeur d'Alene, Maryland
  - Local Institution, Cumberland, Maryland
  - Local Institution, Springfield, Massachusetts
  - Local Institution, Duluth, Minnesota
  - Local Institution, Lincoln, Nebraska
  - Local Institution, New Brunswick, New Jersey
  - Local Institution, Albuquerque, New Mexico
  - Local Institution, Albany, New York
  - Local Institution, Binghamton, New York
  - Local Institution, Mineola, New York
  - Local Institution, New York, New York
  - Local Institution, Syracuse, New York
  - Local Institution, The Bronx, New York
  - Local Institution, Wilmington, North Carolina
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Duncansville, Pennsylvania
  - Local Institution, Norristown, Pennsylvania
  - Local Institution, Sellersville, Pennsylvania
  - Local Institution, Willow Grove, Pennsylvania
  - Local Institution, North Charleston, South Carolina
  - Local Institution, Austin, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Arlington, Virginia
  - Local Institution, Milwaukee, Wisconsin

REFERENCES:
- [Result] Kremer JM, Genant HK, Moreland LW, Russell AS, Emery P, Abud-Mendoza C, Szechinski J, Li T, Ge Z, Becker JC, Westhovens R. Effects of abatacept in patients with methotrexate-resistant active rheumatoid arthritis: a randomized trial. Ann Intern Med. 2006 Jun 20;144(12):865-76. doi: 10.7326/0003-4819-144-12-200606200-00003. PMID 16785475
- [Derived] Kremer JM, Peterfy C, Russell AS, Emery P, Abud-Mendoza C, Sibilia J, Becker JC, Westhovens R, Genant HK. Longterm safety, efficacy, and inhibition of structural damage progression over 5 years of treatment with abatacept in patients with rheumatoid arthritis in the abatacept in inadequate responders to methotrexate trial. J Rheumatol. 2014 Jun;41(6):1077-87. doi: 10.3899/jrheum.130263. Epub 2014 May 1. PMID 24786925
- [Derived] Kremer JM, Genant HK, Moreland LW, Russell AS, Emery P, Abud-Mendoza C, Szechinski J, Li T, Teng J, Becker JC, Westhovens R. Results of a two-year followup study of patients with rheumatoid arthritis who received a combination of abatacept and methotrexate. Arthritis Rheum. 2008 Apr;58(4):953-63. doi: 10.1002/art.23397. PMID 18383390

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in this evaluation were enrolled 116 sites worldwide: 31 sites in the United States; 32 sites in Europe, 13 sites in Canada; 4 sites in Australia; 7 sites in Argentina; 7 sites in Brazil; 7 sites in Mexico; 3 sites in Peru; 5 sites in South Africa; 3 sites in Taiwan; and 4 sites in Turkey.
Pre-assignment Details: Of 1250 participants enrolled, 594 participants were not randomized (519 no longer met study criteria, 37 for unknown reasons, 33 withdrew consent, 3 lost to follow-up, 1 administrative reason by sponsor, and 1 adverse event). Four participants (2 per group) were randomized but never treated; 2 no longer met study criteria and 2 withdrew consent.
Groups:
- Abatacept (ABA) + Methotrexate (MTX) DB: Abatacept was dosed intravenously by weight with participants weighing < 60 kg received 500 mg, participants weighing 60 kg to 100 kg received 750 mg, and participants weighing > 100 kg received 1 gram. Study medication was administered on Days 1, 15, 29, and every 28 days thereafter for a total of 14 doses. Each dose was infused intravenously over approximately 30 minutes on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337. Participants also received MTX at a minimum dose of (10-30 mg/wk), although doses of < 10 mg/wk were acceptable if due to toxicity.
- MTX + Placebo DB: Control group receiving MTX treatment in combination with placebo. Participants received MTX at a minimum dose of (10-30 mg/wk), although doses of < 10 mg/wk were acceptable if due to toxicity. Placebo was administered IV on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337.
- ABA + MTX [Open-label (OL)]: Abatacept was dosed intravenously by weight at 10 mg/kg in the OL period under tiered dosing such that participants weighing < 60 kg received abatacept 500 mg; participants ≥ 60 kg and ≤ 100 kg received abatacept 750 mg; and participants > 100 kg received abatacept 1 g. MTX was continued at the dose used in the DB period.
Period: Double-Blind Period Days 1 to 169
Arm/Group | Abatacept (ABA) + Methotrexate (MTX) DB | MTX + Placebo DB | ABA + MTX [Open-label (OL)]
Started | 433 | 219 | 0
Completed | 401 | 174 | 0
Not Completed | 32 | 45 | 0
Not completed — Adverse Event | 11 | 3 | 0
Not completed — Lack of Efficacy | 11 | 33 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 4 | 0
Not completed — Unknown Reasons | 2 | 4 | 0
Period: Double-Blind Period Days 170 to 365
Arm/Group | Abatacept (ABA) + Methotrexate (MTX) DB | MTX + Placebo DB | ABA + MTX [Open-label (OL)]
Started | 401 | 174 | 0
Completed | 385 | 162 | 0
Not Completed | 16 | 12 | 0
Not completed — Death | 1 | 1 | 0
Not completed — Adverse Event | 7 | 1 | 0
Not completed — Lack of Efficacy | 2 | 7 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0
Not completed — Poor/Non-Compliance | 0 | 1 | 0
Not completed — Pregnancy | 2 | 0 | 0
Not completed — No Longer Met Study Criteria | 1 | 1 | 0
Period: Open-Label Period
Arm/Group | Abatacept (ABA) + Methotrexate (MTX) DB | MTX + Placebo DB | ABA + MTX [Open-label (OL)]
Started | 0 | 0 | 539
Completed | 0 | 0 | 379
Not Completed | 0 | 0 | 160
Not completed — Death | 0 | 0 | 13
Not completed — Adverse Event | 0 | 0 | 49
Not completed — Lack of Efficacy | 0 | 0 | 32
Not completed — Withdrawal by Subject | 0 | 0 | 26
Not completed — Pregnancy | 0 | 0 | 5
Not completed — No Longer Met Study Criteria | 0 | 0 | 2
Not completed — Administrative Decision By Sponsor | 0 | 0 | 1
Not completed — Unknown Reasons | 0 | 0 | 25
Not completed — Lost to Follow-up | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- ABA + MTX DB: Abatacept was dosed by weight with participants weighing < 60 kg received 500 mg, participants weighing 60 kg to 100 kg received 750 mg, and participants weighing > 100 kg received 1 gram. Study medication was administered on Days 1, 15, 29, and every 28 days thereafter for a total of 14 doses. Each dose was infused intravenously over approximately 30 minutes on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337. Participants also received MTX at a minimum dose of (10-30 mg/wk), although doses of < 10 mg/wk were acceptable if due to toxicity. Placebo and MTX were administered IV on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337.
- Total: Total of all reporting groups
Arm/Group | ABA + MTX DB | MTX + Placebo DB | Total
Number analyzed (Participants) | 433 | 219 | 652
Age Continuous [Mean (Standard Deviation); unit: years] | 51.5 (12.9) | 50.4 (12.4) | 51.1 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 40 | 136
  Male | 337 | 179 | 516
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 18 | 10 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 4 | 14
  White | 379 | 193 | 572
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 23 | 11 | 34
Duration of Rheumatoid Arthritis (RA) Disease [Number; unit: Participants] — Number of participants with RA duration <= 2 years, > 2 years to <= 5 years, > 5 years to <= 10 years, and > 10 years as evaluated at baseline.
  Participants
    <= 2 years | 99 | 45 | 144
    > 2 years to <= 5 years | 93 | 46 | 139
    > 5 years to <=10 years | 106 | 54 | 160
    > 10 years | 135 | 74 | 209

OUTCOME MEASURES:

1. Primary Outcome: Number of American College of Rheumatology 20 (ACR 20) Responders at Day 169
Description: ACR 20 response requires a patient to have a 20% reduction in the number of swollen and tender joints, and a reduction of 20% in three of the following five parameters: physician global assessment of disease, patient global assessment of disease, patient assessment of pain, C-reactive protein or erythrocyte sedimentation rate, and degree of disability in Health Assessment Questionnaire (HAQ) score. A participant achieved a sustained ACR 20 response if the participant had ACR 20 observed for at least 2 consecutive study visits.
Time Frame: Day 169
Population: Analyses of efficacy were based on the intent-to-treat population. Due to the non-compliance of a single site, 9 participants in the abatacept group and 5 in the placebo group were not included in this analysis.
Measure: Number; unit: Participants
Groups:
- ABA + MTX DB: Abatacept was dosed intravenously by weight with participants weighing < 60 kg received 500 mg, participants weighing 60 kg to 100 kg received 750 mg, and participants weighing > 100 kg received 1 gram. Study medication was administered on Days 1, 15, 29, and every 28 days thereafter for a total of 14 doses. Each dose was infused intravenously over approximately 30 minutes on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337. Participants also received MTX at a minimum dose of 10-30 mg/wk, although doses of < 10 mg/wk were acceptable if due to toxicity.
- MTX + Placebo DB: Control group receiving MTX treatment in combination with placebo. Participants received MTX at a minimum dose of 10-30 mg/wk, although doses of < 10 mg/wk were acceptable if due to toxicity. Placebo and MTX were administered IV on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337.
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Participants | 288 | 85
Statistical Analysis 1: Comparison: ABA + MTX DB vs MTX + Placebo DB; The study had a 99% power to detect a difference of 20% in ACR 20 between the 2 groups at the 5% level; Test type: Superiority or Other; p < 0.001, Chi-squared, Corrected; Estimated Difference = 28.2, 95% CI 2-sided [19.8 to 36.7] — Estimated difference between ABA + MTX and MTX + PLA is the estimated difference between ABA+MTX and MTX + PLA in the proportion of participants achieving ACR 20 response

2. Primary Outcome: Number of Participants Achieving Clinically Meaningful Improvement in Health Assessment Questionnaire (HAQ) at Day 365
Description: The HAQ-DI includes 20 questions to assess physical function in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip, and common activities. The domain questions are evaluated on a 4-point scale: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=unable to do. HAQ-DI=sum of worst scores in each domain dividied by the number of domains answered. HAQ-DI ranges from 0 to a maximum overall score of 3.0. Clinically meaningful HAQ response was defined as an improvement of at least 0.3 units from baseline in HAQ DI.
Time Frame: Day 365
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Participants | 270 | 84
Statistical Analysis 1: Comparison: ABA + MTX DB vs MTX + Placebo DB; Test type: Superiority or Other; p < 0.001, Chi-squared, Corrected — Based on the hierarchical testing procedure for the co-primary measures, the study had 98% power to detect 18% difference in HAQ response rate between the two arms at the 5% level; This model includes treatment as the main factor and baseline value as a covariate; Estimated Difference = 24.4, 95% CI 2-sided [15.9 to 32.9] — Estimated difference between ABA + MTX and MTX + PLA is the estimated difference between ABA+MTX and MTX + PLA in the proportion of participants achieving HAQ response at Day 365

3. Primary Outcome: Baseline and Mean Change From Baseline (BL) in Radiographic Erosion Score Results at Day 365
Description: To assess joint damage progression, the Genant-modified Sharp scoring method was used to evaluate radiographs of hands/wrists and feet for erosions. The erosion score range is 0 (no radiographic damage) to 145 (worst possible radiographic damage). Change from baseline = Post-baseline - Baseline value
Time Frame: BL (Day 0), Day 365
Population: All randomized and treated participants in the DB period with radiographic data available at baseline and Day 365. Due to the compliance issues of a single site, 9 participants in the abatacept group and 5 in the placebo group were not included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 391 | 195
Units on a Scale
  BL | 21.68 (18.07) | 21.83 (18.63)
  Mean Change From BL | 0.63 (1.77) [0.00 to 1.02] | 1.14 (2.81) [0.00 to 1.27]
Statistical Analysis 1: Comparison: ABA + MTX DB vs MTX + Placebo DB; Test type: Superiority or Other; p = 0.029, Nonparametric ANCOVA; The rank of the change from baseline=dependent variable, treatment=the main factor, rank of baseline value as covariate

4. Secondary Outcome: Mean Number of Tender Joints and Swollen Joints at DB BL
Time Frame: BL (Day 0)
Population: All randomized and treated participants in the DB period.
Measure: Mean (Standard Deviation); unit: Joints
Groups:
- ABA + MTX DB: Abatacept was dosed by weight with participants weighing < 60 kg received 500 mg, subjects weighing 60 kg to 100 kg received 750 mg, and subjects weighing > 100 kg received 1 gram. Study medication was administered on Days 1, 15, 29, and every 28 days thereafter for a total of 14 doses. Each dose was infused intravenously over approximately 30 minutes on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337. Participants also received MTX at a minimum dose of (10-30 mg/wk), although doses of < 10 mg/wk were acceptable if due to toxicity.
- MTX + Placebo DB: Control group receiving MTX treatment in combination with placebo. Participants received MTX at a minimum dose of (10-30 mg/wk), although doses of < 10 mg/wk were acceptable if due to toxicity. Placebo and MTX were administered IV on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337.
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 433 | 219
Joints
  Tender Joints | 31.0 (13.2) | 32.3 (13.6)
  Swollen Joints | 21.4 (8.8) | 22.1 (8.8)

5. Secondary Outcome: Mean DB BL Participant Physical Pain Assessment, Participant Global Assessment, and Physician Global Assessment
Description: Participant physical pain assessment was determined at baseline on the Visual Analog Scale (VAS) of 0 mm to 100 mm where 0mm is no pain and 100mm is worst pain possible. The mean participant global assessment is a measure of overall disease burden and is a component of the ACR and evaluated using the VAS 100 mm. The physician global assessment is a measure of overall disease burden and is a component of the ACR and evaluated using the VAS 0mm to 100 mm with 0mm indicating no disease burden and 100mm indicating worse disease burden possible.
Time Frame: BL (Day 0)
Population: All randomized and treated participants in the DB period.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 433 | 219
Units on a Scale
  Participant Physical Pain Assessment | 63.3 (21.1) | 65.9 (20.6)
  Participant Global Assessment | 62.7 (21.2) | 62.8 (21.6)
  Physician Global Assessment | 68.0 (16.0) | 67.4 (17.0)

6. Secondary Outcome: BL Rheumatoid Factor (RF) Status for Participants Continuing in the OL Period
Description: This analysis determined whether participants in the OL period were RF positive or RF negative based on serum samples. A positive value for RF was > 20 IU/ml; a negative value for RF was ≤ 20 IU/mL.
Time Frame: BL (Day 365)
Population: All treated participants in the OL period (treatment groups represent treatment received in the DB period).
Measure: Number; unit: Participants
Groups:
- ABA + MTX DB: Abatacept was dosed intravenously by weight at 10 mg/kg in the OL period under tiered dosing such that participants weighing < 60 kg received abatacept 500 mg; participants ≥ 60 kg and ≤ 100 kg received abatacept 750 mg; and participants > 100 kg received abatacept 1 g. MTX was continued at the dose used in the DB period.
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 378 | 161
Participants
  RF Negative | 42 | 18
  RF Positive | 312 | 130

7. Secondary Outcome: ACR 20 Responders at Day 365
Description: ACR 20 response requires a patient to have a 20% reduction in the number of swollen and tender joints, and a reduction of 20% in three of the following five parameters: physician global assessment of disease, patient global assessment of disease, patient assessment of pain, C-reactive protein or erythrocyte sedimentation rate, and degree of disability in HAQ score. A participant achieved a sustained ACR 20 response if the participant had ACR 20 observed for at least 2 consecutive study visits.
Time Frame: Day 365
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Participants | 310 | 85
Statistical Analysis 1: Comparison: ABA + MTX DB vs MTX + Placebo DB; Test type: Superiority or Other; p < 0.001, Chi-squared, Corrected; Estimated Difference = 33.4, 95% CI 2-sided [25.1 to 41.7] — Estimated difference between ABA + MTX and MTX + PLA is the estimated difference between ABA+MTX and MTX + PLA in the proportion of participants achieving ACR 20 response at Day 365

8. Secondary Outcome: ACR 20 Responders in the Double-Blind (DB) Period
Description: ACR 20 response requires a patient to have a 20% reduction in the number of swollen and tender joints, and a reduction of 20% in three of the following five parameters: physician global assessment of disease, patient global assessment of disease, patient assessment of pain, C-reactive protein or erythrocyte sedimentation rate, and degree of disability in HAQ score.
Time Frame: Day 15, Day 29, Day 57, Day 85, Day 113, Day 141, Day 169, Day 225, Day 281, Day 365
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Participants
  Day 15 | 97 | 30
  Day 29 | 155 | 51
  Day 57 | 237 | 75
  Day 85 | 262 | 80
  Day 113 | 283 | 86
  Day 141 | 291 | 93
  Day 169 | 288 | 85
  Day 225 | 318 | 91
  Day 281 | 312 | 94
  Day 365 | 310 | 85

9. Secondary Outcome: ACR 50 Responders at Day 169
Description: ACR 50 response requires a patient to have a 50% reduction in the number of swollen and tender joints, and a reduction of 50% in three of the following five parameters: physician global assessment of disease, patient global assessment of disease, patient assessment of pain, C-reactive protein or erythrocyte sedimentation rate, and degree of disability in HAQ score. A participant achieved a sustained ACR 50 response if the participant had ACR 50 observed for at least 2 consecutive study visits.
Time Frame: Day 169
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Participants | 169 | 36
Statistical Analysis 1: Comparison: ABA + MTX DB vs MTX + Placebo DB; Test type: Superiority or Other; p < 0.001, Chi-squared, Corrected; Estimated Difference = 23.0, 95% CI 2-sided [15.0 to 31.1] — Estimated difference between ABA + MTX and MTX + PLA is the estimated difference between ABA+MTX and MTX + PLA in the proportion of participants achieving ACR 50 response at Day 169

10. Secondary Outcome: ACR 50 Responders at Day 365
Description: ACR 50 response requires a patient to have a 50% reduction in the number of swollen and tender joints, and a reduction of 50% in three of the following five parameters: physician global assessment of disease, patient global assessment of disease, patient assessment of pain, C-reactive protein or erythrocyte sedimentation rate, and degree of disability in HAQ score.
Time Frame: Day 365
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Participants | 205 | 39
Statistical Analysis 1: Comparison: ABA + MTX DB vs MTX + Placebo DB; Test type: Superiority or Other; p < 0.001, Chi-squared, Corrected; Estimated Difference = 30.1, 95% CI 2-sided [21.8 to 38.5] — Estimated difference between ABA + MTX and MTX + PLA is the estimated difference between ABA+MTX and MTX + PLA in the proportion of participants achieving ACR 50 response at Day 365

11. Secondary Outcome: ACR 50 Responders in the DB Period
Description: as for outcome 9
Time Frame: Day 15, Day 29, Day 57, Day 85, Day 113, Day 141, Day 169, Day 225, Day 281, Day 365
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Participants
  Day 15 | 12 | 2
  Day 29 | 36 | 9
  Day 57 | 87 | 16
  Day 85 | 135 | 17
  Day 113 | 148 | 27
  Day 141 | 162 | 39
  Day 169 | 169 | 36
  Day 225 | 197 | 42
  Day 281 | 200 | 38
  Day 365 | 205 | 39

12. Secondary Outcome: ACR 70 Responders at Day 169
Description: ACR 70 response requires a patient to have a 70% reduction in the number of swollen and tender joints, and a reduction of 70% in three of the following five parameters: physician global assessment of disease, patient global assessment of disease, patient assessment of pain, C-reactive protein or erythrocyte sedimentation rate, and degree of disability in HAQ score.
Time Frame: Day 169
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Participants | 84 | 14
Statistical Analysis 1: Comparison: ABA + MTX DB vs MTX + Placebo DB; Test type: Superiority or Other; p < 0.001, Chi-squared, Corrected; Estimated Difference = 13.3, 95% CI 2-sided [7.0 to 19.5] — Estimated difference between ABA + MTX and MTX + PLA is the estimated difference between ABA + MTX and MTX + PLA in the proportion of participants achieving ACR 70 response at Day 169

13. Secondary Outcome: ACR 70 Responders at Day 365
Description: as for outcome 12
Time Frame: Day 365
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Participants | 122 | 13
Statistical Analysis 1: Comparison: ABA + MTX DB vs MTX + Placebo DB; Test type: Superiority or Other; p < 0.001, Chi-squared, Corrected; Mean Difference (Final Values) = 22.7, 95% CI 2-sided [15.6 to 29.8]

14. Secondary Outcome: ACR 70 Responders in the DB Period
Description: as for outcome 12
Time Frame: Day 15, Day 29, Day 57, Day 85, Day 113, Day 141, Day 169, Day 225, Day 281, Day 365
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Participants
  Day 15 | 4 | 1
  Day 29 | 8 | 2
  Day 57 | 27 | 6
  Day 85 | 54 | 7
  Day 113 | 57 | 12
  Day 141 | 75 | 12
  Day 169 | 84 | 14
  Day 225 | 103 | 16
  Day 281 | 106 | 19
  Day 365 | 122 | 13

15. Secondary Outcome: Number of Participants Achieving Major Clinical Response By Day 365
Description: A Major Clinical Response (MCR) is defined as maintenance of an ACR 70 response over a continuous 6-month period.
Time Frame: Day 1 to Day 365. Data were collected monthly during the first 6 months and then every other month (with the exception of Day 337) during the second 6 months of the DB period.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Participants | 60 | 4
Statistical Analysis 1: Comparison: ABA + MTX DB vs MTX + Placebo DB; Test type: Superiority or Other; p < 0.001, Chi-squared, Corrected; Estimated Difference = 12.3, 95% CI 2-sided [7.3 to 17.2] — Estimated difference between ABA + MTX and MTX + PLA is the estimated difference between ABA+MTX and MTX + PLA in the proportion of participants achieving MCR

16. Secondary Outcome: Mean BL and Disease Activity Score 28 (DAS-28; Erythrocyte Sedimentation Rate [ESR]) at Day 169 and Day 365
Description: The DAS 28 is an assessment of disease activity measured on a visual analog scale (VAS)of 100 mm. The scale reports from 1 to 10, with increasing number indicating increasing extent of disease progression. Scores for disease activity are defined as high (>5.1); low (≤3.2); remission (<2.6). Time-matched BL(Day 0) values and post-BL vales were presented for each post-BL visit and represent only that cohort of participants with measurements available at that post-BL assessment.
Time Frame: BL (Day 0), Day 169, Day 365, Day 169, Day 365
Population: Analyses of efficacy were based on the intent-to-treat population. Due to the non-compliance of a single site, 9 participants in the abatacept group and 5 in the placebo group were not included in this analysis. Last Observation Carried Forward (LOCF) analysis. N = participants analyzed and n = participants with measurements for that time point.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Units on a Scale
  BL (Day 0) for Day 169 Cohort (n=366, 179) | 6.82 (0.87) | 6.84 (0.82)
  BL (Day 0) for Day 169 Cohort (n=366, 179) | 4.34 (1.38) | 5.50 (1.35)
  BL (Day 0) for Day 365 Cohort (n=375, 183) | 6.82 (0.87) | 6.83 (0.82)
  BL (Day 0) for Day 365 Cohort (n=375, 183) | 3.97 (1.40) | 5.36 (1.32)
Statistical Analysis 1: Comparison: ABA + MTX DB vs MTX + Placebo DB; Test type: Superiority or Other; p < 0.001, ANCOVA; Estimated Difference on Day 169 = -1.15, 95% CI 2-sided [-1.38 to -0.91] — Estimated difference between ABA + MTX and MTX + PLA on Day 169
Statistical Analysis 2: Comparison: ABA + MTX DB vs MTX + Placebo DB; Test type: Superiority or Other; p < 0.001, ANCOVA; Estimated Difference on Day 365 = -1.39, 95% CI 2-sided [-1.63 to -1.16] — Estimated difference between ABA + MTX and MTX + PLA on Day 365

17. Secondary Outcome: Number of Participants With Death, Serious Adverse Events (SAEs), Related SAEs, Discontinuation Due to SAEs, AEs, Related AEs, or Discontinued Due to AEs in the DB Period
Description: AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. SAE was defined as any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event.
Time Frame: Day 1 to Day 365
Population: All treated subjects in the DB period.
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 433 | 219
Participants
  Deaths | 1 | 1
  SAEs | 65 | 26
  Related SAEs | 15 | 1
  Discontinuations Due to SAEs | 10 | 3
  AEs | 378 | 184
  Related AEs | 214 | 104
  Discontinued Due to AEs | 18 | 4

18. Secondary Outcome: Mean DB BL and Mean Change From BL in Joint Space Narrowing (JSN) and Total Score (TS)
Description: To assess joint damage progression, the Genant-modified Sharp scoring method was used to evaluate radiographs of hands/wrists and feet for erosions and joint space narrowing (JSN). The total Genant-modified Sharp score ranges from 0 (no radiographic damage) to 290 (worst possible radiographic damage) and is the sum of the erosion score (range 0-145) and the joint space narrowing score (range 0-145). Higher scores indicated more damage. Change from baseline = Post-baseline - Baseline value.
Time Frame: BL (Day 0), Day 365
Population: All randomized and treated participants in the DB period with radiographic data available at baseline and Day 365. Due to the non-compliance of a single site, 9 participants in the abatacept group and 5 in the placebo group were not included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 391 | 195
Units on a Scale
  Baseline Mean JSN | 22.79 (20.16) | 23.02 (20.36)
  Mean Change From Baseline JSN Day 365 | 0.58 (1.54) | 1.18 (2.58)
  Baseline Mean TS | 44.47 (37.33) | 44.85 (37.72)
  Mean Change From Baseline TS Day 365 | 1.21 (2.94) | 2.32 (5.04)

19. Secondary Outcome: Mean DB BL Physical Component Summary of Health-Related Quality of Life (SF-36)
Description: The SF-36 covers 8 health dimensions including 4 physical subscales (physical function, role-physical, bodily pain, and general health) and 4 mental subscales (vitality, social function, role-emotional, and mental health). The scores range from a minimum of 0 to a maximum of 100, with a higher score indicating better quality of life. Improvements of > 3 points were considered clinically meaningful. Time-matched BL(Day 0) values and post-BL vales were presented for each post-BL visit and represent only that cohort of participants with measurements available at that post-BL assessment.
Time Frame: BL (Day 0), Day 169, Day 365
Population: Analyses of efficacy were based on the intent-to-treat population.Due to the non-compliance of a single site, 9 participants in the abatacept group and 5 in the placebo group were not included in this analysis. Last Observation Carried Forward (LOCF) analysis. N = participants analyzed and n = participants with measurements for that time point.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Units on a Scale
  BL (Day 0) for Day 169 Cohort (n= 416, 207) | 30.49 (7.18) | 30.61 (7.42)
  BL (Day 0) for Day 365 Cohort (n=417, 207) | 30.51 (7.17) | 30.62 (7.42)

20. Secondary Outcome: Adjusted Mean Change From BL in the Physical Component Summary of Health-Related Quality of Life (SF-36) in the DB Period
Description: The SF-36 covers 8 health dimensions including 4 physical subscales (physical function, role-physical, bodily pain, and general health) and 4 mental subscales (vitality, social function, role-emotional, and mental health). All subscales were scored using norm-based methods that standardized the scores to a mean of 50 and a standard deviation of 10 in the general population. The scores range from a minimum of 0 to a maximum of 100, with a higher score indicating better quality of life. Improvements of > 3 points were considered clinically meaningful.
Time Frame: BL (Day 0), Day 169, Day 365
Population: as for outcome 19
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Units on a Scale
  Day 169 (n=416, 207) | 8.82 (0.42) | 4.77 (0.59)
  Day 365 (n=417, 207) | 9.12 (0.43) | 4.97 (0.61)
Statistical Analysis 1: Comparison: ABA + MTX DB vs MTX + Placebo DB; Adjustment based on ANCOVA model with treatment as factor and baseline value as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; Adjusted Mean Difference at Day 169 = 4.06, 95% CI 2-sided [2.64 to 5.57]
Statistical Analysis 2: Comparison: ABA + MTX DB vs MTX + Placebo DB; Adjustment based on ANCOVA model with treatment as factor and baseline value as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; Adjusted Mean Difference at Day 365 = 4.15, 95% CI 2-sided [2.69 to 5.62]

21. Secondary Outcome: Participants in the DB Period Achieving an Extended Major Clinical Response
Description: An extended major clinical response (MCR) was defined as a continuous ACR 70 response over any nine month treatment period with study medications. ACR 70 response criteria requires a patient to have a 70% reduction in the number of swollen and tender joints, and a reduction of 70% in three of the following five parameters: physician global assessment of disease, patient global assessment of disease, patient assessment of pain, C-reactive protein or erythrocyte sedimentation rate, and degree of disability in HAQ score.
Time Frame: Day 1 to Day 365
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Participants | 26 | 1
Statistical Analysis 1: Comparison: ABA + MTX DB vs MTX + Placebo DB; Test type: Superiority or Other; p = 0.002, Chi-squared, Corrected; Estimated Difference = 5.7, 95% CI 2-sided [2.4 to 9.0] — Estimated difference between ABA + MTX and MTX + PLA is the estimated difference between ABA+MTX and MTX + PLA in the proportion of participants achieving extended MCR

22. Secondary Outcome: Mean BL DAS-28 C-Reactive Protein (CRP) and ESR in the DB Period
Description: The mean baseline CRP and ESR in the DB period on Day 169 and Day 365 was evaluated for all treated participants. Time-matched BL(Day 0) values and post-BL vales were presented for each post-BL visit and represent only that cohort of participants with measurements available at that post-BL assessment.
Time Frame: BL (Day 0), Day 169, Day 365
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg / mL
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
mg / mL
  BL (Day 0) CRP for Day 169 Cohort (n=418, 211) | 6.37 (0.83) | 6.36 (0.82)
  BL (Day 0) ESR for Day 169 Cohort (n=418, 211) | 6.82 (0.87) | 6.84 (0.82)
  BL (Day 0) CRP for Day 365 Cohort (n=424, 212) | 6.38 (0.83) | 6.35 (0.82)
  BL (Day 0) ESR for Day 365 Cohort (n=424, 212) | 6.82 (0.87) | 6.83 (0.82)

23. Secondary Outcome: Adjusted Mean Change From BL in DAS-28 CRP and ESR in the DB Period
Description: The mean change from baseline in CRP and ESR in the DB period was evaluated for all treated participants. Adjustment based on ANCOVA model with treatment as factor and baseline value as covariate.
Time Frame: BL (Day 0), Day 169, Day 365
Population: Due to the closure of a single site, 9 participants in the abatacept group and 5 in the placebo group were not included in this analysis. N = number of participants analyzed and n = the number of participants with measurements for that time point.
Measure: Mean (Standard Error); unit: mg / mL
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
mg / mL
  DAS-28 CRP Day 169 (n=418, 211) | -2.38 (0.06) | -1.29 (0.09)
  DAS-28 ESR Day 169 (n=418, 211) | -2.48 (0.07) | -1.33 (0.10)
  DAS-28 CRP Day 365 (n=424, 212) | -2.71 (0.06) | -1.41 (0.09)
  DAS-28 ESR Day 365 (n=424, 212) | -2.85 (0.07) | -1.46 (0.10)

24. Secondary Outcome: Mean BL Soluble Interleukin-2 Receptors (sIL2-r) in the DB Period
Description: The mean baseline sIL2-r in the DB period was evaluated from serum samples for all treated participants.
Time Frame: BL (Day 0), Day 169, Day 365
Population: All treated subjects in the DB period. N = number of participants analyzed and n = the number of participants with measurements for that time point.
Measure: Mean (Standard Deviation); unit: mg / mL
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
mg / mL
  Day 169 (n=370, 171) | 1776.0 (946.5) | 1603.0 (933.1)
  Day 365 (n=235, 106) | 1674.0 (835.1) | 1601.0 (1076.0)

25. Secondary Outcome: Mean Change From BL in Soluble Interleukin-2 Receptors (sIL2-r) in the DB Period
Description: The mean change from baseline in sIL2-r in the DB period was evaluated for all treated participants.
Time Frame: BL (Day 0), Day 169, Day 365
Population: All treated subjects in the DB period.
Measure: Mean (Standard Error); unit: mg / mL
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
mg / mL
  Day 169 (n=370, 171) | -519.00 (23.72) | -85.50 (32.78)
  Day 365 (n=235, 106) | -562.00 (40.82) | -290.00 (87.97)

26. Secondary Outcome: ACR Core Component: Mean Number of Tender Joints at All Post-BL Visits in the DB Period
Description: Time-matched BL(Day 0) values and post-BL vales were presented for each post-BL visit and represent only that cohort of participants with measurements available at that post-BL assessment.
Time Frame: Day 15, Day 29, Day 57, Day 85, Day 113, Day 141, Day 169, Day 225, Day 281, Day 365
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Joints
  BL (Day 0) for Day 15 Cohort (n=416, 210) | 25.19 (14.62) | 27.93 (14.27)
  BL (Day 0) for Day 29 Cohort (n=419, 211) | 21.14 (14.69) | 24.11 (14.97)
  BL (Day 0) for Day 57 Cohort (n=421, 210) | 16.70 (14.06) | 21.41 (14.15)
  BL (Day 0) for Day 85 Cohort (n=417, 208) | 14.84 (13.98) | 20.58 (15.61)
  BL (Day 0) for Day 113 Cohort (n=415, 210) | 13.55 (13.35) | 19.83 (15.29)
  BL (Day 0) for Day 141 Cohort (n=420, 211) | 12.59 (13.39) | 19.78 (15.74)
  BL (Day 0) for Day 169 Cohort (n=420, 211) | 11.69 (12.37) | 18.70 (15.42)
  BL (Day 0) for Day 225 Cohort (n=419, 212) | 10.42 (12.04) | 18.22 (15.46)
  BL (Day 0) for Day 281Cohort (n=419, 211) | 9.92 (11.37) | 17.10 (16.04)
  BL (Day 0) for Day 365 Cohort (n=424, 212) | 9.96 (11.87) | 18.31 (15.72)

27. Secondary Outcome: ACR Core Component: Mean Number of Swollen Joints at All Post-BL Visits in the DB Period
Description: The mean number of swollen joints in the DB period was evaluated based on the swollen joint core component of the ACR scoring system where increasing score indicates increasing level of severity. Time-matched BL(Day 0) values and post-BL vales were presented for each post-BL visit and represent only that cohort of participants with measurements available at that post-BL assessment.
Time Frame: Day 15, Day 29, Day 57, Day 85, Day 113, Day 141, Day 169, Day 225, Day 281, Day 365
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
joints
  BL (Day 0) for Day 15 Cohort (n=416, 210) | 16.40 (8.63) | 18.49 (9.92)
  BL (Day 0) for Day 29 Cohort (n=419, 211) | 14.04 (9.26) | 16.03 (9.23)
  BL (Day 0) for Day 57 Cohort (n=421, 210) | 11.02 (8.64) | 14.77 (9.85)
  BL (Day 0) for Day 85 Cohort (n=417, 208) | 9.76 (8.99) | 14.56 (10.83)
  BL (Day 0) for Day 113 Cohort (n=415, 210) | 8.73 (8.64) | 13.93 (10.69)
  BL (Day 0) for Day 141 Cohort (n=420, 211) | 7.84 (8.10) | 13.28 (10.70)
  BL (Day 0) for Day 169 Cohort (n=420, 211) | 7.54 (7.77) | 13.14 (11.05)
  BL (Day 0) for Day 225 Cohort (n=419, 212) | 6.80 (7.57) | 12.78 (11.06)
  BL (Day 0) for Day 281 Cohort (n=419, 211) | 6.50 (7.52) | 12.46 (10.98)
  BL (Day 0) for Day 365 Cohort (n=424, 212) | 6.31 (7.16) | 12.69 (10.84)

28. Secondary Outcome: ACR Core Component: Mean Participant Pain Assessment at All Post-BL Visits in the DB Period
Description: Participant self-reported pain assessment core component of the ACR scoring system where increasing score indicates increasing level of severity as indicated on a 100mm Visual Analog Scale (VAS) with 0mm representing no pain and 100mm representing the most pain possible.
Time Frame: Day 15, Day 29, Day 57, Day 85, Day 113, Day 141, Day 169, Day 225, Day 281, Day 365
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Units on a Scale
  Day 15 (n=413, 210) | 52.39 (22.85) | 60.08 (21.90)
  Day 29 (n=418, 211) | 47.03 (23.84) | 54.69 (23.86)
  Day 57 (n=419, 209) | 40.34 (24.29) | 50.11 (25.16)
  Day 85 (n=417, 207) | 35.97 (24.01) | 48.36 (25.53)
  Day 113 (n=418, 210) | 34.31 (23.61) | 48.60 (26.99)
  Day 141 (n=420, 211) | 33.93 (25.47) | 48.26 (27.19)
  Day 169 (n=421, 211) | 32.69 (24.32) | 49.21 (27.13)
  Day 225 (n=418, 211) | 31.39 (24.01) | 47.20 (26.77)
  Day 281 (n=419, 210) | 31.06 (24.58) | 46.18 (27.23)
  Day 365 (n=424, 212) | 29.78 (24.20) | 48.17 (27.82)

29. Secondary Outcome: ACR Core Component: Mean Participant Physical Function Assessment at All Post-BL Visits in the DB Period
Description: as for outcome 2
Time Frame: Day 15, Day 29, Day 57, Day 85, Day 113, Day 141, Day 169, Day 225, Day 281, Day 365
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Units on a Scale
  Day 15 (n=405, 206) | 1.51 (0.64) | 1.58 (0.56)
  Day 29 (n=406, 207) | 1.41 (0.64) | 1.47 (0.60)
  Day 57 (n=412, 205) | 1.29 (0.65) | 1.42 (0.63)
  Day 85 (n=407, 203) | 1.18 (0.68) | 1.32 (0.65)
  Day 113 (n=409, 206) | 1.16 (0.67) | 1.35 (0.68)
  Day 141 (n=411, 207) | 1.13 (0.71) | 1.35 (0.70)
  Day 169 (n=413, 207) | 1.11 (0.70) | 1.31 (0.69)
  Day 225 (n=409, 207) | 1.06 (0.70) | 1.35 (0.70)
  Day 281 (n=408, 207) | 1.05 (0.70) | 1.31 (0.68)
  Day 365 (n=415, 208) | 1.04 (0.70) | 1.34 (0.70)

30. Secondary Outcome: ACR Core Component: Mean Participant Global Assessment at All Post-BL Visits in the DB Period
Description: Participant self-reported global RA assessment core component of the ACR scoring system where increasing score indicates increasing level of severity as indicated on a 100mm Visual Analog Scale (VAS) with 0mm representing no pain and 100mm representing the most pain possible.
Time Frame: Day 15, Day 29, Day 57, Day 85, Day 113, Day 141, Day 169, Day 225, Day 281, Day 365
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Units on a Scale
  Day 15 (n=413, 210) | 50.90 (22.42) | 56.66 (22.33)
  Day 29 (n=418, 211) | 45.26 (22.72) | 53.11 (22.81)
  Day 57 (n=419, 209) | 39.78 (23.02) | 49.34 (23.98)
  Day 85 (n=417, 207) | 35.07 (23.37) | 46.82 (24.71)
  Day 113 (n=418, 210) | 33.98 (22.59) | 47.26 (25.69)
  Day 141 (n=420, 211) | 33.52 (24.06) | 47.52 (26.57)
  Day 169 (n=421, 211) | 32.37 (23.26) | 47.93 (26.24)
  Day 225 (n=418, 210) | 30.63 (22.48) | 46.06 (26.21)
  Day 281 (n=419, 211) | 29.98 (23.25) | 44.45 (26.13)
  Day 365 (n=424, 212) | 28.95 (23.60) | 45.62 (26.92)

31. Secondary Outcome: ACR Core Component: Mean Physician Global Assessment at All Post-BL Visits in the DB Period
Description: Physician global RA assessment core component of the ACR scoring system where increasing score indicates increasing level of severity as indicated on a 100mm Visual Analog Scale (VAS) with 0mm representing very good global RA assessment and 100mm representing very poor global RA assessment.
Time Frame: Day 15, Day 29, Day 57, Day 85, Day 113, Day 141, Day 169, Day 225, Day 281, Day 365
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Units on a Scale
  Day 15 (n=415, 209) | 52.79 (19.24) | 56.68 (18.93)
  Day 29 (n=418, 211) | 45.24 (20.58) | 51.83 (20.14)
  Day 57 (n=421, 210) | 35.89 (19.84) | 45.21 (22.61)
  Day 85 (n=416, 208) | 31.07 (20.12) | 42.59 (23.87)
  Day 113 (n=412, 209) | 29.01 (20.40) | 42.20 (24.72)
  Day 141 (n=420, 211) | 26.71 (20.38) | 41.22 (25.33)
  Day 169 (n=421, 211) | 25.44 (19.65) | 41.75 (25.79)
  Day 225 (n=418, 212) | 24.34 (19.27) | 40.68 (26.15)
  Day 281 (n=419, 210) | 23.33 (19.09) | 38.76 (26.70)
  Day 365 (n=424, 212) | 21.58 (19.53) | 41.04 (25.91)

32. Secondary Outcome: ACR Core Component: Mean CRP at All Post-BL Visits in the DB Period
Description: CRP core component of the ACR scoring system was evaluated from serum samples in which increasing levels indicate increasing level of disease.
Time Frame: Day 15, Day 29, Day 57, Day 85, Day 113, Day 141, Day 169, Day 225, Day 281, Day 365
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: IU / mL
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
IU / mL
  Day 15 (n=401, 199) | 3.27 (3.13) | 2.65 (2.34)
  Day 29 (n=410, 208) | 1.94 (1.99) | 2.65 (2.48)
  Day 57 (n=416, 209) | 1.70 (2.02) | 2.36 (2.34)
  Day 85 (n=412, 203) | 1.53 (1.97) | 2.53 (2.39)
  Day 113 (n=417, 209) | 1.49 (1.69) | 2.55 (2.59)
  Day 141 (n=414, 209) | 1.27 (1.52) | 2.48 (2.61)
  Day 169 (n=420, 211) | 1.42 (1.67) | 2.56 (2.43)
  Day 225 (n=414, 212) | 1.30 (1.55) | 2.46 (2.70)
  Day 281 (n=412, 210) | 1.36 (1.80) | 2.60 (3.09)
  Day 365 (n=424, 212) | 1.27 (1.63) | 2.41 (2.58)

33. Secondary Outcome: Number of Participants Discontinuing in the DB Period
Description: Participants that discontinued treatment during the DB period for any reason were evaluated after 6 months and 1 year of treatment.
Time Frame: Day 1 to Day 169, Day 170 to Day 365
Population: All randomized and treated participants in the DB period.
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 433 | 219
Participants
  Day 1 to 169 Discontinuations (DC) - All Causes | 32 | 45
  Day 1 to 169 DC Due to Lack of Efficacy | 11 | 33
  Day 170 to Day 365 DC - All Causes | 16 | 12
  Day 170 to Day 365 DC Due to Lack of Efficacy | 2 | 7

34. Secondary Outcome: Change From BL in Joint Narrowing Score (JSN), Erosion Score (ES), and Total Score (TS) by Category in the DB Period
Description: To assess joint damage progression, the Genant-modified Sharp scoring method was used to evaluate radiographs of hands/wrists and feet for erosions and joint space narrowing (JSN). The total Genant-modified Sharp score ranges from 0 (no radiographic damage) to 290 (worst possible radiographic damage) and is the sum of the erosion score (range 0-145) and the joint space narrowing score (range 0-145). Higher scores indicated more damage. Improvement=decreases from BL, stable=same as BL, worsening=increases from BL.
Time Frame: BL (Day 0), Day 365
Population: This analysis was not completed.
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 0 | 0

35. Primary Outcome: Participants With Deaths, Adverse Events (AEs) and SAEs in the Open-Label (OL) Period
Description: as for outcome 17
Time Frame: Day 365 to Day 2,185
Population: All treated participants in the OL period.
Measure: Number; unit: Participants
Groups:
- ABA + MTX OL: Abatacept was dosed intravenously by weight at 10 mg/kg in the OL period under tiered dosing such that participants weighing < 60 kg received abatacept 500 mg; participants ≥ 60 kg and ≤ 100 kg received abatacept 750 mg; and participants > 100 kg received abatacept 1 g. MTX was continued at the dose used in the DB period.
Arm/Group | ABA + MTX OL
Number analyzed (Participants) | 539
Participants
  Deaths | 17
  SAEs | 215
  Related SAEs | 60
  Discontinuations Due to SAEs | 36
  AEs | 518
  Related AEs | 323
  Discontinued Due to AEs | 49

36. Primary Outcome: Participants With Hematology Values Meeting the Marked Abnormality Criteria in the OL Period
Description: Marked abnormality criteria are: Hemoglobin (HGB): >3 g/dL decrease from BL; Hematocrit: <0.75 * BL; Erythrocytes: <0.75 * BL; Platelets (PLT): <0.67 * LLN/>1.5 * ULN, or if BL < LLN then use <0.5 * BL and <100,000 mm^3; Leukocytes: <0.75 * LLN/ >1.25 * ULN, or if BL<LLN then use <0.8 * BL or >ULN, or if BL>ULN then use >1.2 * BL or <LLN; neutrophils+bands: <1.0 * 10^3 c/uL; eosinophils: >0.750 * 10^3 c/uL; basophils: > 400 mm^3; monocytes: >2000 mm^3; lymphocytes: <0.750 * 10^3 c/uL/ >7.50 * 10^3 c/uL.
Time Frame: Day 365 to Day 2,185
Population: All treated participants in the OL period.
Measure: Number; unit: Participants
Arm/Group | ABA + MTX OL
Number analyzed (Participants) | 536
Participants
  Low Hemoglobin (LLN 11.5 g/dL) | 21
  Low Hematocrit (LLN 34%) | 20
  Low Erythrocytes (LLN 38 x 10^6 c/µL) | 15
  Low Platelet Count (LLN 140 x 10^3 c/µL) | 9
  High Platelet Count (ULN 415 x 10^3 c/µL) | 4
  Low Leukocytes (LLN 4 x 10^3 c/µL) | 53
  High Leukocytes (ULN 10.5 x 10^3 c/µL) | 68
  Low Absolute Neutrophils (LLN 1.8 x 10^3 c/µL) | 14
  Low Absolute Lymphocytes (LLN 0.7 x 10^3 c/µL) | 109
  High Absolute Lymphocytes (ULN 4.5 x 10^3 c/µL) | 4
  High Absolute Monocytes (ULN 1.0 x 10^3 c/µL) | 9
  High Absolute Basophils (ULN 0.2 x 10^3 c/µL) | 3
  High Absolute Eosinophils (ULN 0.4 x 10^3 c/µL) | 49

37. Primary Outcome: Participants With Liver and Kidney Function Values Meeting the Marked Abnormality Criteria in the OL Period
Description: as for outcome 36
Time Frame: Day 365 to Day 2,185
Population: All treated participants in the OL period.
Measure: Number; unit: Participants
Arm/Group | ABA + MTX OL
Number analyzed (Participants) | 536
Participants
  High ALP (ULN 150 U/L) | 3
  High AST (ULN 40 U/L) | 14
  High ALT (ULN 55 U/L) | 20
  High GGT (ULN 65 U/L) | 36
  High Bilirubin (ULN 1.2 mg/dL) | 6
  High BUN (ULN 26 mg/dL) | 40
  High Creatinine (ULN 1.5 mg/dL) | 92

38. Primary Outcome: Participants With Electrolyte Values Meeting the Marked Abnormality Criteria in the OL Period
Description: Sodium < 0.9 * LLN or > 1.05 * ULN or if BL < LLN then use < 0.95 * BL or > ULN or if BL > ULN then use >1.05 *BL or < LLN; Potassium: < 0.9 * LLN or > 1.1 * ULN or if BL < LLN then use < 0.9 * BL or > ULN or if BL > ULN then use 1.1 * BL or < LLN; Chloride: < 0.9 * LLN or > 1.1 * ULN or if BL < LLN then use <0.9 * BL or >ULN or if BL > ULN then use > 1.1 * BL or < LLN; Calcium <0.8 * LLN or > 1.2 * ULN or if BL < LLN then use <0.67 * BL or > ULN or if BL > ULN then use > 1.3 * BL or < LLN.
Time Frame: Day 365 to Day 2,185
Population: All treated participants in the OL period.
Measure: Number; unit: Participants
Arm/Group | ABA + MTX OL
Number analyzed (Participants) | 536
Participants
  Low Sodium (LLN 135 mmol/L) | 11
  High Sodium (ULN 148 mmol/L) | 2
  Low Potassium (LLN 3.5 mmol/L) | 11
  High Potassium (ULN 5.5 mmol/L) | 32
  Low Chloride (LLN 96 mmol/L) | 1
  High Chloride (ULN 109 mmol/L) | 0
  Low Calcium (LLN 8.5 mg/dL) | 0
  High Calcium (ULN 10.6 mg/dL) | 1
  Low Phosphorous (LLN 2.5 mg/dL) | 16
  High Phosphorous (ULN 5.6 mg/dL) | 8

39. Primary Outcome: Participants With Glucose, Protein, Metabolites, and Urinalysis Values Meeting the Marked Abnormality Criteria in the OL Period
Description: Glucose: < 65 mg/dL or > 220 mg/dL; Fasting Glucose: <0.8 * LLN or > 1.5 * ULN or if BL < LLN then use < 0.8 * BL or > ULN or if BL > ULN then use 1.1 * BL or < LLN; Total protein: < 0.9 * LLN or 1.1 * ULN or if BL < LLN then use 0.9 * BL or > ULN or if BL > ULN then use 1.1 * BL or < LLN; Albumin: < 0.9 * LLN or if BL < LLN then use 0.75 * BL; Uric acid: > 1.5 * ULN or if BL > ULN then use > 2.0 * BL. All urinalysis abnormalities were defined as: if missing BL then use >= 2 or if value >=4, or if BL = 0 or 0.5 then use >= 2, or if BL = 1.0 then use >= 3, or if BL = 2.0 then use >=4.
Time Frame: Day 365 to Day 2,185
Population: All treated participants in the OL period.
Measure: Number; unit: Participants
Arm/Group | ABA + MTX OL
Number analyzed (Participants) | 536
Participants
  Low Serum Glucose (LLN 64 mg/dL) | 120
  High Serum Glucose (ULN 140 mg/dL) | 36
  Low Serum Fasting Glucose (LLN 65 mg/dL) | 25
  High Serum Fasting Glucose (ULN 109 mg/dL) | 22
  Low Total Protein (LLN 6 g/dL) | 11
  High Total Protein (ULN 8.5 g/dL) | 6
  Low Albumin (LLN 3.5 g/dL) | 15
  High Uric Acid (ULN 8.7 mg/dL) | 4
  High Urine Protein (ULN Trace) | 39
  High Urine Glucose (ULN Trace) | 39
  High Urine Ketones (ULN Positive) | 1
  High Urine Blood (ULN >=0) | 141
  High Urine Leukocyte Esterase (ULN >=0) | 35
  High Urine White Blood Count (ULN 12 hpf) | 232
  High Urine Red Blood Count (ULN 8 hpf) | 181

40. Secondary Outcome: Participants Experiencing Clinically Significant Changes in Vital Signs in the DB Period
Description: All changes in participant vital signs were monitored on each day of study drug administration prior to dosing and 60 minutes after dosing. Vital signs included body temperature, heart rate, and seated blood pressure. Clinical significance was defined as any change from baseline that resulted in a value outside the normal limits for the participant.
Time Frame: Day 1 to Day 365
Population: All randomized and treated participants.
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 433 | 219
Participants | 0 | 0

41. Secondary Outcome: Participants Experiencing AEs of Special Interest in the DB Period
Description: AEs were defined as any new untoward medical occurrence or worsening of a pre- existing medical condition which does not necessarily have a causal relationship with this treatment. AEs were identified as those which may be associated with the use of immunomodulatory agents or infusion of therapeutic proteins. Acute infusional AEs were defined as those that occurred within 1 hour after the start of the infusion.
Time Frame: Day 1 to Day 365
Population: All treated participants in the DB period.
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 433 | 219
Participants
  Infections/Infestations | 50 | 12
  Neoplasms | 14 | 9
  Autoimmune Disorders | 13 | 2
  Acute Infusional AEs | 38 | 9

42. Secondary Outcome: Mean BL Individual Components of the HAQ DI at Day 169 and Day 365
Description: as for outcome 2
Time Frame: BL (Day 0), Day 169, Day 365
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Units on a Scale
  HAQ DI Day 169 (n=373, 159) | 1.68 (0.63) | 1.70 (0.59)
  HAQ DI Day 365 (n=369, 160) | 1.68 (0.63) | 1.70 (0.58)
  Dressing and Grooming Day 169 (n=374, 159) | 1.48 (0.75) | 1.48 (0.73)
  Dressing and Grooming Day 365 (n=372, 160) | 1.47 (0.75) | 1.49 (0.73)
  Arising Day 169 (n=373, 159) | 1.42 (0.83) | 1.45 (0.79)
  Arising Day 365 (n=372, 160) | 1.42 (0.82) | 1.46 (0.78)
  Eating Day 169 (n=374, 159) | 1.63 (0.97) | 1.67 (0.84)
  Eating Day 365 (n=372, 160) | 1.63 (0.97) | 1.68 (0.84)
  Walking Day 169 (n=373, 158) | 1.40 (0.83) | 1.36 (0.78)
  Walking Day 365 (n=372, 158) | 1.40 (0.83) | 1.37 (0.78)
  Hygiene Day 169 (n=373, 159) | 1.93 (0.90) | 1.91 (0.89)
  Hygiene Day 365 (n=370, 160) | 1.93 (0.90) | 1.91 (0.89)
  Reaching Day 169 (n=373, 159) | 1.94 (0.86) | 1.97 (0.80)
  Reaching Day 365 (n=370, 160) | 1.94 (0.86) | 1.97 (0.80)
  Gripping Day 169 (n=374, 159) | 1.80 (0.76) | 1.90 (0.67)
  Gripping Day 365 (n=371, 160) | 1.80 (0.76) | 1.90 (0.67)
  Activities Day 169 (n=373, 159) | 1.87 (0.79) | 1.86 (0.82)
  Activities Day 365 (n=369, 160) | 1.87 (0.79) | 1.86 (0.82)

43. Secondary Outcome: Adjusted Mean Change From BL in Individual Components of the HAQ DI at Day 169
Description: as for outcome 2
Time Frame: Day 169
Population: Analyses of efficacy were based on the intent-to-treat population. Due to the non-compliance of a single site, 9 participants in the abatacept group and 5 in the placebo group were not included in this analysis. Last observation carried forward (LOCF) analysis.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Units on a Scale
  HAQ DI | -0.62 (0.03) | -0.52 (0.05)
  Dressing and Grooming | -0.73 (0.04) | -0.55 (0.05)
  Arising | -0.69 (0.03) | -0.65 (0.05)
  Eating | -0.68 (0.04) | -0.48 (0.06)
  Walking | -0.58 (0.04) | -0.45 (0.05)
  Hygiene | -0.48 (0.05) | -0.40 (0.07)
  Reaching | -0.64 (0.04) | -0.52 (0.06)
  Gripping | -0.53 (0.04) | -0.43 (0.06)
  Activities | -0.57 (0.04) | -0.43 (0.06)

44. Secondary Outcome: Adjusted Mean Change From BL in Individual Components of the HAQ DI at Day 365
Description: as for outcome 2
Time Frame: Day 365
Population: as for outcome 43
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Units on a Scale
  HAQ DI | -0.68 (0.03) | -0.51 (0.06)
  Dressing and Grooming | -0.78 (0.04) | -0.61 (0.06)
  Arising | -0.75 (0.04) | -0.58 (0.05)
  Eating | -0.81 (0.04) | -0.44 (0.06)
  Walking | -0.61 (0.04) | -0.50 (0.06)
  Hygiene | -0.53 (0.05) | -0.37 (0.07)
  Reaching | -0.70 (0.04) | -0.59 (0.07)
  Gripping | -0.65 (0.04) | -0.44 (0.07)
  Activities | -0.66 (0.44) | -0.47 (0.07)

45. Secondary Outcome: Number of Participants With Immunogenicity to Abatacept in the DB Period
Description: Participants with titers to abatacept in the DB period. Serum samples from abatacept-treated adult participants with active RA were screened for the presence of drug-specific antibodies using two validated direct-format enzyme-linked immunosorbent assays (ELISAs) to determine the presence of antibodies to abatacept and/or CTLA4-T.
Time Frame: Day 1 to Day 365
Population: Participants treated with abatacept in the DB period with at least one immunogenicity sample collected in the DB period.
Measure: Number; unit: Participants
Groups:
- ABA + MTX DB: Abatacept was dosed intravenously by weight at 10 mg/kg in the DB period under tiered dosing such that participants weighing < 60 kg received abatacept 500 mg; particiapnts ≥ 60 kg and ≤ 100 kg received abatacept 750 mg; and particpants > 100 kg received abatacept 1 g. MTX was continued at the dose used in the OL period.
Arm/Group | ABA + MTX DB
Number analyzed (Participants) | 406
Participants | 6

46. Secondary Outcome: Number of New Tender Joints and Number of New Swollen Joints in the DB Period
Description: Tender joints and swollen joints are core components of the ACR 20, 50, and 70. The incidences of new tender joints and new swollen joints were evaluated in the DB period after 6 months and 1 year of treatment.
Time Frame: Day 169, Day 365
Population: These data were not summarized as it was determined that no meaningful information would be obtained.
Measure: Number; unit: Joints
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 0 | 0

47. Secondary Outcome: Number of Participants Experiencing a 100% Reduction in Tender Joints or 100% Reduction in Swollen Joints in the DB Period
Time Frame: Day 169, Day 365
Population: as for outcome 43
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
Participants
  100% Reduction in New Tender Joints Day 169 | 43 | 9
  100% Reduction in New Swollen Joints Day 169 | 59 | 14
  100% Reduction in New Tender Joints Day 365 | 67 | 8
  100% Reduction in New Swollen Joints Day 365 | 78 | 9

48. Secondary Outcome: Number of Participants With Hematology Laboratories Meeting Marked Abnormality Criteria in the DB Period
Description: Marked abnormality criteria were: Hemoglobin (HGB): >3 g/dL decrease from BL; Hematocrit: <0.75 * BL; Erythrocytes: <0.75 * BL; Platelets (PLT): <0.67 * LLN/>1.5 * ULN, or if BL < LLN then use <0.5 * BL and <100,000 mm^3; Leukocytes: <0.75 * LLN/ >1.25 * ULN, or if BL<LLN then use <0.8 * BL or >ULN, or if BL>ULN then use >1.2 * BL or <LLN; neutrophils+bands: <1.0 * 10^3 c/uL; eosinophils: >0.750 * 10^3 c/uL; basophils: > 400 mm^3; monocytes: >2000 mm^3; lymphocytes: <0.750 * 10^3 c/uL/ >7.50 * 10^3 c/uL.
Time Frame: Day 1 to Day 365
Population: All treated participants in the DB period.
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 433 | 219
Participants
  Low Hemoglobin (LLN 11.5 g/dL) | 7 | 4
  Low Hematocrit (LLN 34%) | 4 | 3
  Low Platelet Count (LLN 140 x 10^3 c/uL) | 4 | 1
  High Platelet Count (ULN 415 x 10^3 c/uL) | 1 | 0
  Low Leukocytes (LLN 4.0 x 10^3 c/uL) | 15 | 4
  High Leukocytes (ULN 10.5 x 10^3 c/uL) | 45 | 33
  Low Absolute Neutrophils (LLN 1.8 x 10^3 c/uL) | 10 | 3

49. Secondary Outcome: Number of Participants With Liver and Kidney Function Tests Meeting Marked Abnormality Criteria in the DB Period
Description: Marked abnormality criteria were: Aspartate Aminotransferase (AST) >3 * ULN or if BL > ULN then use >4 *BL; Alanine Aminotransferase (ALT) >3 * ULN or if BL > ULN then use > 4 * BL; Creatinine > 1.5 * BL.
Time Frame: Day 1 to Day 365
Population: All treated participants in the DB period.
Measure: Number; unit: Participants
Groups:
- Placebo + MTX DB: Control group receiving MTX treatment in combination with placebo. Participants received MTX at a minimum dose of 10-30 mg/wk, although doses of < 10 mg/wk were acceptable if due to toxicity. Placebo and MTX were administered IV on Days 1, 15, 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337.
Arm/Group | ABA + MTX DB | Placebo + MTX DB
Number analyzed (Participants) | 433 | 219
Participants
  High AST (ULN 40 U/L) | 4 | 2
  High ALT (ULN 55 U/L) | 7 | 5
  High Creatinine (ULN 1.5 mg/ dL) | 23 | 15

50. Secondary Outcome: Mean BL ESR and CRP Levels in the OL Period
Description: Mean baseline values are reported for each cohort at each time point.
Time Frame: BL (Day 0), Day 365, Day 729, Day 1,093, Day 1,457, Day 1,821, Day 1,989, Day 2,185
Population: All treated participants in the OL period. Treatment groups represent treatment received in the DB period. N = number of participants analyzed and n = the number of participants with measurements for that time point.
Measure: Mean (Standard Deviation); unit: IU / mL
Groups:
- ABA + MTX DB: Abatacept was dosed intravenously by weight at 10 mg/kg in the OL period under tiered dosing such that participants weighing < 60 kg received abatacept 500 mg; particiapnts ≥ 60 kg and ≤ 100 kg received abatacept 750 mg; and particpants > 100 kg received abatacept 1 g. MTX was continued at the dose used in the DB period.
- MTX + Placebo DB: Participants that received MTX + placebo in the DB treatment period (Day 1 to Day 365) but are currently receiving treatment with ABA +MTX in the OL period. Abatacept was dosed intravenously by weight at 10 mg/kg in the OL period under tiered dosing such that participants weighing < 60 kg received abatacept 500 mg; particiapnts ≥ 60 kg and ≤ 100 kg received abatacept 750 mg; and particpants > 100 kg received abatacept 1 g. MTX was continued at the dose used in the DB period.
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 378 | 161
IU / mL
  ESR Day 365 (n=343, 141) | 43.56 (22.98) | 43.61 (25.25)
  CRP Day 365 (n=373, 160) | 32.48 (31.41) | 24.72 (20.74)
  ESR Day 729 (n=307, 132) | 43.74 (23.44) | 41.37 (24.15)
  CRP Day 729 (n=348, 153) | 32.12 (30.99) | 23.46 (19.65)
  ESR Day 1,093 (n=283, 123) | 43.57 (23.34) | 42.41 (25.25)
  CRP Day 1,093 (n=306, 131) | 31.96 (30.35) | 24.09 (19.85)
  ESR Day 1,457 (n=270, 111) | 43.49 (23.71) | 42.87 (24.27)
  CRP Day 1,457 (n=295, 132) | 32.13 (30.14) | 23.20 (19.22)
  ESR Day 1,821 (n=257, 109) | 43.03 (22.86) | 41.83 (24.01)
  CRP Day 1,821 (n=275, 124) | 31.41 (29.30) | 22.14 (18.34)
  ESR Day 1,989 (n=114, 49) | 42.61 (24.00) | 38.78 (19.64)
  CRP Day 1,989 (n=128, 61) | 33.22 (34.65) | 20.39 (14.43)
  ESR Day 2,185 (n=76, 29) | 45.04 (23.46) | 39.17 (21.30)
  CRP Day 2,185 (n=83, 38) | 34.73 (36.05) | 22.08 (15.69)

51. Secondary Outcome: Mean Change From BL in ESR in the OL Period
Description: Serum samples were evaluated from study participants to determine the mean change from baseline in ESR values.
Time Frame: BL (Day 0), Day 365, Day 729, Day 1,093, Day 1,457, Day 1,821, Day 1,989, Day 2,185
Population: as for outcome 50
Measure: Mean (Standard Error); unit: IU / mL
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 378 | 161
IU / mL
  Day 365 (n=343, 141) | -17.9 (1.21) | -6.85 (1.74)
  Day 729 (n=307, 132) | -19.3 (1.29) | -16.3 (1.91)
  Day 1,093 (n=283, 123) | -17.2 (1.55) | -16.6 (2.15)
  Day 1,457 (n=270, 111) | -17.7 (1.41) | -16.3 (2.33)
  Day 1,821 (n=257, 109) | -17.7 (1.46) | -16.6 (2.26)
  Day 1,989 (n=114, 49) | -17.3 (2.33) | -13.3 (3.12)
  Day 2,185 (n=76, 29) | -22.1 (2.92) | -21.0 (4.45)

52. Secondary Outcome: Participant RF Seroconversion in the OL Period
Description: This analysis determined participant RF status (positive or RF negative) based on serum samples at each specified timepoint. A positive value for RF was > 20 IU/ml; a negative value for RF was ≤ 20 IU/mL.
Time Frame: Day 365, Day 729, Day 1,093, Day 1,457, Day 1,821, Day 2,185
Population: as for outcome 50
Measure: Number; unit: Participants
Groups:
- MTX + Placebo DB: Participants that received MTX + placebo in the DB treatment period (Day 1 to Day 365) but are currently receiving treatment with ABA +MTX in the OL period. Abatacept was dosed intravenously by weight at 10 mg/kg in the OL period under tiered dosing such that participants weighing < 60 kg received abatacept 500 mg; participants ≥ 60 kg and ≤ 100 kg received abatacept 750 mg; and participants > 100 kg received abatacept 1 g. MTX was continued at the dose used in the DB period.
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 378 | 161
Participants
  Positive Seroconversion Day 365 (n=347, 146) | 2 | 3
  Negative Seroconversion Day 365 (n=347, 146) | 31 | 2
  Positive Seroconversion Day 729 (n=330, 143) | 8 | 1
  Negative Seroconversion Day 729 (n=330, 143) | 31 | 10
  Positive Seroconversion Day 1,093 (n=280, 119) | 6 | 3
  Negative Seroconversion Day 1,093 (n=280, 119) | 27 | 7
  Positive Seroconversion Day 1,457 (n=275, 118) | 5 | 4
  Negative Seroconversion Day 1,457 (n=275, 118) | 27 | 8
  Positive Seroconversion Day 1,821 (n=255, 115) | 4 | 5
  Negative Seroconversion Day 1,821 (n=255, 115) | 25 | 9
  Positive Seroconversion Day 2,185 (n=75, 31) | 3 | 3
  Negative Seroconversion Day 2,185 (n=75, 31) | 7 | 2

53. Secondary Outcome: Number of ACR 20 Responders in the DB and OL Periods
Description: ACR 20 response requires a patient to have a 20% reduction in the number of swollen and tender joints, and a reduction of 20% in three of the following five parameters: physician global assessment of disease, patient global assessment of disease, patient assessment of pain, CRP or ESR, and degree of disability in HAQ score. A participant achieved a sustained ACR 20 response if the participant had ACR 20 observed for at least 2 consecutive study visits.
Time Frame: Day 15, Day 29, Day 57, Day 85, Day 113, Day 141, Day 169, Day 225, Day 281, Day 365, Day 449, Day 533, Day 617, Day 729, Day 813, Day 897, Day 981, Day 1,083, Day 1,177, Day 1,261, Day 1,345, Day 1,497, Day 1,625, Day 1,821
Population: All treated participants in the OL period (Treatment groups represent treatment received in the DB period). Due to the non-compliance of a single site, 3 participants were not included in this analysis. N = number of participants analyzed and n = the number of participants with measurements for that time point.
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Participants
  Day 15 (n = 370, n = 158) | 95 | 26
  Day 29 (n = 368, n=158) | 145 | 44
  Day 57 (n = 371, n = 159) | 218 | 66
  Day 85 (n = 367, n = 158) | 246 | 70
  Day 113 (n = 367, n = 159) | 266 | 79
  Day 141 (n = 368, n = 159) | 275 | 85
  Day 169 (n = 371, n = 159) | 272 | 79
  Day 225 (n = 369, n = 158) | 302 | 86
  Day 281 (n = 367, n = 159) | 299 | 92
  Day 365 (n = 373, n = 159) | 307 | 86
  Day 449 (n = 363, n = 155) | 299 | 122
  Day 533 (n = 353, n = 155) | 300 | 127
  Day 617 (n = 347, n = 155) | 299 | 127
  Day 729 (n = 337, n = 147) | 296 | 122
  Day 813 (n = 322, n = 143) | 273 | 124
  Day 897 (n = 311, n = 136) | 260 | 117
  Day 981 (n = 298, n = 133) | 243 | 110
  Day 1,093 (n = 303, n = 134) | 257 | 111
  Day 1,177 (n = 265, n = 117) | 228 | 101
  Day 1,261 (n = 289, n = 131) | 251 | 107
  Day 1,345 (n = 133, n = 53) | 108 | 43
  Day 1,457 (n = 288, n = 128) | 253 | 110
  Day 1,625 (n = 273, n= 126) | 236 | 112
  Day 1,821 (n = 268, n = 123) | 224 | 106
  Day 1,989 (n = 119, n = 54) | 103 | 45
  Day 2,185 (n = 85, n = 37) | 72 | 34

54. Secondary Outcome: Number of ACR 50 Responders in the DB and OL Periods
Description: ACR 50 response requires a patient to have a 50% reduction in the number of swollen and tender joints, and a reduction of 50% in three of the following five parameters: physician global assessment of disease, patient global assessment of disease, patient assessment of pain, CRP or ESR, and degree of disability in HAQ score.
Time Frame: as for outcome 53
Population: as for outcome 53
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Participants
  Day 15 (n = 371, n = 160) | 12 | 2
  Day 29 (n = 368, n=158) | 35 | 8
  Day 57 (n = 373, n = 159) | 82 | 15
  Day 85 (n = 367, n = 158) | 128 | 16
  Day 113 (n = 368, n = 159) | 142 | 25
  Day 141 (n = 371, n = 159) | 157 | 38
  Day 169 (n = 373, n = 159) | 163 | 35
  Day 225 (n = 370, n = 159) | 188 | 42
  Day 281 (n = 369, n = 159) | 193 | 38
  Day 365 (n = 372, n = 160) | 202 | 40
  Day 449 (n = 366, n = 155) | 214 | 70
  Day 533 (n = 348, n = 156) | 213 | 82
  Day 617 (n = 346, n = 155) | 213 | 87
  Day 729 (n = 338, n = 147) | 207 | 93
  Day 813 (n = 321, n = 145) | 196 | 85
  Day 897 (n = 314, n = 136) | 184 | 78
  Day 981 (n = 302, n = 133) | 182 | 79
  Day 1,093 (n = 306, n = 135) | 194 | 77
  Day 1,177 (n = 266, n = 118) | 158 | 64
  Day 1,261 (n = 289, n = 130) | 176 | 76
  Day 1,345 (n = 141, n = 56) | 83 | 31
  Day 1,457 (n = 288, n = 127) | 193 | 75
  Day 1,625 (n = 274, n= 126) | 181 | 84
  Day 1,821 (n = 270, n = 123) | 165 | 75
  Day 1,989 (n = 121, n = 55) | 78 | 33
  Day 2,185 (n = 83, n = 37) | 46 | 22

55. Secondary Outcome: Number of ACR 70 Responders in the DB and OL Periods
Description: ACR 70 response requires a patient to have a 70% reduction in the number of swollen and tender joints, and a reduction of 70% in three of the following five parameters: physician global assessment of disease, patient global assessment of disease, patient assessment of pain, CRP or ESR, and degree of disability in HAQ score. A participant achieved a sustained ACR 70 response if the participant had ACR 70 observed for at least 2 consecutive study visits.
Time Frame: as for outcome 53
Population: as for outcome 53
Measure: Number; unit: Participants
Groups:
- ABA + MTX: Abatacept was dosed intravenously by weight at 10 mg/kg in the OL period under tiered dosing such that participants weighing < 60 kg received abatacept 500 mg; participants ≥ 60 kg and ≤ 100 kg received abatacept 750 mg; and particpants > 100 kg received abatacept 1 g. MTX was continued at the dose used in the DB period.
- MTX + Placebo: Participants that received MTX + placebo in the DB treatment period (Day 1 to Day 365) but are currently receiving treatment with ABA +MTX in the OL period. Abatacept was dosed intravenously by weight at 10 mg/kg in the OL period under tiered dosing such that participants weighing < 60 kg received abatacept 500 mg; particiapnts ≥ 60 kg and ≤ 100 kg received abatacept 750 mg; and particpants > 100 kg received abatacept 1 g. MTX was continued at the dose used in the DB period.
Arm/Group | ABA + MTX | MTX + Placebo
Number analyzed (Participants) | 376 | 160
Participants
  Day 15 (n = 371, n = 160) | 4 | 1
  Day 29 (n = 369, n=159) | 8 | 2
  Day 57 (n = 374, n = 159) | 27 | 6
  Day 85 (n = 370, n = 158) | 51 | 7
  Day 113 (n = 371, n = 159) | 56 | 10
  Day 141 (n = 371, n = 159) | 73 | 12
  Day 169 (n = 374, n = 159) | 83 | 14
  Day 225 (n = 369, n = 160) | 100 | 16
  Day 281 (n = 372, n = 160) | 104 | 20
  Day 365 (n = 374, n = 160) | 121 | 14
  Day 449 (n = 367, n = 157) | 122 | 33
  Day 533 (n = 350, n = 156) | 126 | 47
  Day 617 (n = 347, n = 154) | 116 | 51
  Day 729 (n = 340, n = 147) | 130 | 49
  Day 813 (n = 325, n = 146) | 117 | 42
  Day 897 (n = 314, n = 138) | 109 | 40
  Day 981 (n = 306, n = 134) | 116 | 39
  Day 1,093 (n = 309, n = 137) | 116 | 44
  Day 1,177 (n = 265, n = 122) | 94 | 40
  Day 1,261 (n = 289, n = 132) | 105 | 45
  Day 1,345 (n = 139, n = 57) | 52 | 18
  Day 1,457 (n = 288, n = 128) | 121 | 47
  Day 1,625 (n = 278, n= 125) | 115 | 50
  Day 1,821 (n = 270, n = 125) | 107 | 46
  Day 1,989 (n = 119, n = 54) | 50 | 22
  Day 2,185 (n = 83, n = 37) | 32 | 14

56. Secondary Outcome: Number of Participants Continuing in the OL Period With DAS-28 Remission or Low DAS-28 Activity Over Time
Description: The DAS 28 is a continuous measure evaluating extent of disease activity in RA, and is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, erythrocyte sedimentation rate (ESR) and participant assessment of disease activity measure on a visual analog scale (VAS) of 100 mm. The scale reports from 1 to 10, with increasing number indicating increasing extent of disease progression. Scores for disease activity are defined as high (> 5.1); low (≤ 3.2); remission (< 2.6).
Time Frame: Day 15, Day 29, Day 57, Day 85, Day 113, Day 141, Day 169, Day 225, Day 281, Day 365, Day 449, Day 533, Day 617, Day 729, Day 813, Day 897, Day 981, Day 1,083, Day 1,177, Day 1,261, Day 1,345, Day 1,497, Day 1,625, Day 1,821, Day 1,989, Day 2,185
Population: as for outcome 53
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Participants
  Remission Day 15 (n = 355, n = 152) | 1 | 0
  Low Disease Activity Day 15 (n=355, 152) | 5 | 1
  Remission Day 29 (n = 362, n =157) | 8 | 0
  Low Disease Activity Day 29 (n=362, 157) | 24 | 2
  Remission Day 57 (n = 367, n = 156) | 19 | 1
  Low Disease Activity Day 57 (n=367, 156) | 44 | 7
  Remission Day 85 (n = 366, n = 152) | 39 | 3
  Low Disease Activity Day 85 (n=366, 152) | 76 | 16
  Remission Day 113 (n = 367, n = 159) | 39 | 9
  Low Disease Activity Day 113 (n=367, 159) | 89 | 20
  Remission Day 141 (n = 366, n = 158) | 57 | 7
  Low Disease Activity Day 141 (n=366, 158) | 104 | 20
  Remission Day 169 (n = 371, n = 159) | 63 | 6
  Low Disease Activity Day 169 (n=371, 159) | 117 | 19
  Remission Day 225 (n = 366, n = 158) | 75 | 9
  Low Disease Activity Day 225 (n=366, 158) | 147 | 21
  Remission Day 281 (n = 364, n = 159) | 89 | 14
  Low Disease Activity Day 281 (n=364, 159) | 150 | 33
  Remission Day 365 (n = 370, n = 159) | 94 | 4
  Low Disease Activity Day 365 (n=370, 159) | 163 | 19
  Remission Day 449 (n = 357, n = 150) | 100 | 32
  Low Disease Activity Day 449 (n=357, 150) | 162 | 55
  Remission Day 533 (n = 343, n = 150) | 101 | 42
  Low Disease Activity Day 553 (n=343, 150) | 158 | 61
  Remission Day 617 (n = 334, n = 153) | 100 | 46
  Low Disease Activity Day 617 (n=334, 153) | 159 | 74
  Remission Day 729 (n = 337, n = 148) | 97 | 45
  Low Disease Activity Day 729 (n=337, 148) | 175 | 77
  Remission Day 813 (n = 317, n = 143) | 97 | 46
  Low Disease Activity Day 813 (n=317, 143) | 160 | 72
  Remission Day 897 (n = 303, n = 135) | 91 | 48
  Low Disease Activity Day 897 (n=303, 135) | 152 | 70
  Remission Day 981 (n = 297, n = 133) | 102 | 46
  Low Disease Activity Day 981 (n=297, 133) | 168 | 72
  Remission Day 1,093 (n = 300, n = 129) | 112 | 42
  Low Disease Activity Day 1,093 (n=300, 129) | 160 | 77
  Remission Day 1,177 (n = 158, n = 71) | 55 | 27
  Low Disease Activity Day 1,177 (n=158, 71) | 84 | 42
  Remission Day 1,261 (n = 267, n = 119) | 91 | 50
  Low Disease Activity Day 1,261 (n=267, 119) | 146 | 70
  Remission Day 1,457 (n = 284, n = 129) | 111 | 51
  Low Disease Activity Day 1,457 (n=284, 129) | 161 | 79
  Remission Day 1,625 (n = 272, n= 124) | 96 | 47
  Low Disease Activity Day 1,625 (n=272, 124) | 145 | 71
  Remission Day 1,821 (n = 270, n = 124) | 89 | 47
  Low Disease Activity Day 1,821 (n=270, 124) | 147 | 73
  Remission Day 1,989 (n=118, 54) | 43 | 21
  Low Disease Activity Day 1,989 (n=118, 54) | 65 | 31
  Remission Day 2,185 (n=82, 37) | 25 | 18
  Low Disease Activity Day 2,185 (n=82, 37) | 41 | 22

57. Secondary Outcome: Mean BL DAS-28 CRP Over Time for Participants Continuing in the OL Period
Description: Time-matched BL (Day 0) values and post-BL vales were presented for each post-BL visit and represent only that cohort of participants with measurements available at that post-BL assessment.
Time Frame: BL(Day 0), Day 15, Day 29,Day 57,Day 85, Day 113, Day 141, Day 169, Day 225, Day 281, Day 365, Day 449, Day 533, Day 617, Day 729, Day 813, Day 897, Day 981, Day 1,083, Day 1,177, Day 1,261, Day 1,345, Day 1,497, Day 1,625, Day 1,821, Day 1,989, Day 2,185
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: mg / mL
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
mg / mL
  BL (Day 0) for Day 15 Cohort (n=352, 150) | 6.36 (0.81) | 6.32 (0.81)
  BL (Day 0) for Day 29 Cohort (n=357, 154) | 6.36 (0.81) | 6.35 (0.81)
  BL (Day 0) for Day 57 Cohort (n=362, 153) | 6.36 (0.81) | 6.35 (0.79)
  BL (Day 0) for Day 85 Cohort (n=362, 149) | 6.35 (0.81) | 6.33 (0.81)
  BL (Day 0) for Day 113 Cohort (n=362, 149) | 6.35 (0.81) | 6.34 (0.81)
  BL (Day 0) for Day 141 Cohort (n=361, 155) | 6.34 (0.80) | 6.33 (0.82)
  BL (Day 0) for Day 169 Cohort (n=366, 156) | 6.35 (0.80) | 6.34 (0.80)
  BL (Day 0) for Day 225 Cohort (n=361, 155) | 6.35 (0.81) | 6.33 (0.81)
  BL (Day 0) for Day 281 Cohort (n=359, 156) | 6.35 (0.81) | 6.33 (0.81)
  BL (Day 0) for Day 365 Cohort (n=365, 156) | 6.36 (0.81) | 6.33 (0.81)
  BL (Day 0) for Day 449 Cohort (n=352, 147) | 6.37 (0.81) | 6.34 (0.81)
  BL (Day 0) for Day 533 Cohort (n=338, 147) | 6.38 (0.81) | 6.35 (0.80)
  BL (Day 0) for Day 617 Cohort (n=329, 150) | 6.37 (0.80) | 6.35 (0.81)
  BL (Day 0) for Day 729 Cohort (n=333, 145) | 6.37 (0.81) | 6.36 (0.83)
  BL (Day 0) for Day 813 Cohort (n=313, 140) | 6.39 (0.82) | 6.37 (0.82)
  BL (Day 0) for Day 897 Cohort (n=301, 133) | 6.38 (0.83) | 6.37 (0.83)
  BL (Day 0) for Day 981 Cohort (n=294, 131) | 6.39 (0.82) | 6.37 (0.83)
  BL (Day 0) for Day 1,093 Cohort (n=296, 127) | 6.37 (0.83) | 6.37 (0.84)
  BL (Day 0) for Day 1,177 Cohort (n=156, 70) | 6.43 (0.85) | 6.38 (0.86)
  BL (Day 0) for Day 1,261 Cohort (n=267, 117) | 6.39 (0.80) | 6.34 (0.85)
  BL (Day 0) for Day 1,457 Cohort (n=281, 126) | 6.40 (0.82) | 6.35 (0.81)
  BL (Day 0) for Day 1,625 Cohort (n=269, 121) | 6.39 (0.81) | 6.40 (0.77)
  BL (Day 0) for Day 1,821 Cohort (n=267, 122) | 6.39 (0.81) | 6.33 (0.76)
  BL (Day 0) for Day 1,989 Cohort (n=118, 53) | 6.53 (0.77) | 6.49 (0.75)
  BL (Day 0) for Day 2,185 Cohort (n=82, 36) | 6.41 (0.77) | 6.38 (0.82)

58. Secondary Outcome: Mean Change From BL in DAS-28 CRP Over Time for Participants Continuing in the OL Period
Description: Change from baseline in participant were calculated at all study visits in the DB and OL periods.
Time Frame: BL(Day 0),Day 15,Day 29, Day 57, Day 85, Day 113, Day 141, Day 169, Day 225, Day 281, Day 365, Day 449, Day 533, Day 617, Day 729, Day 813, Day 897, Day 981, Day 1,083, Day 1,177, Day 1,261, Day 1,345, Day 1,497, Day 1,625, Day 1,821, Day 1,989, Day 2,185
Population: as for outcome 53
Measure: Mean (Standard Error); unit: mg / mL
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
mg / mL
  Day 15 (n=352, 150) | -0.83 (0.04) | -0.47 (0.06)
  Day 29 (n=357, 154) | -1.27 (0.05) | -0.87 (0.08)
  Day 57 (n=362, 153) | -1.80 (0.06) | -1.17 (0.09)
  Day 85 (n=362, 149) | -2.12 (0.06) | -1.37 (0.10)
  Day 113 (n=362, 149) | -2.30 (0.06) | -1.47 (0.11)
  Day 141 (n=361, 155) | -2.46 (0.07) | -1.52 (0.11)
  Day 169 (n=366, 156) | -2.48 (0.07) | -1.57 (0.11)
  Day 225 (n=361, 155) | -2.72 (0.07) | -1.70 (0.11)
  Day 281 (n=359, 156) | -2.81 (0.07) | -1.87 (0.10)
  Day 365 (n=365, 156) | -2.83 (0.07) | -1.68 (0.10)
  Day 449 (n=352, 147) | -2.91 (0.07) | -2.68 (0.10)
  Day 533 (n=338, 147) | -3.01 (0.07) | -2.79 (0.11)
  Day 617 (n=329, 150) | -3.00 (0.07) | -2.92 (0.11)
  Day 729 (n=333, 145) | -3.10 (0.07) | -3.02 (0.11)
  Day 813 (n=313, 140) | -3.09 (0.07) | -3.05 (0.12)
  Day 897 (n=301, 133) | -3.06 (0.07) | -3.11 (0.11)
  Day 981 (n=294, 131) | -3.21 (0.08) | -3.14 (0.12)
  Day 1,093 (n=296, 127) | -3.21 (0.08) | -3.15 (0.12)
  Day 1,177 (n=156, 70) | -3.27 (0.11) | -3.21 (0.16)
  Day 1,261 (n=267, 117) | -3.22 (0.08) | -3.15 (0.13)
  Day 1,457 (n=281, 126) | -3.29 (0.08) | -3.23 (0.11)
  Day 1,625 (n=269, 121) | -3.23 (0.08) | -3.34 (0.11)
  Day 1,821 (n=267, 122) | -3.14 (0.08) | -3.26 (0.12)
  Day 1,989 (n=118, 53) | -3.39 (0.12) | -3.31 (0.19)
  Day 2,185 (n=82, 36) | -3.04 (0.16) | -3.30 (0.23)

59. Secondary Outcome: Mean BL DAS-28 ESR Over Time in the OL Period
Description: Mean baseline values are reported for each cohort at each time point. Time-matched BL(Day 0) values and post-BL vales were presented for each post-BL visit and represent only that cohort of participants with measurements available at that post-BL assessment.
Time Frame: BL (Day 0), Day 365, Day 449, Day 533, Day 617, Day 729, Day 813, Day 897, Day 981, Day 1,083, Day 1,177, Day 1,261, Day 1,345, Day 1,497, Day 1,625, Day 1,821, Day 1,989, Day 2,185
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: IU / mL
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
IU / mL
  BL (Day 0) for Day 365 Cohort (n=352, 148) | 6.82 (0.85) | 6.88 (0.85)
  BL (Day 0) for Day 449 Cohort (n=345, 145) | 6.82 (0.86) | 6.89 (0.85)
  BL (Day 0) for Day 533 Cohort (n=332, 146) | 6.83 (0.86) | 6.88 (0.86)
  BL (Day 0) for Day 617 Cohort (n=325, 148) | 6.85 (0.86) | 6.86 (0.86)
  BL (Day 0) for Day 729 Cohort (n=315, 139) | 6.82 (0.88) | 6.87 (0.88)
  BL (Day 0) for Day 813 Cohort (n=303, 134) | 6.82 (0.87) | 6.90 (0.88)
  BL (Day 0) for Day 897 Cohort (n=296, 128) | 6.83 (0.88) | 6.85 (0.90)
  BL (Day 0) for Day 981 Cohort (n=282, 119) | 6.82 (0.87) | 6.88 (0.88)
  BL (Day 0) for Day 1,093 Cohort (n=287, 130) | 6.83 (0.88) | 6.87 (0.89)
  BL (Day 0) for Day 1,177 Cohort (n=241, 110) | 6.86 (0.87) | 6.89 (0.92)
  BL (Day 0) for Day 1,261 Cohort (n=271, 121) | 6.82 (0.87) | 6.86 (0.89)
  BL (Day 0) for Day 1,457 Cohort (n=269, 117) | 6.87 (0.85) | 6.88 (0.87)
  BL (Day 0) for Day 1,625 Cohort (n=260, 118) | 6.86 (0.85) | 6.86 (0.86)
  BL (Day 0) for Day 1,821 Cohort (n=259, 114) | 6.85 (0.86) | 6.87 (0.84)
  BL (Day 0) for Day 1,989 Cohort (n=108, 47) | 6.95 (0.83) | 7.04 (0.85)
  BL (Day 0) for Day 2,185 Cohort (n=76, 31) | 6.90 (0.82) | 6.97 (0.92)

60. Secondary Outcome: Mean Change From BL in DAS-28 ESR Over Time in the OL Period
Description: Change from baseline in participant serum values of ESR were calculated at all study visits in the OL period.
Time Frame: as for outcome 59
Population: as for outcome 53
Measure: Mean (Standard Error); unit: IU / mL
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
IU / mL
  Day 365 (n=352, 148) | -2.96 (0.07) | -1.76 (0.11)
  Day 449 (n=345, 145) | -3.04 (0.08) | -2.87 (0.11)
  Day 533 (n=332, 146) | -3.14 (0.08) | -2.95 (0.12)
  Day 617 (n=325, 148) | -3.17 (0.08) | -3.02 (0.11)
  Day 729 (n=315, 139) | -3.27 (0.07) | -3.20 (0.12)
  Day 813 (n=303, 134) | -3.13 (0.08) | -3.18 (0.12)
  Day 897 (n=296, 128) | -3.11 (0.08) | -3.10 (0.12)
  Day 981 (n=282, 119) | -3.26 (0.09) | -3.19 (0.14)
  Day 1,093 (n=287, 130) | -3.23 (0.08) | -3.22 (0.13)
  Day 1,177 (n=241, 110) | -3.33 (0.09) | -3.29 (0.15)
  Day 1,261 (n=271, 121) | -3.25 (0.08) | -3.18 (0.14)
  Day 1,457 (n=269, 117) | -3.32 (0.08) | -3.23 (0.12)
  Day 1,625 (n=260, 118) | -3.30 (0.09) | -3.27 (0.12)
  Day 1,821 (n=259, 114) | -3.22 (0.09) | -3.34 (0.12)
  Day 1,989 (n=108, 47) | -3.41 (0.13) | -3.42 (0.23)
  Day 2,185 (n=76, 31) | -3.25 (0.17) | -3.66 (0.33)

61. Primary Outcome: Mean BL Immunoglobulins Over Time in the OL Period
Description: Mean baseline values are those that are reported for each cohort at each time point on Day 365, Day 729, and Day 1,093.
Time Frame: BL (Day 0), Day 365, Day 729, Day 1,093
Population: All treated participants in the OL period (treatment groups represent treatment received in the double-blind period).
Measure: Mean (Standard Deviation); unit: mg / mL
Arm/Group | ABA + MTX DB | Placebo + MTX DB
Number analyzed (Participants) | 378 | 161
mg / mL
  Immunoglobulin A (IgA) Day 365 | 327.0 (135.2) | 319.2 (145.1)
  Immunoglobulin G (IgG) Day 365 | 1278 (412.4) | 1317 (425.4)
  Immunoglobulin M (IgM) Day 365 | 145.1 (86.72) | 154.3 (85.53)
  IgA Day 729 | 328.0 (133.8) | 317.0 (145.0)
  IgG Day 729 | 1280 (410.4) | 1315 (425.3)
  IgM Day 729 | 146.2 (87.34) | 153.1 (85.80)
  IgA Day 1,093 | 321.8 (133.4) | 318.5 (145.7)
  IgG Day 1,093 | 1273 (392.3) | 1319 (436.8)
  IgM Day 1,093 | 148.6 (91.01) | 153.5 (88.82)

62. Primary Outcome: Mean Change From BL in Immunoglobulins in the OL Period
Time Frame: BL (Day 0), Day 365, Day 729, Day 1,093
Population: All treated participants in the OL period (treatment groups represent treatment received in the double-blind period).
Measure: Mean (Standard Error); unit: mg / mL
Arm/Group | ABA + MTX DB | Placebo + MTX DB
Number analyzed (Participants) | 378 | 161
mg / mL
  IgA Day 365 | -47.8 (3.16) | -8.30 (6.41)
  IgG Day 365 | -212 (12.77) | -52.7 (18.96)
  IgM Day 365 | -5.05 (1.98) | 6.95 (9.73)
  IgA Day 729 | -38.6 (4.24) | -26.6 (9.95)
  IgG Day 729 | -215 (14.10) | -206 (21.86)
  IgM Day 729 | 8.04 (3.96) | 6.49 (5.76)
  IgA Day 1,093 | -46.8 (4.76) | -37.9 (9.66)
  IgG Day 1,093 | -236 (15.94) | -245 (25.44)
  IgM Day 1,093 | 4.38 (3.19) | 6.01 (5.01)

63. Primary Outcome: Participants With Immunogenicity to Abatacept in the Cumulative DB + OL Period
Description: Participants with titers to abatacept in the DB and OL periods. Serum samples from abatacept-treated adult participants with active Rheumatoid Arthritis (RA) were screened for the presence of drug-specific antibodies using two validated direct-format enzyme-linked immunosorbent assays (ELISAs) to determine the presence of antibodies to abatacept and or CTLA4-T.
Time Frame: Day 1 to Day 1,821
Population: Participants with serum samples available for evaluation of titers to abatacept.
Measure: Number; unit: Participants
Groups:
- ABA + MTX Cumulative DB + OL Periods: Abatacept was dosed intravenously by weight at 10 mg/kg in the DB and OL periods under tiered dosing such that participants weighing < 60 kg received abatacept 500 mg; particiapnts ≥ 60 kg and ≤ 100 kg received abatacept 750 mg; and particpants > 100 kg received abatacept 1 g. MTX was continued at the dose used in the DB period.
Arm/Group | ABA + MTX Cumulative DB + OL Periods
Number analyzed (Participants) | 586
Participants | 56

64. Secondary Outcome: Number of Participants Achieving HAQ Response Over Time for Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: as for outcome 53
Population: as for outcome 53
Measure: Number; unit: Participants
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Participants
  Day 15 (n = 367, n = 160) | 115 | 46
  Day 29 (n = 365, n = 159) | 148 | 57
  Day 57 (n = 372, n = 157) | 199 | 73
  Day 85 (n = 366, n = 156) | 228 | 76
  Day 113 (n = 369, n = 159) | 239 | 85
  Day 141 (n = 370, n = 159) | 238 | 85
  Day 169 (n = 373, n = 159) | 247 | 89
  Day 225 (n = 368, n = 159) | 252 | 87
  Day 281 (n = 368, n = 160) | 249 | 89
  Day 365 (n = 369, n = 160) | 265 | 86
  Day 449 (n = 366, n = 157) | 268 | 114
  Day 533 (n = 354, n = 157) | 259 | 109
  Day 617 (n = 348, n = 154) | 257 | 107
  Day 729 (n = 337, n = 148) | 248 | 100
  Day 813 (n = 325, n= 146) | 237 | 98
  Day 897 (n = 318, n = 140) | 232 | 99
  Day 981 (n = 312, n = 137) | 227 | 91
  Day 1,093 (n = 308, n = 137) | 225 | 94
  Day 1,177 (n = 274, n = 124) | 205 | 85
  Day 1,261 (n = 292, n = 134) | 214 | 88
  Day 1,345 (n = 152, n = 62) | 106 | 40
  Day 1,457 (n = 289, n = 129) | 218 | 94
  Day 1,625 (n =280, n = 126) | 210 | 92
  Day 1,821 (n = 271, n = 125) | 201 | 90
  Day 1,989 (n = 119, n = 55) | 90 | 35
  Day 2,185 (n = 85, n = 38) | 63 | 26

65. Secondary Outcome: BL and Mean Change From BL in Radiographic Erosion, Joint Space Narrowing (JSN), and Total Scores (TS) in the OL Period
Description: Change from baseline in the Genant-modified Sharp erosion score, JSN, TS were evaluated for all participants at the end of the OL period. The total Genant-modified Sharp score (TS) ranges from 0 (no radiographic damage) to 290 (worst possible radiographic damage) and is the sum of the erosion score (range 0-145) and the joint space narrowing score (range 0-145).Higher scores indicated more damage. Time-matched BL (Day 0) values and post-BL vales were presented for each post-BL visit and represent only that cohort of participants with measurements available at that post-BL assessment.
Time Frame: BL (Day 0), Day 365, Day 729, Day 1,093, Day 1,457, Day 1,821
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  BL (Day 0) for Day 365 Cohort Erosion (n=291, 131) | 17.65 (15.81) | 18.69 (17.12)
  Day 365 Erosion Change From BL (n=291, 131) | 0.42 (1.20) | 0.84 (1.93)
  BL (Day 0) for Day 365 Cohort JSN (n=291, 131) | 10.83 (14.02) | 12.02 (14.53)
  Day 365 JSN Change From BL(n=291, 131) | 0.38 (1.05) | 0.64 (1.67)
  BL (Day 0) for Day 365 Cohort TS (n=291, 131) | 28.48 (29.01) | 30.71 (30.84)
  Day 365 TS Change From BL (n=291, 131) | 0.80 (1.99) | 1.48 (3.35)
  BL (Day 0) for Day 729 Cohort Erosion (n=290, 130) | 17.40 (15.41) | 18.88 (17.18)
  Day 729 Erosion Change From BL (n=291, 131) | 0.59 (1.67) | 1.14 (2.74)
  BL (Day 0) for Day 729 Cohort JSN (n=291, 131) | 10.65 (13.80) | 12.21 (14.56)
  Day 729 JSN Change From BL(n=291, 131) | 0.55 (1.40) | 1.05 (2.79)
  BL (Day 0) for Day 729 Cohort TS (n=291, 131) | 28.05 (28.41) | 31.09 (30.93)
  Day 729 TS Change From BL(n=291, 131) | 1.14 (2.69) | 2.19 (5.22)
  BL (Day 0) for Day 1093 Cohort Erosion (n=293,130) | 17.66 (15.78) | 18.69 (17.12)
  Day 1093 Erosion Change From BL (n=293, 130) | 0.92 (2.60) | 1.48 (3.65)
  BL (Day 0) for Day 1093 Cohort JSN (n=293, 130) | 10.84 (13.97) | 12.02 (14.53)
  Day 1093 JSN Change From BL (n=293, 130) | 0.73 (2.02) | 1.31 (3.40)
  BL (Day 0) for Day 1093 Cohort TS (n=293, 130) | 28.50 (28.94) | 30.71 (30.84)
  Day 1093 Total Score Change From BL (n=293, 130) | 1.65 (4.20) | 2.79 (6.60)
  BL (Day 0) for Day 1457 Cohort Erosion (n=290,128) | 17.46 (15.46) | 18.94 (17.30)
  Day 1457 Erosion Change From BL (n=290, 128) | 1.16 (3.14) | 1.76 (4.30)
  BL (Day 0) for Day 1457 Cohort JSN (n=290, 128) | 10.66 (13.71) | 12.12 (14.64)
  Day 1457 JSN Change From BL (n=290, 128) | 0.85 (2.30) | 1.51 (3.73)
  BL (Day 0) for Day 1457 Cohort TS (n=290, 128) | 28.12 (28.35) | 31.06 (31.16)
  Day 1457 TS Change From BL (n=290, 128) | 2.01 (5.00) | 3.27 (7.55)
  BL (Day 0) for Day 1821 Cohort Erosion (n=233,114) | 17.62 (15.62) | 18.93 (17.37)
  Day 1821 Erosion Change From BL (n=233, 114) | 1.12 (2.99) | 2.05 (4.88)
  BL (Day 0) for Day 1821 Cohort JSN (n=233, 114) | 10.77 (13.73) | 12.01 (14.47)
  Day 1821 JSN Change From BL (n=233, 114) | 0.90 (2.54) | 1.73 (4.11)
  BL (Day 0) for Day 1821 Cohort TS (n=233, 114) | 28.39 (28.50) | 30.94 (30.99)
  Day 1821 TS Change From BL (n=233, 114) | 2.02 (4.93) | 3.78 (8.46)

66. Secondary Outcome: Mean BL Physical Component Summary of the SF-36 by Visit in the OL Period
Description: as for outcome 19
Time Frame: BL (Day 0), Day 365, Day 449, Day 533, Day 617, Day 729, Day 813, Day 897, Day 981, Day 1,093, Day 1,177, Day 1,261, Day 1,345, Day 14,57, Day 1,625, Day 1,821, Day 1,989, Day 2,185
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- ABA + MTX DB: Abatacept was dosed intravenously by weight at 10 mg/kg in the OL period under tiered dosing such that participants weighing < 60 kg received abatacept 500 mg; participants ≥ 60 kg and ≤ 100 kg received abatacept 750 mg; and participants > 100 kg received abatacept 1 g. MTX was continued at the dose used in the OL period.
- MTX + Placebo DB: Participants that received MTX + placebo in the DB treatment period (Day 1 to Day 365) but are currently receiving treatment with ABA + MTX in the OL period. Abatacept was dosed intravenously by weight at 10 mg/kg in the OL period under tiered dosing such that participants weighing < 60 kg received abatacept 500 mg; participants ≥ 60 kg and ≤ 100 kg received abatacept 750 mg; and participants > 100 kg received abatacept 1 g. MTX was continued at the dose used in the DB period.
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  BL (Day 0) for Day 365 Cohort (n=370, 157) | 30.69 (6.84) | 30.94 (7.32)
  BL (Day 0) for Day 449 Cohort (n=362, 156) | 30.55 (6.78) | 30.95 (7.34)
  BL (Day 0) for Day 533 Cohort (n=355, 155) | 30.64 (6.79) | 30.86 (7.34)
  BL (Day 0) for Day 617 Cohort (n=348, 153) | 30.70 (6.81) | 30.88 (7.37)
  BL (Day 0) for Day 729 Cohort (n=338, 146) | 30.75 (6.78) | 30.88 (7.25)
  BL (Day 0) for Day 813 Cohort (n=323, 145) | 30.58 (6.66) | 31.00 (7.29)
  BL (Day 0) for Day 897 Cohort (n=320, 139) | 30.52 (6.69) | 30.87 (7.41)
  BL (Day 0) for Day 981 Cohort (n=312, 136) | 30.49 (6.64) | 30.98 (7.46)
  BL (Day 0) for Day 1,093 Cohort (n=308, 137) | 30.51 (6.67) | 30.93 (7.45)
  BL (Day 0) for Day 1,177 Cohort (n=273, 124) | 30.58 (6.78) | 30.87 (7.19)
  BL (Day 0) for Day 1,261 Cohort (n=289, 133) | 30.64 (6.86) | 31.02 (7.47)
  BL (Day 0) for Day 1,345 Cohort (n=146, 60) | 30.40 (6.32) | 29.37 (7.07)
  BL (Day 0) for Day 1,457 Cohort (n=288, 128) | 30.51 (6.76) | 31.23 (7.46)
  BL (Day 0) for Day 1,625 Cohort (n=278, 125) | 30.70 (6.78) | 30.90 (7.30)
  BL (Day 0) for Day 1,821 Cohort (n=273, 124) | 30.54 (6.81) | 31.27 (7.42)
  BL (Day 0) for Day 1,989 Cohort (n=118, 54) | 29.80 (6.72) | 30.66 (7.61)
  BL (Day 0) for Day 2,185 Cohort (n=84, 38) | 28.80 (5.77) | 29.74 (5.72)

67. Secondary Outcome: Mean Change From BL by Visit in the Physical Component Summary of the SF-36 in the OL Period
Description: as for outcome 20
Time Frame: as for outcome 66
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  Day 365 (n=370, 157) | 9.70 (0.50) | 6.61 (0.74)
  Day 449 (n=362, 156) | 10.51 (0.50) | 9.91 (0.78)
  Day 533 (n=355, 155) | 10.27 (0.51) | 10.53 (0.86)
  Day 617 (n=348, 153) | 10.46 (0.52) | 10.74 (0.85)
  Day 729 (n=338, 146) | 10.71 (0.53) | 10.36 (0.84)
  Day 813 (n=323, 145) | 10.79 (0.55) | 10.41 (0.84)
  Day 897 (n=320, 139) | 10.30 (0.53) | 9.87 (0.85)
  Day 981 (n=312, 136) | 11.05 (0.58) | 10.78 (0.87)
  Day 1,093 (n=308, 137) | 10.83 (0.55) | 11.07 (0.94)
  Day 1,177 (n=273, 124) | 11.02 (0.61) | 11.20 (1.01)
  Day 1,261 (n=289, 133) | 10.40 (0.60) | 11.34 (0.94)
  Day 1,345 (n=146, 60) | 9.81 (0.87) | 10.81 (1.55)
  Day 1,457 (n=288, 128) | 11.12 (0.58) | 10.68 (0.97)
  Day 1,625 (n=278, 125) | 10.76 (0.61) | 11.05 (0.90)
  Day 1,821 (n=273, 124) | 10.81 (0.63) | 10.09 (0.91)
  Day 1,989 (n=118, 54) | 11.69 (0.93) | 9.65 (1.47)
  Day 2,185 (n=84, 38) | 9.69 (0.99) | 11.39 (1.71)

68. Secondary Outcome: Mean BL Mental Component Summary of the SF-36 by Visit in the OL Period
Description: The SF-36 covers 8 health dimensions including 4 physical subscales (physical function, role-physical, bodily pain, and general health) and 4 mental subscales (vitality, social function, role-emotional, and mental health). The scores range from a minimum of 0 to a maximum of 100, with a higher score indicating better quality of life. Improvements of > 3 points were considered clinically meaningful.Time-matched BL(Day 0) values and post-BL vales were presented for each post-BL visit and represent only that cohort of participants with measurements available at that post-BL assessment.
Time Frame: BL (Day 0), Day 365, Day 449, Day 533, Day 617, Day 729, Day 813, Day 897, Day 981, Day 1,093, Day 1,177, Day 1,261, Day 1,345, Day 1,457, Day 1,625, Day 1,821, Day 1,989, Day 2,185
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  BL (Day 0) for Day 365 Cohort (n=370, 157) | 41.40 (11.35) | 40.56 (11.18)
  BL (Day 0) for Day 449 Cohort (n=362, 156) | 41.20 (11.29) | 40.47 (11.11)
  BL (Day 0) for Day 533 Cohort (n=355, 156) | 41.28 (11.20) | 40.53 (11.25)
  BL (Day 0) for Day 617 Cohort (n=348, 153) | 41.23 (11.28) | 40.67 (11.26)
  BL (Day 0) for Day 729 Cohort (n=338, 146) | 41.21 (11.28) | 40.24 (11.11)
  BL (Day 0) for Day 813 Cohort (n=323, 145) | 41.23 (11.34) | 40.19 (11.20)
  BL (Day 0) for Day 897 Cohort (n=320, 139) | 41.36 (11.41) | 40.28 (11.33)
  BL (Day 0) for Day 981 Cohort (n=312, 136) | 41.40 (11.39) | 40.32 (11.45)
  BL (Day 0) for Day 1,093 Cohort (n=308, 137) | 41.40 (11.25) | 40.33 (11.41)
  BL (Day 0) for Day 1,177 Cohort (n=273, 124) | 41.28 (11.47) | 40.19 (11.06)
  BL (Day 0) for Day 1,261 Cohort (n=289, 133) | 41.29 (11.45) | 40.26 (11.50)
  BL (Day 0) for Day 1,345 Cohort (n=146, 60) | 42.11 (11.81) | 39.99 (10.83)
  BL (Day 0) for Day 1,457 Cohort (n=288, 128) | 41.35 (11.45) | 40.06 (11.35)
  BL (Day 0) for Day 1,625 Cohort (n=278, 125) | 41.25 (11.60) | 40.16 (11.44)
  BL (Day 0) for Day 1,821 Cohort (n=273, 124) | 41.39 (11.60) | 40.03 (11.23)
  BL (Day 0) for Day 1,989 Cohort (n=118, 54) | 41.73 (11.58) | 39.61 (9.98)
  BL (Day 0) for Day 2,185 Cohort (n=84, 38) | 42.00 (11.97) | 37.55 (9.95)

69. Secondary Outcome: Mean Change From BL by Visit in the Mental Component Summary of the SF-36 in the OL Period
Description: as for outcome 20
Time Frame: as for outcome 68
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  Day 365 (n=370, 157) | 7.29 (0.60) | 6.41 (0.85)
  Day 449 (n=362, 156) | 6.84 (0.63) | 7.73 (0.97)
  Day 533 (n=355, 156) | 7.30 (0.62) | 7.20 (0.96)
  Day 617 (n=348, 153) | 7.15 (0.64) | 6.88 (0.94)
  Day 729 (n=338, 146) | 7.31 (0.61) | 8.07 (1.01)
  Day 813 (n=323, 145) | 6.98 (0.67) | 7.15 (1.01)
  Day 897 (n=320, 139) | 7.26 (0.69) | 8.54 (1.02)
  Day 981 (n=312, 136) | 6.82 (0.69) | 7.76 (1.02)
  Day 1,093 (n=308, 137) | 7.79 (0.69) | 6.09 (1.04)
  Day 1,177 (n=273, 124) | 6.93 (0.73) | 7.65 (1.09)
  Day 1,261 (n=289, 133) | 7.33 (0.74) | 7.04 (1.05)
  Day 1,345 (n=146, 60) | 6.37 (1.00) | 7.42 (1.43)
  Day 1,457 (n=288, 128) | 6.82 (0.74) | 7.19 (1.12)
  Day 1,625 (n=278, 125) | 6.60 (0.74) | 6.99 (1.15)
  Day 1,821 (n=273, 124) | 6.75 (0.75) | 9.08 (1.10)
  Day 1,989 (n=118, 54) | 5.53 (1.14) | 8.74 (1.60)
  Day 2,185 (n=84, 38) | 5.28 (1.28) | 9.91 (1.72)

70. Secondary Outcome: Mean BL Physical Function Component of the SF-36 by Visit in the OL Period
Description: as for outcome 19
Time Frame: as for outcome 68
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  BL (Day 0) for Day 365 Cohort (n=373, 160) | 28.79 (9.12) | 28.09 (8.88)
  BL (Day 0) for Day 449 Cohort (n=367, 157) | 28.62 (9.06) | 28.07 (8.95)
  BL (Day 0) for Day 533 Cohort (n=355, 157) | 28.63 (9.13) | 28.05 (8.91)
  BL (Day 0) for Day 617 Cohort (n=348, 155) | 28.71 (9.13) | 28.02 (8.91)
  BL (Day 0) for Day 729 Cohort(n=338, 148) | 28.68 (9.20) | 28.01 (8.93)
  BL (Day 0) for Day 813 Cohort (n=324, 147) | 28.41 (8.97) | 28.01 (9.01)
  BL (Day 0) for Day 897 Cohort (n=320, 140) | 28.36 (8.99) | 27.93 (9.11)
  BL (Day 0) for Day 981 Cohort (n=312, 137) | 28.43 (9.01) | 28.10 (9.15)
  BL (Day 0) for Day 1,093 Cohort (n=310, 138) | 28.43 (8.98) | 28.10 (9.11)
  BL (Day 0) for Day 1,177 Cohort (n=275, 125) | 28.70 (8.95) | 27.91 (8.85)
  BL (Day 0) for Day 1,261 Cohort (n=292, 135) | 28.62 (9.12) | 28.17 (9.13)
  BL (Day 0) for Day 1,345 Cohort (n=147, 61) | 28.70 (8.97) | 26.49 (8.34)
  BL (Day 0) for Day 1,457 Cohort (n=290, 129) | 28.35 (9.11) | 28.24 (9.03)
  BL (Day 0) for Day 1,625 Cohort (n=279, 126) | 28.68 (9.10) | 27.98 (8.87)
  BL (Day 0) for Day 1,821 Cohort (n=273, 125) | 28.50 (9.07) | 28.50 (9.03)
  BL (Day 0) for Day 1,989 Cohort (n=118, 55) | 27.78 (8.86) | 27.75 (9.35)
  BL (Day 0) for Day 2,185 Cohort (n=85, 38) | 26.94 (7.79) | 26.25 (7.45)

71. Primary Outcome: Number of Participants Experiencing Clinically Significant Changes in Vital Signs in the OL Period
Description: Vital signs included body temperature, heart rate, and seated blood pressure. Clinically significant changes were defined as those that were not within the normal range for the participant.
Time Frame: Day 365 to Day 1,821. All changes in participant vital signs were monitored on each day of study drug administration prior to dosing and 60 minutes after dosing.
Population: All treated participants entering the OL period.
Measure: Number; unit: Participants
Arm/Group | ABA + MTX OL
Number analyzed (Participants) | 529
Participants
  Body Temperature | 0
  Heart Rate | 0
  Blood Pressure | 0

72. Primary Outcome: Number of Participants Experiencing AEs of Special Interest in the OL Period
Description: AEs were defined as any new untoward medical occurrence or worsening of a pre- existing medical condition which does not necessarily have a causal relationship with this treatment. AEs of special interest have been identified to be those which may be associated with the use of immunomodulatory agents or infusion of therapeutic proteins. Acute infusional AEs were defined as those that occurred within 1 hour after the start of the infusion.
Time Frame: Day 365 to Day 2,185
Population: All treated participants in the OL period.
Measure: Number; unit: Participants
Arm/Group | ABA + MTX OL
Number analyzed (Participants) | 529
Participants
  Infections/Infestations | 452
  Neoplasms | 71
  Autoimmune Disorders | 52
  Acute Infusional AEs | 30
  Peri-Infusional AEs | 86

73. Primary Outcome: Mean BL Hematocrit in the OL Period
Description: Mean baseline values are those that are reported for each cohort at each time point on Day 365 to Day 2,185.
Time Frame: Baseline (Day 0), Day 365, Day 729, Day 1,093, Day 1,457, Day 1,821, Day 1,905, Day 1,989, Day 2,073, Day 2,185
Population: All treated participants in the OL period (treatment groups represent treatment received in the double-blind period). N = number of participants analyzed and n = the number of participants with measurements for that time point.
Measure: Mean (Standard Deviation); unit: Percentage of Red Blood Cells
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 378 | 161
Percentage of Red Blood Cells
  Day 365 (n=365, 157) | 38.79 (4.60) | 39.38 (4.32)
  Day 729 (n=328, 143) | 38.72 (4.52) | 39.39 (4.19)
  Day 1,093 (n=312, 138) | 38.69 (4.57) | 39.46 (4.33)
  Day 1,457 (n=292, 130) | 38.59 (4.48) | 39.40 (4.27)
  Day 1,821 (n=262,124) | 38.70 (4.44) | 39.48 (4.43)
  Day 1,905 (n=134, 68) | 38.11 (4.56) | 39.83 (3.90)
  Day 1,989 (n=121,56) | 38.07 (4.78) | 39.99 (4.12)
  Day 2,073 (n=81,38) | 37.11 (3.92) | 39.12 (3.45)
  Day 2,185 (n=82,37) | 37.25 (3.83) | 39.02 (3.45)

74. Primary Outcome: Mean Change From BL in Participant Hematocrit in the OL Period
Description: All changes in participant laboratory parameters were monitored on each day of study drug administration.
Time Frame: BL (Day 0), Day 365, Day 729, Day 1,093, Day 1,457, Day 1,821, Day 1,905, Day 1,989, Day 2,073, Day 2,185
Population: All treated participants in the OL period (treatment groups represent treatment received in the double-blind period).N = number of participants analyzed and n = the number of participants with measurements for that time point.
Measure: Mean (Standard Error); unit: Percentage Blood Volume Occupied by RBCs
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 378 | 161
Percentage Blood Volume Occupied by RBCs
  Day 365 (n=365, 157) | 1.87 (0.21) | -0.04 (0.24)
  Day 729 (n=328, 143) | 2.16 (0.20) | 1.36 (0.31)
  Day 1,093 (n=312, 138) | 1.41 (0.20) | 0.56 (0.35)
  Day 1,457 (n=292, 130) | 1.60 (0.23) | 1.01 (0.38)
  Day 1,821 (n=262,124) | 0.85 (0.25) | 0.78 (0.34)
  Day 1,905 (n=134, 68) | 1.63 (0.34) | 0.59 (0.48)
  Day 1,989 (n=121,56) | 1.42 (0.38) | 0.94 (0.49)
  Day 2,073 (n=81,38) | 1.79 (0.42) | 0.20 (0.62)
  Day 2,185 (n=82,37) | 1.42 (0.37) | 0.65 (0.61)

75. Primary Outcome: Mean BL Platelet Count in the OL Period
Description: Mean baseline values are those that are reported for each cohort at each time point on Day 365 to Day 2,185.
Time Frame: BL (Day 0), Day 365, Day 729, Day 1,093, Day 1,457, Day 1,821, Day 1,905, Day 1,989, Day 2,073, Day 2,185
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: 10^9 c/L
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 378 | 161
10^9 c/L
  Day 365 (n=365, 157) | 352.7 (108.5) | 339.2 (97.92)
  Day 729 (n=328, 143) | 351.8 (110.4) | 334.2 (91.41)
  Day 1,093 (n=312, 138) | 351.7 (107.9) | 334.8 (96.35)
  Day 1,457 (n=292, 130) | 352.7 (106.4) | 335.0 (98.59)
  Day 1,821 (n=262,124) | 351.1 (98.28) | 334.2 (97.52)
  Day 1,905 (n=134, 68) | 365.7 (113.9) | 333.7 (89.66)
  Day 1,989 (n=121,56) | 366.1 (115.3) | 326.6 (86.82)
  Day 2,073 (n=81,38) | 375.2 (118.6) | 321.2 (90.51)
  Day 2,185 (n=82,37) | 380.4 (119.7) | 320.3 (91.59)

76. Primary Outcome: Mean Change From BL in Participant Platelet Count in the OL Period
Description: All changes in participant laboratory parameters were monitored on each day of study drug administration.
Time Frame: BL (Day 0), Day 365, Day 729, Day 1,093, Day 1,457, Day 1,821, Day 1,905, Day 1,989, Day 2,073, Day 2,185
Population: as for outcome 73
Measure: Mean (Standard Error); unit: 10^9 c/L
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 378 | 161
10^9 c/L
  Day 365 (n=365, 157) | -66.9 (4.29) | -29.9 (5.58)
  Day 729 (n=328, 143) | -59.5 (4.64) | -45.4 (6.64)
  Day 1,093 (n=312, 138) | -53.5 (5.10) | -36.8 (7.21)
  Day 1,457 (n=292, 130) | -59.0 (5.64) | -48.7 (7.40)
  Day 1,821 (n=262,124) | -68.9 (4.92) | -59.2 (7.38)
  Day 1,905 (n=134, 68) | -55.1 (14.57) | -47.5 (10.71)
  Day 1,989 (n=121,56) | -63.7 (8.33) | -50.3 (9.83)
  Day 2,073 (n=81,38) | -69.6 (10.64) | -55.3 (11.68)
  Day 2,185 (n=82,37) | -80.5 (10.68) | -53.9 (10.34)

77. Primary Outcome: Mean BL Hemoglobin, Total Protein, and Albumin in the OL Period
Description: Mean baseline values are those that are reported for each cohort at each time point on Day 365 to Day 2,185.
Time Frame: BL (Day 0), Day 365, Day 729, Day 1,093, Day 1,457, Day 1,821, Day 1,905, Day 1,989, Day 2,073, Day 2,185
Population: as for outcome 73
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 378 | 161
g/dL
  Hemoglobin Day 365 (n=365, 157) | 12.49 (1.57) | 12.70 (1.56)
  Total Protein Day 365 (n=365, 157) | 7.23 (0.52) | 7.35 (0.56)
  Albumin Day 365 (n=365, 157) | 4.03 (0.33) | 4.13 (0.30)
  Hemoglobin Day 729 (n=328, 143) | 12.50 (1.54) | 12.72 (1.49)
  Total Protein Day 729 (n=328, 143) | 7.22 (0.52) | 7.34 (0.55)
  Albumin Day 729 (n=328, 143) | 4.01 (0.33) | 4.12 (0.29)
  Hemoglobin Day 1,093 (n=312, 138) | 12.48 (1.55) | 12.75 (1.55)
  Total Protein Day 1,093 (n=312, 138) | 7.23 (0.51) | 7.34 (0.55)
  Albumin Day 1,093 (n=312, 138) | 4.02 (0.33) | 4.11 (0.30)
  Hemoglobin Day 1,457 (n=292, 130) | 12.46 (1.54) | 12.74 (1.50)
  Total Protein Day 1,457 (n=292, 130) | 7.23 (0.51) | 7.35 (0.57)
  Albumin Day 1,457 (n=292, 130) | 4.02 (0.33) | 4.12 (0.30)
  Hemoglobin Day 1,821 (n=262,124) | 12.49 (1.51) | 12.79 (1.57)
  Total Protein Day 1,821 (n=262,124) | 7.23 (0.49) | 7.37 (0.56)
  Albumin Day 1,821 (n=262,124) | 4.02 (0.33) | 4.13 (0.30)
  Hemoglobin Day 1,905 (n=134, 68) | 12.35 (1.55) | 12.88 (1.33)
  Total Protein Day 1,905 (n=134, 68) | 7.27 (0.52) | 7.35 (0.53)
  Albumin Day 1,905 (n=134, 68) | 4.03 (0.32) | 4.13 (0.30)
  Hemoglobin Day 1,989 (n=121,56) | 12.35 (1.60) | 12.98 (1.46)
  Total Protein Day 1,989 (n=121,56) | 7.25 (0.51) | 7.38 (0.55)
  Albumin Day 1,989 (n=121,56) | 4.03 (0.33) | 4.12 (0.30)
  Hemoglobin Day 2,073 (n=81,38) | 12.21 (1.46) | 12.84 (1.18)
  Total Protein Day 2,073 (n=81,38) | 7.18 (0.47) | 7.27 (0.44)
  Albumin Day 2,073 (n=81,38) | 3.98 (0.33) | 4.08 (0.33)
  Hemoglobin Day 2,185 (n=82,37) | 12.25 (1.44) | 12.82 (1.19)
  Total Protein Day 2,185 (n=82,37) | 7.18 (0.47) | 7.28 (0.45)
  Albumin Day 2,185 (n=82,37) | 3.97 (0.32) | 4.08 (0.33)

78. Primary Outcome: Mean Change From BL in Hemoglobin, Total Protein, and Albumin in the OL Period
Description: All changes in participant laboratory parameters were monitored on each day of study drug administration.
Time Frame: BL (Day 0), Day 365, Day 729, Day 1,093, Day 1,457, Day 1,821, Day 1,905, Day 1,989, Day 2,073, Day 2,185
Population: as for outcome 73
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 378 | 161
g/dL
  Hemoglobin Day 365 (n=365, 157) | 0.62 (0.07) | -0.09 (0.08)
  Total Protein Day 365 (n=365, 157) | -0.26 (0.02) | -0.25 (0.04)
  Albumin Day 365 (n=365, 157) | 0.22 (0.02) | 0.02 (0.02)
  Hemoglobin Day 729 (n=328, 143) | 0.95 (0.07) | 0.61 (0.10)
  Total Protein Day 729 (n=328, 143) | -0.01 (0.03) | -0.05 (0.05)
  Albumin Day 729 (n=328, 143) | 0.31 (0.02) | 0.23 (0.03)
  Hemoglobin Day 1,093 (n=312, 138) | 0.75 (0.07) | 0.40 (0.11)
  Total Protein Day 1,093 (n=312, 138) | -0.16 (0.03) | -0.26 (0.04)
  Albumin Day 1,093 (n=312, 138) | 0.13 (0.02) | 0.02 (0.03)
  Hemoglobin Day 1,457 (n=292, 130) | 0.80 (0.07) | 0.52 (0.12)
  Total Protein Day 1,457 (n=292, 130) | -0.28 (0.03) | -0.35 (0.05)
  Albumin Day 1,457 (n=292, 130) | 0.07 (0.02) | -0.02 (0.03)
  Hemoglobin Day 1,821 (n=262,124) | 0.79 (0.08) | 0.70 (0.11)
  Total Protein Day 1,821 (n=262,124) | -0.27 (0.03) | -0.35 (0.05)
  Albumin Day 1,821 (n=262,124) | 0.06 (0.02) | -0.05 (0.03)
  Hemoglobin Day 1,905 (n=134, 68) | 0.74 (0.12) | 0.39 (0.16)
  Total Protein Day 1,905 (n=134, 68) | -0.32 (0.05) | -0.31 (0.07)
  Albumin Day 1,905 (n=134, 68) | 0.05 (0.03) | -0.06 (0.04)
  Hemoglobin Day 1,989 (n=121,56) | 0.59 (0.13) | 0.41 (0.17)
  Total Protein Day 1,989 (n=121,56) | -0.29 (0.05) | -0.33 (0.07)
  Albumin Day 1,989 (n=121,56) | 0.08 (0.03) | 0.01 (0.05)
  Hemoglobin Day 2,073 (n=81,38) | 0.78 (0.15) | 0.23 (0.22)
  Total Protein Day 2,073 (n=81,38) | -0.21 (0.04) | -0.24 (0.09)
  Albumin Day 2,073 (n=81,38) | 0.22 (0.03) | 0.09 (0.06)
  Hemoglobin Day 2,185 (n=82,37) | 0.69 (0.14) | 0.40 (0.21)
  Total Protein Day 2,185 (n=82,37) | -0.20 (0.04) | -0.12 (0.09)
  Albumin Day 2,185 (n=82,37) | 0.30 (0.03) | 0.25 (0.06)

79. Secondary Outcome: Mean Change From BL by Visit in the Physical Function Component of the SF-36 in the OL Period
Description: as for outcome 20
Time Frame: as for outcome 68
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  Day 365 (n=373, 160) | 8.61 (0.58) | 6.44 (0.84)
  Day 449 (n=367, 157) | 9.44 (0.57) | 9.13 (0.93)
  Day 533 (n=355, 157) | 9.43 (0.59) | 9.46 (0.97)
  Day 617 (n=348, 155) | 9.43 (0.57) | 9.80 (0.98)
  Day 729 (n=338, 148) | 9.51 (0.61) | 9.63 (1.03)
  Day 813 (n=324, 147) | 10.17 (0.62) | 9.71 (1.06)
  Day 897 (n=320, 140) | 9.95 (0.60) | 9.39 (1.07)
  Day 981 (n=312, 137) | 10.23 (0.63) | 10.45 (1.10)
  Day 1,093 (n=310, 138) | 9.40 (0.63) | 10.35 (1.15)
  Day 1,177 (n=275, 125) | 9.74 (0.71) | 10.57 (1.17)
  Day 1,261 (n=292, 135) | 9.95 (0.68) | 9.92 (1.14)
  Day 1,345 (n=147, 61) | 9.18 (1.00) | 10.75 (1.84)
  Day 1,457 (n=290, 129) | 10.55 (0.70) | 10.03 (1.15)
  Day 1,625 (n=279, 126) | 9.80 (0.72) | 9.68 (1.13)
  Day 1,821 (n=273, 125) | 9.48 (0.75) | 9.08 (1.10)
  Day 1,989 (n=118, 55) | 11.35 (1.17) | 9.22 (1.92)
  Day 2,185 (n=85, 38) | 10.06 (1.22) | 10.90 (2.25)

80. Secondary Outcome: Mean BL Role-Physical Component of the SF-36 by Visit in the OL Period
Description: The SF-36 covers 8 health dimensions including 4 physical subscales (physical function, role-physical, bodily pain, and general health) and 4 mental subscales (vitality, social function, role-emotional, and mental health). The scores range from a minimum of 0 to a maximum of 100, with a higher score indicating better quality of life. Improvements of > 3 points were considered clinically meaningful. Time-matched BL (Day 0) values and post-BL vales were presented for each post-BL visit and represent only that cohort of participants with measurements available at that post-BL assessment.
Time Frame: as for outcome 68
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  BL (Day 0) for Day 365 Cohort (n=372, 160) | 32.06 (7.78) | 32.08 (7.34)
  BL (Day 0) for Day 449 Cohort (n=367, 157) | 31.88 (7.64) | 32.02 (7.40)
  BL (Day 0) for Day 533 Cohort (n=355, 157) | 32.02 (7.78) | 32.11 (7.39)
  BL (Day 0) for Day 617 Cohort (n=348, 156) | 32.04 (7.81) | 32.14 (7.41)
  BL (Day 0) for Day 729 Cohort (n=338, 148) | 32.12 (7.86) | 31.79 (6.83)
  BL (Day 0) for Day 813 Cohort (n=324, 147) | 31.93 (7.65) | 31.91 (7.14)
  BL (Day 0) for Day 897 Cohort (n=320, 140) | 31.91 (7.56) | 32.01 (7.27)
  BL (Day 0) for Day 981 Cohort (n=312, 137) | 31.83 (7.52) | 32.05 (7.32)
  BL (Day 0) for Day 1,093 Cohort (n=309, 138) | 31.82 (7.52) | 32.02 (7.31)
  BL (Day 0) for Day 1,177 Cohort (n=275, 125) | 31.84 (7.55) | 31.88 (7.22)
  BL (Day 0) for Day 1,261 Cohort (n=292, 134) | 31.83 (7.56) | 32.09 (7.38)
  BL (Day 0) for Day 1,345 Cohort (n=147, 61) | 31.90 (7.13) | 31.66 (6.53)
  BL (Day 0) for Day 1,457 Cohort (n=289, 129) | 31.82 (7.57) | 32.08 (7.34)
  BL (Day 0) for Day 1,625 Cohort (n=279, 126) | 31.88 (7.60) | 31.96 (7.25)
  BL (Day 0) for Day 1,821 Cohort (n=273, 125) | 31.87 (7.71) | 31.71 (6.95)
  BL (Day 0) for Day 1,989 Cohort (n=118, 55) | 31.79 (7.72) | 31.43 (6.92)
  BL (Day 0) for Day 2,185 Cohort (n=84, 38) | 30.98 (6.88) | 30.56 (5.05)

81. Secondary Outcome: Mean Change From BL by Visit in the Role-Physical Component of the SF-36 in the OL Period
Description: as for outcome 20
Time Frame: as for outcome 68
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  Day 365 (n=372, 160) | 10.10 (0.67) | 7.59 (0.96)
  Day 449 (n=367, 157) | 10.66 (0.70) | 10.89 (1.04)
  Day 533 (n=355, 157) | 11.18 (0.70) | 10.98 (1.02)
  Day 617 (n=348, 156) | 10.93 (0.73) | 11.61 (1.05)
  Day 729 (n=338, 148) | 11.33 (0.72) | 11.50 (1.04)
  Day 813 (n=324, 147) | 10.56 (0.73) | 10.57 (1.00)
  Day 897 (n=320, 140) | 10.13 (0.74) | 10.96 (1.06)
  Day 981 (n=312, 137) | 10.96 (0.76) | 10.88 (1.07)
  Day 1,093 (n=309, 138) | 11.82 (0.76) | 9.72 (1.04)
  Day 1,177 (n=275, 125) | 11.32 (0.82) | 11.09 (1.18)
  Day 1,261 (n=292, 134) | 10.25 (0.82) | 11.61 (1.08)
  Day 1,345 (n=147, 61) | 9.09 (1.13) | 10.32 (1.67)
  Day 1,457 (n=289, 129) | 10.57 (0.79) | 11.39 (1.13)
  Day 1,625 (n=279, 126) | 10.11 (0.80) | 11.10 (1.10)
  Day 1,821 (n=273, 125) | 11.25 (0.84) | 10.62 (1.15)
  Day 1,989 (n=118, 55) | 10.79 (1.31) | 10.42 (1.71)
  Day 2,185 (n=84, 38) | 9.04 (1.41) | 12.84 (1.96)

82. Secondary Outcome: Mean BL Bodily Pain Component of the SF-36 by Visit in the OL Period
Description: as for outcome 80
Time Frame: as for outcome 68
Population: AlAll treated participants in the OL period (Treatment groups represent treatment received in the DB period). Due to the non-compliance of a single site, 3 participants were not included in this analysis. N = number of participants analyzed and n = the number of participants with measurements for that time point.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  BL (Day 0) for Day 365 Cohort (n=373, 160) | 33.13 (7.37) | 33.43 (7.53)
  BL (Day 0) for Day 449 Cohort (n=367, 157) | 32.95 (7.36) | 33.47 (7.56)
  BL (Day 0) for Day 533 Cohort (n=355, 157) | 33.05 (7.36) | 33.27 (7.49)
  BL (Day 0) for Day 617 Cohort (n=348, 156) | 33.00 (7.30) | 33.49 (7.59)
  BL (Day 0) for Day 729 Cohort (n=338, 148) | 32.94 (7.38) | 33.44 (7.57)
  BL (Day 0) for Day 813 Cohort (n=324, 147) | 32.80 (7.27) | 33.53 (7.65)
  BL (Day 0) for Day 897 Cohort (n=320, 140) | 32.80 (7.33) | 33.29 (7.67)
  BL (Day 0) for Day 981 Cohort (n=312, 137) | 32.79 (7.28) | 33.29 (7.74)
  BL (Day 0) for Day 1,093 Cohort (n=309, 138) | 32.88 (7.30) | 33.29 (7.71)
  BL (Day 0) for Day 1,177 Cohort (n=275, 125) | 32.84 (7.34) | 33.13 (7.71)
  BL (Day 0) for Day 1,261 Cohort (n=291, 134) | 32.81 (7.50) | 33.31 (7.77)
  BL (Day 0) for Day 1,345 Cohort (n=147, 61) | 32.57 (7.37) | 31.83 (6.61)
  BL (Day 0) for Day 1,457 Cohort (n=289, 129) | 32.73 (7.35) | 33.48 (7.74)
  BL (Day 0) for Day 1,625 Cohort (n=279, 126) | 32.78 (7.36) | 33.20 (7.52)
  BL (Day 0) for Day 1,821 Cohort (n=273, 125) | 32.85 (7.44) | 33.56 (7.71)
  BL (Day 0) for Day 1,989 Cohort (n=118, 55) | 31.98 (7.20) | 32.81 (7.66)
  BL (Day 0) for Day 2,185 Cohort (n=85, 38) | 31.49 (6.81) | 31.40 (5.91)

83. Secondary Outcome: Mean Change From BL by Visit in the Bodily Pain Component of the SF-36 in the OL Period
Description: as for outcome 20
Time Frame: as for outcome 68
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  Day 365 (n=373, 160) | 12.08 (0.51) | 7.98 (0.76)
  Day 449 (n=367, 157) | 12.38 (0.53) | 11.78 (0.82)
  Day 533 (n=355, 157) | 11.94 (0.55) | 12.53 (0.86)
  Day 617 (n=348, 156) | 12.52 (0.56) | 11.97 (0.90)
  Day 729 (n=338, 148) | 12.84 (0.57) | 12.06 (0.88)
  Day 813 (n=324, 147) | 13.13 (0.60) | 12.25 (0.85)
  Day 897 (n=320, 140) | 12.44 (0.59) | 11.84 (0.85)
  Day 981 (n=312, 137) | 12.86 (0.63) | 12.87 (0.87)
  Day 1,093 (n=309, 138) | 13.34 (0.60) | 12.93 (0.91)
  Day 1,177 (n=275, 125) | 13.21 (0.67) | 13.44 (1.02)
  Day 1,261 (n=291, 134) | 12.83 (0.68) | 13.31 (0.94)
  Day 1,345 (n=147, 61) | 12.44 (0.98) | 13.40 (1.42)
  Day 1,457 (n=289, 129) | 13.13 (0.60) | 11.74 (0.97)
  Day 1,625 (n=279, 126) | 12.89 (0.63) | 13.36 (0.89)
  Day 1,821 (n=273, 125) | 12.56 (0.67) | 12.65 (0.95)
  Day 1,989 (n=118, 55) | 13.45 (0.98) | 13.19 (1.41)
  Day 2,185 (n=85, 38) | 10.44 (1.18) | 14.28 (1.47)

84. Secondary Outcome: Mean BL General Health Component of the SF-36 by Visit in the OL Period
Description: as for outcome 80
Time Frame: as for outcome 68
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  BL (Day 0) for Day 365 Cohort (n=373, 160) | 35.43 (8.41) | 35.27 (7.73)
  BL (Day 0) for Day 449 Cohort (n=367, 157) | 35.33 (8.45) | 35.28 (7.80)
  BL (Day 0) for Day 533 Cohort (n=355, 157) | 35.34 (8.40) | 35.17 (7.73)
  BL (Day 0) for Day 617 Cohort (n=348, 156) | 35.41 (8.38) | 35.21 (7.72)
  BL (Day 0) for Day 729 Cohort (n=338, 148) | 35.47 (8.46) | 35.16 (7.61)
  BL (Day 0) for Day 813 Cohort (n=324, 147) | 35.59 (8.45) | 35.19 (7.62)
  BL (Day 0) for Day 897 Cohort (n=320, 140) | 35.72 (8.50) | 35.22 (7.78)
  BL (Day 0) for Day 981 Cohort (n=312, 137) | 35.67 (8.46) | 35.38 (7.79)
  BL (Day 0) for Day 1,093 Cohort (n=312, 138) | 35.69 (8.52) | 35.32 (7.80)
  BL (Day 0) for Day 1,177 Cohort (n=275, 125) | 35.50 (8.38) | 35.54 (7.87)
  BL (Day 0) for Day 1,261 Cohort (n=291, 135) | 35.65 (8.38) | 35.31 (7.88)
  BL (Day 0) for Day 1,345 Cohort (n=147, 61) | 35.88 (8.68) | 33.78 (7.96)
  BL (Day 0) for Day 1,457 Cohort (n=290, 129) | 35.56 (8.48) | 35.43 (7.85)
  BL (Day 0) for Day 1,625 Cohort (n=280, 126) | 35.67 (8.33) | 35.23 (7.91)
  BL (Day 0) for Day 1,821 Cohort (n=273, 125) | 35.61 (8.46) | 35.56 (7.83)
  BL (Day 0) for Day 1,989 Cohort (n=119, 55) | 34.87 (8.65) | 34.94 (8.67)
  BL (Day 0) for Day 2,185 Cohort (n=85, 38) | 34.29 (9.03) | 33.71 (8.26)

85. Secondary Outcome: Mean Change From BL by Visit in the General Health Component of the SF-36 in the OL Period
Description: as for outcome 20
Time Frame: as for outcome 68
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  Day 365 (n=373, 160) | 6.88 (0.46) | 5.43 (0.58)
  Day 449 (n=367, 157) | 6.94 (0.46) | 7.32 (0.71)
  Day 533 (n=355, 157) | 6.82 (0.47) | 7.88 (0.68)
  Day 617 (n=348, 156) | 7.22 (0.45) | 7.87 (0.70)
  Day 729 (n=338, 148) | 7.31 (0.46) | 7.90 (0.68)
  Day 813 (n=324, 147) | 6.89 (0.49) | 7.63 (0.69)
  Day 897 (n=320, 140) | 6.86 (0.52) | 8.24 (0.79)
  Day 981 (n=312, 137) | 7.31 (0.53) | 8.45 (0.79)
  Day 1,093 (n=312, 138) | 7.24 (0.55) | 8.36 (0.82)
  Day 1,177 (n=275, 125) | 7.48 (0.57) | 8.55 (0.94)
  Day 1,261 (n=291, 135) | 7.18 (0.58) | 8.17 (0.83)
  Day 1,345 (n=147, 61) | 6.19 (0.73) | 8.45 (1.36)
  Day 1,457 (n=290, 129) | 7.07 (0.57) | 8.32 (0.86)
  Day 1,625 (n=280, 126) | 7.27 (0.57) | 8.10 (0.81)
  Day 1,821 (n=273, 125) | 7.50 (0.60) | 7.53 (0.81)
  Day 1,989 (n=119, 55) | 6.55 (0.81) | 7.05 (1.14)
  Day 2,185 (n=85, 38) | 5.93 (1.02) | 8.76 (1.38)

86. Secondary Outcome: Mean BL Social Functioning Component of the SF-36 by Visit in the OL Period
Description: as for outcome 19
Time Frame: as for outcome 68
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  BL (Day 0) for Day 365 Cohort (n=373, 160) | 35.58 (10.10) | 34.98 (9.72)
  BL (Day 0) for Day 449 Cohort (n=368, 157) | 35.42 (10.13) | 34.91 (9.75)
  BL (Day 0) for Day 533 Cohort (n=355, 157) | 35.52 (10.18) | 34.94 (9.80)
  BL (Day 0) for Day 617 Cohort (n=348, 156) | 35.46 (10.14) | 35.01 (9.80)
  BL (Day 0) for Day 729 Cohort (n=338, 148) | 35.70 (10.24) | 34.51 (9.61)
  BL (Day 0) for Day 813 Cohort (n=324, 147) | 35.47 (10.17) | 34.57 (9.73)
  BL (Day 0) for Day 897 Cohort (n=320, 140) | 35.47 (10.20) | 34.65 (9.82)
  BL (Day 0) for Day 981 Cohort (n=312, 137) | 35.46 (10.17) | 34.67 (9.90)
  BL (Day 0) for Day 1,093 Cohort (n=312, 138) | 35.60 (10.07) | 34.68 (9.86)
  BL (Day 0) for Day 1,177 Cohort (n=275, 125) | 35.52 (10.10) | 34.51 (9.60)
  BL (Day 0) for Day 1,261 Cohort (n=292, 134) | 35.48 (10.24) | 34.82 (9.93)
  BL (Day 0) for Day 1,345 Cohort (n=147, 62) | 35.65 (10.53) | 33.24 (9.09)
  BL (Day 0) for Day 1,457 Cohort (n=289, 129) | 35.56 (10.28) | 34.83 (9.82)
  BL (Day 0) for Day 1,625 Cohort (n=280, 126) | 35.44 (10.45) | 34.73 (9.90)
  BL (Day 0) for Day 1,821 Cohort (n=273, 125) | 35.56 (10.42) | 34.86 (9.52)
  BL (Day 0) for Day 1,989 Cohort (n=118, 55) | 34.50 (10.41) | 33.75 (8.92)
  BL (Day 0) for Day 2,185 Cohort (n=85, 38) | 34.66 (10.43) | 31.85 (8.21)

87. Secondary Outcome: Mean Change From BL by Visit in the Social Functioning Component of the SF-36 in the OL Period
Description: as for outcome 20
Time Frame: as for outcome 68
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  Day 365 (n=373, 160) | 9.01 (0.61) | 7.12 (0.77)
  Day 449 (n=368, 157) | 9.74 (0.61) | 9.47 (0.91)
  Day 533 (n=355, 157) | 9.88 (0.62) | 9.44 (0.92)
  Day 617 (n=348, 156) | 9.48 (0.62) | 8.66 (0.92)
  Day 729 (n=338, 148) | 9.99 (0.63) | 9.90 (0.94)
  Day 813 (n=324, 147) | 9.80 (0.67) | 8.97 (0.92)
  Day 897 (n=320, 140) | 9.96 (0.67) | 9.81 (0.99)
  Day 981 (n=312, 137) | 9.71 (0.66) | 9.51 (1.00)
  Day 1,093 (n=312, 138) | 10.16 (0.68) | 8.61 (0.98)
  Day 1,177 (n=275, 125) | 9.28 (0.71) | 9.64 (1.06)
  Day 1,261 (n=292, 134) | 9.54 (0.73) | 9.92 (0.99)
  Day 1,345 (n=147, 62) | 9.01 (1.11) | 8.84 (1.42)
  Day 1,457 (n=289, 129) | 10.16 (0.72) | 9.26 (1.01)
  Day 1,625 (n=280, 126) | 9.67 (0.73) | 9.05 (0.99)
  Day 1,821 (n=273, 125) | 8.93 (0.75) | 8.16 (0.91)
  Day 1,989 (n=118, 55) | 9.34 (1.17) | 10.17 (1.37)
  Day 2,185 (n=85, 38) | 7.98 (1.31) | 10.57 (1.40)

88. Secondary Outcome: Mean BL Role-Emotional Component of the SF-36 by Visit in the OL Period
Description: as for outcome 80
Time Frame: as for outcome 68
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  BL (Day 0) for Day 365 Cohort (n= 370, 158) | 35.78 (13.63) | 33.40 (12.53)
  BL (Day 0) for Day 449 Cohort (n=365, 157) | 35.71 (13.61) | 33.26 (12.44)
  BL (Day 0) for Day 533 Cohort (n=355, 156) | 35.61 (13.57) | 33.39 (12.61)
  BL (Day 0) for Day 617 Cohort (n=348, 155) | 35.66 (13.55) | 33.52 (12.60)
  BL (Day 0) for Day 729 Cohort (n=338, 147) | 35.49 (13.49) | 33.34 (12.45)
  BL (Day 0) for Day 813 Cohort (n=324, 146) | 35.38 (13.42) | 33.26 (12.52)
  BL (Day 0) for Day 897 Cohort (n=320, 139) | 35.46 (13.40) | 33.13 (12.60)
  BL (Day 0) for Day 981 Cohort (n=312, 136) | 35.42 (13.36) | 33.19 (12.65)
  BL (Day 0) for Day 1,093 Cohort (n=309, 137) | 35.40 (13.36) | 33.27 (12.64)
  BL (Day 0) for Day 1,177 Cohort (n=275, 124) | 35.46 (13.34) | 33.42 (12.57)
  BL (Day 0) for Day 1,261 Cohort (n=291, 133) | 35.61 (13.44) | 33.00 (12.51)
  BL (Day 0) for Day 1,345 Cohort (n=146, 60) | 36.00 (13.78) | 32.69 (12.39)
  BL (Day 0) for Day 1,457 Cohort (n=289, 128) | 35.36 (13.44) | 32.79 (12.31)
  BL (Day 0) for Day 1,625 Cohort (n=279, 125) | 35.33 (13.39) | 32.92 (12.48)
  BL (Day 0) for Day 1,821 Cohort (n=273, 124) | 35.43 (13.50) | 32.74 (12.14)
  BL (Day 0) for Day 1,989 Cohort (n=118, 54) | 35.61 (13.67) | 30.76 (11.58)
  BL (Day 0) for Day 2,185 Cohort (n=85, 38) | 35.26 (13.76) | 29.28 (10.32)

89. Secondary Outcome: Mean Change From BL by Visit in the Role-Emotional Component of the SF-36 in the OL Period
Description: as for outcome 20
Time Frame: as for outcome 68
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  Day 365 (n= 370, 158) | 8.97 (0.81) | 8.60 (1.25)
  Day 449 (n=365, 157) | 8.02 (0.86) | 10.80 (1.28)
  Day 533 (n=355, 156) | 8.44 (0.88) | 10.13 (1.30)
  Day 617 (n=348, 155) | 8.60 (0.88) | 10.47 (1.34)
  Day 729 (n=338, 147) | 8.96 (0.86) | 10.89 (1.34)
  Day 813 (n=324, 146) | 8.71 (0.89) | 11.04 (1.37)
  Day 897 (n=320, 139) | 8.48 (0.90) | 11.67 (1.41)
  Day 981 (n=312, 136) | 8.61 (0.92) | 11.70 (1.42)
  Day 1,093 (n=309, 137) | 9.31 (0.94) | 9.46 (1.41)
  Day 1,177 (n=275, 124) | 8.35 (1.01) | 11.17 (1.48)
  Day 1,261 (n=291, 133) | 8.43 (1.00) | 10.53 (1.42)
  Day 1,345 (n=146, 60) | 7.22 (1.35) | 11.41 (2.23)
  Day 1,457 (n=289, 128) | 7.51 (0.98) | 10.70 (1.46)
  Day 1,625 (n=279, 125) | 7.91 (1.02) | 9.44 (1.53)
  Day 1,821 (n=273, 124) | 7.39 (0.71) | 6.56 (1.09)
  Day 1,989 (n=118, 54) | 7.81 (1.60) | 12.49 (2.18)
  Day 2,185 (n=85, 38) | 7.06 (1.69) | 16.08 (2.17)

90. Secondary Outcome: Mean BL Vitality Component of the SF-36 by Visit in the OL Period
Description: as for outcome 80
Time Frame: as for outcome 68
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  BL (Day 0) for Day 365 Cohort (n=373, 159) | 40.93 (9.14) | 41.29 (8.35)
  BL (Day 0) for Day 449 Cohort (n=368, 156) | 40.77 (9.11) | 41.21 (8.38)
  BL (Day 0) for Day 533 Cohort (n=355, 156) | 40.68 (8.99) | 41.21 (8.40)
  BL (Day 0) for Day 617 Cohort (n=348, 155) | 40.77 (9.02) | 41.40 (8.37)
  BL (Day 0) for Day 729 Cohort (n=338, 147) | 40.74 (9.11) | 41.19 (8.34)
  BL (Day 0) for Day 813 Cohort (n=323, 146) | 40.60 (9.06) | 41.27 (8.46)
  BL (Day 0) for Day 897 Cohort (n=320, 140) | 40.79 (9.11) | 41.34 (8.45)
  BL (Day 0) for Day 981 Cohort (n=312, 137) | 40.85 (9.00) | 41.43 (8.45)
  BL (Day 0) for Day 1,093 Cohort (n=312, 138) | 40.85 (9.07) | 41.33 (8.50)
  BL (Day 0) for Day 1,177 Cohort (n=273, 125) | 40.69 (9.23) | 41.23 (8.42)
  BL (Day 0) for Day 1,261 Cohort (n=292, 134) | 40.78 (9.15) | 41.31 (8.57)
  BL (Day 0) for Day 1,345 Cohort (n=147, 62) | 41.30 (9.39) | 40.64 (7.84)
  BL (Day 0) for Day 1,457 Cohort (n=290, 129) | 40.79 (9.21) | 41.47 (8.17)
  BL (Day 0) for Day 1,625 Cohort (n=280, 126) | 40.84 (9.18) | 41.23 (8.29)
  BL (Day 0) for Day 1,821 Cohort (n=273, 125) | 40.82 (9.27) | 41.47 (8.36)
  BL (Day 0) for Day 1,989 Cohort (n=118, 55) | 42.19 (8.85) | 41.72 (8.01)
  BL (Day 0) for Day 2,185 Cohort (n=85, 38) | 41.16 (9.08) | 39.88 (8.31)

91. Secondary Outcome: Mean Change From BL by Visit in the Vitality Component of the SF-36 in the OL Period
Description: as for outcome 20
Time Frame: as for outcome 68
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  Day 365 (n=373, 159) | 8.58 (0.55) | 6.04 (0.68)
  Day 449 (n=368, 156) | 8.29 (0.55) | 8.70 (0.76)
  Day 533 (n=355, 156) | 8.68 (0.52) | 8.09 (0.81)
  Day 617 (n=348, 155) | 8.61 (0.53) | 8.46 (0.79)
  Day 729 (n=338, 147) | 8.69 (0.55) | 8.41 (0.80)
  Day 813 (n=323, 146) | 8.99 (0.58) | 8.22 (0.83)
  Day 897 (n=320, 140) | 8.69 (0.57) | 8.53 (0.81)
  Day 981 (n=312, 137) | 8.85 (0.58) | 7.52 (0.83)
  Day 1,093 (n=312, 138) | 8.98 (0.56) | 7.53 (0.82)
  Day 1,177 (n=273, 125) | 9.08 (0.63) | 8.08 (0.85)
  Day 1,261 (n=292, 134) | 8.39 (0.64) | 8.14 (0.84)
  Day 1,345 (n=147, 62) | 8.29 (0.91) | 6.39 (1.25)
  Day 1,457 (n=290, 129) | 9.19 (0.62) | 7.57 (0.87)
  Day 1,625 (n=280, 126) | 8.77 (0.64) | 8.20 (0.85)
  Day 1,821 (n=273, 125) | 8.96 (0.66) | 7.42 (0.84)
  Day 1,989 (n=118, 55) | 7.60 (0.99) | 7.99 (1.26)
  Day 2,185 (n=85, 38) | 7.06 (1.11) | 9.61 (1.28)

92. Secondary Outcome: Mean BL Mental Health Component of the SF-36 by Visit in the OL Period
Description: as for outcome 80
Time Frame: as for outcome 68
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  BL (Day 0) for Day 365 Cohort (n=373, 159) | 39.08 (11.55) | 39.43 (11.09)
  BL (Day 0) for Day 449 Cohort (n=368, 156) | 38.87 (11.46) | 39.33 (11.14)
  BL (Day 0) for Day 533 Cohort (n=355, 156) | 38.89 (11.44) | 39.40 (11.18)
  BL (Day 0) for Day 617 Cohort (n=348, 155) | 38.76 (11.46) | 39.49 (11.14)
  BL (Day 0) for Day 729 Cohort (n=338, 147) | 38.75 (11.56) | 39.05 (11.18)
  BL (Day 0) for Day 813 Cohort (n=323, 146) | 38.85 (11.57) | 39.01 (11.19)
  BL (Day 0) for Day 897 Cohort (n=320, 140) | 38.96 (11.66) | 39.03 (11.35)
  BL (Day 0) for Day 981 Cohort (n=312, 137) | 39.06 (11.58) | 39.09 (11.46)
  BL (Day 0) for Day 1,093 Cohort (n=312, 138) | 39.16 (11.47) | 39.08 (11.42)
  BL (Day 0) for Day 1,177 Cohort (n=273, 125) | 38.88 (11.54) | 38.67 (11.22)
  BL (Day 0) for Day 1,261 Cohort (n=292, 134) | 38.81 (11.56) | 39.15 (11.49)
  BL (Day 0) for Day 1,345 Cohort (n=147, 62) | 39.91 (11.46) | 39.33 (11.21)
  BL (Day 0) for Day 1,457 Cohort (n=290, 129) | 38.83 (11.62) | 38.93 (11.42)
  BL (Day 0) for Day 1,625 Cohort (n=280, 126) | 38.88 (11.66) | 38.97 (11.46)
  BL (Day 0) for Day 1,821 Cohort (n=273, 125) | 39.06 (11.72) | 38.95 (11.44)
  BL (Day 0) for Day 1,989 Cohort (n=118, 55) | 38.95 (10.99) | 39.90 (10.63)
  BL (Day 0) for Day 2,185 Cohort (n=85, 38) | 39.32 (12.04) | 37.40 (10.09)

93. Secondary Outcome: Mean Change From BL by Visit in the Mental Health Component of the SF-36 in the OL Period
Description: as for outcome 20
Time Frame: as for outcome 68
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  Day 365 (n=373, 159) | 7.02 (0.59) | 5.31 (0.78)
  Day 449 (n=368, 156) | 7.27 (0.58) | 6.45 (0.89)
  Day 533 (n=355, 156) | 7.72 (0.61) | 6.49 (0.88)
  Day 617 (n=348, 155) | 7.60 (0.61) | 6.03 (0.93)
  Day 729 (n=338, 147) | 7.49 (0.61) | 7.38 (0.96)
  Day 813 (n=323, 146) | 7.26 (0.66) | 5.72 (0.93)
  Day 897 (n=320, 140) | 7.65 (0.67) | 7.29 (0.96)
  Day 981 (n=312, 137) | 7.13 (0.65) | 6.97 (1.00)
  Day 1,093 (n=312, 138) | 7.85 (0.62) | 5.81 (0.99)
  Day 1,177 (n=273, 125) | 7.67 (0.68) | 7.02 (1.07)
  Day 1,261 (n=292, 134) | 8.18 (0.70) | 6.14 (1.03)
  Day 1,345 (n=147, 62) | 6.80 (0.93) | 7.01 (1.25)
  Day 1,457 (n=290, 129) | 7.75 (0.70) | 6.51 (1.01)
  Day 1,625 (n=280, 126) | 6.96 (0.70) | 7.13 (1.10)
  Day 1,821 (n=273, 125) | 7.39 (0.71) | 6.56 (1.09)
  Day 1,989 (n=118, 55) | 6.58 (1.08) | 6.65 (1.57)
  Day 2,185 (n=85, 38) | 5.92 (1.22) | 7.10 (1.60)

94. Secondary Outcome: Mean BL Fatigue in the OL Period
Description: Mean baseline values are reported for each cohort at each time point using the VAS 100 mm where 0= no fatigue to 100 = the worst fatigue imaginable. Time-matched BL(Day 0) values and post-BL vales were presented for each post-BL visit and represent only that cohort of participants with measurements available at that post-BL assessment.
Time Frame: as for outcome 68
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  BL (Day 0) for Day 365 Cohort (n=373, 160) | 63.52 (23.23) | 65.37 (22.96)
  BL (Day 0) for Day 449 Cohort (n=358, 156) | 63.59 (23.51) | 65.28 (23.24)
  BL (Day 0) for Day 533 Cohort (n=353, 157) | 63.25 (23.57) | 65.78 (22.89)
  BL (Day 0) for Day 617 Cohort (n=339, 150) | 63.19 (23.48) | 64.73 (23.42)
  BL (Day 0) for Day 729 Cohort (n=329, 143) | 63.53 (23.15) | 64.59 (23.73)
  BL (Day 0) for Day 813 Cohort (n=318, 141) | 63.77 (22.77) | 64.81 (23.59)
  BL (Day 0) for Day 897 Cohort (n=316, 139) | 63.61 (23.11) | 65.36 (23.29)
  BL (Day 0) for Day 981 Cohort (n=312, 137) | 63.58 (22.99) | 65.51 (23.43)
  BL (Day 0) for Day 1,093 Cohort (n=307, 138) | 63.33 (23.18) | 65.47 (23.34)
  BL (Day 0) for Day 1,177 Cohort (n=271, 123) | 64.05 (22.73) | 65.18 (23.11)
  BL (Day 0) for Day 1,261 Cohort (n=289, 133) | 63.38 (23.37) | 65.56 (23.19)
  BL (Day 0) for Day 1,345 Cohort (n=141, 59) | 65.64 (21.44) | 69.00 (20.57)
  BL (Day 0) for Day 1,457 Cohort (n=283, 129) | 63.66 (23.51) | 65.50 (23.00)
  BL (Day 0) for Day 1,625 Cohort (n=275, 124) | 63.18 (23.78) | 66.34 (22.48)
  BL (Day 0) for Day 1,821 Cohort (n=263, 125) | 62.48 (23.84) | 65.00 (23.15)
  BL (Day 0) for Day 1,989 Cohort (n=115, 53) | 64.36 (23.88) | 67.45 (22.16)
  BL (Day 0) for Day 2,185 Cohort (n=81, 37) | 64.77 (22.45) | 70.17 (19.01)

95. Secondary Outcome: Mean Change From BL in Fatigue in the OL Period
Description: The mean change from baseline in fatigue was measured on the VAS 100 mm where 0= no fatigue to 100 = the worst fatigue imaginable.
Time Frame: as for outcome 68
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  Day 365 (n=373, 160) | -28.0 (1.49) | -22.6 (2.21)
  Day 449 (n=358, 156) | -28.5 (1.55) | -31.1 (2.43)
  Day 533 (n=353, 157) | -29.4 (1.51) | -31.1 (2.46)
  Day 617 (n=339, 150) | -30.4 (1.60) | -30.5 (2.54)
  Day 729 (n=329, 143) | -31.2 (1.60) | -30.0 (2.67)
  Day 813 (n=318, 141) | -29.9 (1.60) | -31.0 (2.42)
  Day 897 (n=316, 139) | -29.7 (1.66) | -30.6 (2.45)
  Day 981 (n=312, 137) | -30.5 (1.69) | -31.1 (2.56)
  Day 1,093 (n=307, 138) | -32.8 (1.61) | -31.3 (2.53)
  Day 1,177 (n=271, 123) | -32.2 (1.83) | -33.3 (2.69)
  Day 1,261 (n=289, 133) | -30.3 (1.70) | -31.2 (2.62)
  Day 1,345 (n=141, 59) | -33.9 (2.42) | -28.2 (3.80)
  Day 1,457 (n=283, 129) | -32.2 (1.65) | -32.6 (2.62)
  Day 1,625 (n=275, 124) | -30.9 (1.69) | -32.3 (2.56)
  Day 1,821 (n=263, 125) | -30.3 (1.82) | -32.0 (2.65)
  Day 1,989 (n=115, 53) | -33.6 (2.80) | -33.7 (4.18)
  Day 2,185 (n=81, 37) | -29.4 (3.22) | -35.0 (4.49)

96. Secondary Outcome: Mean BL Sleep Quality in the OL Period
Description: Mean baseline values are reported for each cohort at each time point using the Medical Outcomes Study Sleep scale (MOS-sleep [assesses the extent of sleep problems and measures six dimensions of sleep on a 12-item participant-reported measure]). An overall Sleep Problems Index (SPI) was generated as a summary measure of different types of sleep problems (sleep disturbance, sleep quantity, sleep adequacy, etc.). The score ranges from 0 to 100, with 0 = no problems with sleep and 100 = the most severe problems with sleep. The mean score of the SPI in a population with chronic conditions is 29.
Time Frame: as for outcome 68
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  BL (Day 0) for Day 365 Cohort (n=373, 160) | 42.42 (19.96) | 43.53 (19.59)
  BL (Day 0) for Day 449 Cohort (n=358, 156) | 42.77 (20.07) | 43.22 (19.64)
  BL (Day 0) for Day 533 Cohort (n=353, 157) | 42.62 (20.11) | 43.24 (19.39)
  BL (Day 0) for Day 617 Cohort (n=339, 150) | 42.51 (20.19) | 43.24 (19.90)
  BL (Day 0) for Day 729 Cohort (n=329, 143) | 42.28 (20.01) | 43.97 (19.75)
  BL (Day 0) for Day 813 Cohort (n=318, 141) | 42.63 (20.07) | 43.58 (19.70)
  BL (Day 0) for Day 897 Cohort (n=316, 139) | 42.60 (20.31) | 43.65 (19.83)
  BL (Day 0) for Day 981 Cohort (n=312, 137) | 42.51 (20.25) | 43.58 (19.78)
  BL (Day 0) for Day 1,093 Cohort (n=307, 138) | 42.69 (20.36) | 43.78 (19.84)
  BL (Day 0) for Day 1,177 Cohort (n=270, 124) | 43.08 (20.28) | 43.51 (19.52)
  BL (Day 0) for Day 1,261 Cohort (n=289, 133) | 42.87 (20.40) | 43.76 (19.83)
  BL (Day 0) for Day 1,345 Cohort (n=141, 59) | 41.78 (21.79) | 48.39 (20.23)
  BL (Day 0) for Day 1,457 Cohort (n=275, 124) | 42.93 (20.82) | 44.14 (19.74)
  BL (Day 0) for Day 1,625 Cohort (n=272, 122) | 42.70 (20.46) | 44.51 (20.00)
  BL (Day 0) for Day 1,821 Cohort (n=263, 125) | 42.04 (20.53) | 43.59 (20.00)
  BL (Day 0) for Day 1,989 Cohort (n=115, 53) | 43.15 (22.33) | 47.62 (20.33)
  BL (Day 0) for Day 2,185 Cohort (n=81, 37) | 42.70 (22.06) | 51.43 (19.75)

97. Secondary Outcome: Mean Change From BL in Sleep Quality in the OL Period
Description: The mean change from baseline in sleep quality was assessed on the Medical Outcomes Study Sleep scale (MOS-sleep [assesses the extent of sleep problems and measures six dimensions of sleep on a 12-item participant-reported measure]). An overall Sleep Problems Index (SPI) was generated as a summary measure of different types of sleep problems (sleep disturbance, sleep quantity, sleep adequacy, etc.). The score ranges from 0 to 100, with 0 = no problems with sleep and 100 = the most severe problems with sleep. The mean score of the SPI in a population with chronic conditions is 29.
Time Frame: as for outcome 68
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  Day 365 (n=373, 160) | -10.8 (0.91) | -7.97 (1.25)
  Day 449 (n=358, 156) | -11.0 (0.97) | -11.4 (1.36)
  Day 533 (n=353, 157) | -11.4 (0.92) | -10.9 (1.42)
  Day 617 (n=339, 150) | -10.6 (0.92) | -11.9 (1.41)
  Day 729 (n=329, 143) | -10.9 (0.99) | -11.3 (1.48)
  Day 813 (n=318, 141) | -10.9 (1.07) | -10.8 (1.57)
  Day 897 (n=316, 139) | -12.2 (1.04) | -12.0 (1.46)
  Day 981 (n=312, 137) | -11.4 (1.05) | -10.8 (1.58)
  Day 1,093 (n=307, 138) | -11.9 (1.09) | -11.3 (1.53)
  Day 1,177 (n=270, 124) | -11.9 (1.19) | -10.8 (1.61)
  Day 1,261 (n=289, 133) | -12.2 (1.16) | -10.1 (1.59)
  Day 1,345 (n=141, 59) | -11.6 (1.68) | -12.5 (2.17)
  Day 1,457 (n=275, 124) | -11.7 (1.16) | -10.4 (1.62)
  Day 1,625 (n=272, 122) | -11.2 (1.19) | -11.6 (1.72)
  Day 1,821 (n=263, 125) | -10.8 (1.23) | -9.10 (1.50)
  Day 1,989 (n=115, 53) | -11.7 (1.98) | -11.0 (2.40)
  Day 2,185 (n=81, 37) | -8.76 (2.03) | -14.6 (2.92)

98. Secondary Outcome: Mean BL Limitations on Activities of Daily Living in the OL Period
Description: Mean baseline values are reported for each cohort at each time point. Activity limitation was measured by the number of days in the past 30 days a participant was unable to perform usual activities due to RA. Time-matched BL (Day 0) values and post-BL vales were presented for each post-BL visit and represent only that cohort of participants with measurements available at that post-BL assessment.
Time Frame: BL (Day 0), Day 365, Day 449, Day 533, Day 729, Day 813, Day 897, Day 981, Day 1,093, Day 1,177, Day 1,261, Day 1,345, Day 1,457
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Days
  BL (Day 0) for Day 365 Cohort (n=360, 153) | 13.80 (10.98) | 13.21 (12.64)
  BL (Day 0) for Day 449 Cohort (n=348, 150) | 13.82 (10.92) | 13.19 (12.65)
  BL (Day 0) for Day 533 Cohort (n=338, 148) | 13.91 (11.06) | 13.55 (12.70)
  BL (Day 0) for Day 617 Cohort (n=332, 140) | 14.01 (11.10) | 13.23 (12.72)
  BL (Day 0) for Day 729 Cohort (n=316, 138) | 13.96 (11.11) | 13.52 (12.78)
  BL (Day 0) for Day 813 Cohort (n=306, 133) | 14.31 (11.14) | 13.38 (12.88)
  BL (Day 0) for Day 897 Cohort (n=302, 131) | 14.08 (11.14) | 13.81 (12.91)
  BL (Day 0) for Day 981 Cohort (n=300, 129) | 14.13 (11.19) | 13.70 (13.03)
  BL (Day 0) for Day 1,093 Cohort (n=292, 130) | 14.34 (11.15) | 13.79 (12.95)
  BL (Day 0) for Day 1,177 Cohort (n=259, 118) | 14.53 (11.17) | 13.80 (13.28)
  BL (Day 0) for Day 1,261 Cohort (n=231, 105) | 15.00 (11.01) | 13.81 (13.16)
  BL (Day 0) for Day 1,345 Cohort (n=133, 57) | 15.71 (11.20) | 15.05 (11.29)
  BL (Day 0) for Day 1,457 Cohort (n=196, 84) | 15.36 (11.16) | 14.87 (13.96)

99. Secondary Outcome: Mean Change From BL in Limitations on Activities of Daily Living in the OL Period
Description: The mean change from baseline in limitations on activities of daily living in the OL period. Activity limitation was measured by the number of days in the past 30 days a participant was unable to perform usual activities due to RA.
Time Frame: as for outcome 98
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Days
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Days
  Day 365 (n=360, 153) | -9.04 (0.60) | -6.39 (1.04)
  Day 449 (n=348, 150) | -8.75 (0.58) | -8.60 (1.03)
  Day 533 (n=338, 148) | -9.21 (0.61) | -9.00 (1.12)
  Day 617 (n=332, 140) | -9.49 (0.63) | -8.62 (1.18)
  Day 729 (n=316, 138) | -9.55 (0.62) | -8.18 (1.21)
  Day 813 (n=306, 133) | -9.87 (0.64) | -8.67 (1.19)
  Day 897 (n=302, 131) | -9.35 (0.65) | -9.22 (1.28)
  Day 981 (n=300, 129) | -9.48 (0.66) | -8.68 (1.26)
  Day 1,093 (n=292, 130) | -10.1 (0.69) | -8.71 (1.25)
  Day 1,177 (n=259, 118) | -10.6 (0.68) | -8.39 (1.34)
  Day 1,261 (n=231, 105) | -9.96 (0.73) | -8.30 (1.51)
  Day 1,345 (n=133, 57) | -11.1 (1.02) | -9.18 (1.61)
  Day 1,457 (n=196, 84) | -9.73 (0.94) | -10.3 (1.61)

100. Primary Outcome: Mean BL White Blood Cells in the OL Period
Description: Mean baseline values are those that are reported for each cohort at each time point on Day 365 to Day 2,185.
Time Frame: BL (Day 0), Day 365, Day 729, Day 1,093, Day 1,457, Day 1,821, Day 1,905, Day 1,989, Day 2,073, Day 2,185
Population: as for outcome 73
Measure: Mean (Standard Deviation); unit: 10^3 c/uL
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 378 | 161
10^3 c/uL
  White Blood Cells Day 365 (n=365, 157) | 8.78 (2.83) | 8.81 (3.01)
  Absolute Neutrophils Day 365 (n=365, 157) | 6.45 (2.63) | 6.39 (2.67)
  Absolute Eosinophils Day 365 (n=365, 157) | 0.18 (0.16) | 0.18 (0.12)
  Absolute Monocytes Day 365 (n=365, 157) | 0.42 (0.25) | 0.41 (0.26)
  White Blood Cells Day 729 (n=328, 143) | 8.89 (2.87) | 8.73 (2.96)
  Absolute Neutrophils Day 729 (n=328, 143) | 6.50 (2.63) | 6.35 (2.66)
  Absolute Eosinophils Day 729 (n=328, 143) | 0.18 (0.16) | 0.18 (0.12)
  Absolute Monocytes Day 729 (n=328, 143) | 0.43 (0.25) | 0.40 (0.25)
  White Blood Cells Day 1,093 (n=312, 138) | 8.81 (2.83) | 8.80 (3.08)
  Absolute Neutrophils Day 1,093 (n=312, 138) | 6.46 (2.63) | 6.37 (2.71)
  Absolute Eosinophils Day 1,093 (n=312, 138) | 0.18 (0.16) | 0.18 (0.12)
  Absolute Monocytes Day 1,093 (n=312, 138) | 0.43 (0.25) | 0.41 (0.27)
  White Blood Cells Day 1,457 (n=292, 130) | 8.80 (2.81) | 8.74 (3.10)
  Absolute Neutrophils Day 1,457 (n=292, 130) | 6.43 (2.59) | 6.32 (2.73)
  Absolute Eosinophils Day 1,457 (n=292, 130) | 0.18 (0.17) | 0.18 (0.12)
  Absolute Monocytes Day 1,457 (n=292, 130) | 0.43 (0.25) | 0.40 (0.25)
  White Blood Cells Day 1,821 (n=262,124) | 8.82 (2.76) | 8.70 (3.06)
  Absolute Neutrophils Day 1,821 (n=262,124) | 6.45 (2.56) | 6.35 (2.72)
  Absolute Eosinophils Day 1,821 (n=262,124) | 0.18 (0.16) | 0.18 (0.12)
  Absolute Monocytes Day 1,821 (n=262,124) | 0.42 (0.24) | 0.39 (0.22)
  White Blood Cells Day 1,905 (n=134, 68) | 9.14 (2.83) | 8.80 (2.91)
  Absolute Neutrophils Day 1,905 (n=134, 68) | 6.78 (2.67) | 6.56 (2.68)
  Absolute Eosinophils Day 1,905 (n=134, 68) | 0.17 (0.16) | 0.16 (0.11)
  Absolute Monocytes Day 1,905 (n=134, 68) | 0.37 (0.21) | 0.34 (0.19)
  White Blood Cells Day 1,989 (n=121,56) | 9.16 (2.87) | 8.81 (2.93)
  Absolute Neutrophils Day 1,989 (n=121,56) | 6.86 (2.77) | 6.69 (2.74)
  Absolute Eosinophils Day 1,989 (n=121,56) | 0.15 (0.14) | 0.15 (0.10)
  Absolute Monocytes Day 1,989 (n=121,56) | 0.35 (0.21) | 0.35 (0.18)
  White Blood Cells Day 2,073 (n=81,38) | 9.64 (3.05) | 9.22 (3.12)
  Absolute Neutrophils Day 2,073 (n=81,38) | 7.25 (2.90) | 6.97 (2.99)
  Absolute Eosinophils Day 2,073 (n=81,38) | 0.12 (0.10) | 0.13 (0.09)
  Absolute Monocytes Day 2,073 (n=81,38) | 0.41 (0.22) | 0.38 (0.19)
  White Blood Cells Day 2,185 (n=82,37) | 9.73 (2.98) | 9.22 (3.16)
  Absolute Neutrophils Day 2,185 (n=82,37) | 7.35 (2.84) | 6.93 (3.03)
  Absolute Eosinophils Day 2,185 (n=82,37) | 0.12 (0.11) | 0.13 (0.09)
  Absolute Monocytes Day 2,185 (n=82,37) | 0.40 (0.22) | 0.38 (0.20)

101. Primary Outcome: Mean Change From BL in White Blood Cells in the OL Period
Description: All changes in participant laboratory parameters were monitored on each day of study drug administration.
Time Frame: BL (Day 0), Day 365, Day 729, Day 1,093, Day 1,457, Day 1,821, Day 1,905, Day 1,989, Day 2,073, Day 2,185
Population: as for outcome 73
Measure: Mean (Standard Error); unit: 10^3 c/uL
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 378 | 161
10^3 c/uL
  White Blood Cells Day 365 (n=365, 157) | -.10 (0.13) | -0.44 (0.17)
  Absolute Neutrophils Day 365 (n=365, 157) | -1.20 (0.12) | -0.43 (0.18)
  Absolute Eosinophils Day 365 (n=365, 157) | -0.02 (0.01) | -0.01 (0.01)
  Absolute Monocytes Day 365 (n=365, 157) | -0.03 (0.01) | -0.03 (0.02)
  White Blood Cells Day 729 (n=328, 143) | -1.35 (0.15) | -1.19 (0.20)
  Absolute Neutrophils Day 729 (n=328, 143) | -1.50 (0.14) | -1.49 (0.19)
  Absolute Eosinophils Day 729 (n=328, 143) | -0.02 (0.01) | -0.04 (0.01)
  Absolute Monocytes Day 729 (n=328, 143) | -0.06 (0.02) | -0.03 (0.02)
  White Blood Cells Day 1,093 (n=312, 138) | -1.50 (0.16) | -1.55 (0.22)
  Absolute Neutrophils Day 1,093 (n=312, 138) | -1.57 (0.15) | -1.66 (0.22)
  Absolute Eosinophils Day 1,093 (n=312, 138) | -0.01 (0.01) | -0.01 (0.01)
  Absolute Monocytes Day 1,093 (n=312, 138) | -0.07 (0.02) | -0.08 (0.02)
  White Blood Cells Day 1,457 (n=292, 130) | -1.36 (0.16) | -1.62 (0.25)
  Absolute Neutrophils Day 1,457 (n=292, 130) | -1.44 (0.15) | -1.68 (0.24)
  Absolute Eosinophils Day 1,457 (n=292, 130) | -0.00 (0.01) | 0.01 (0.02)
  Absolute Monocytes Day 1,457 (n=292, 130) | -0.06 (0.02) | -0.07 (0.02)
  White Blood Cells Day 1,821 (n=262,124) | -1.56 (0.18) | -1.71 (0.24)
  Absolute Neutrophils Day 1,821 (n=262,124) | -1.72 (0.17) | -1.92 (0.23)
  Absolute Eosinophils Day 1,821 (n=262,124) | -0.00 (0.01) | 0.01 (0.02)
  Absolute Monocytes Day 1,821 (n=262,124) | -0.03 (0.02) | -0.04 (0.02)
  White Blood Cells Day 1,905 (n=134, 68) | -0.82 (0.38) | -1.11 (0.32)
  Absolute Neutrophils Day 1,905 (n=134, 68) | -1.30 (0.31) | -1.53 (0.33)
  Absolute Eosinophils Day 1,905 (n=134, 68) | -0.00 (0.02) | -0.02 (0.02)
  Absolute Monocytes Day 1,905 (n=134, 68) | 0.03 (0.02) | 0.05 (0.03)
  White Blood Cells Day 1,989 (n=121,56) | -1.07 (0.26) | -0.97 (0.30)
  Absolute Neutrophils Day 1,989 (n=121,56) | -.152 (0.26) | -1.47 (0.33)
  Absolute Eosinophils Day 1,989 (n=121,56) | 0.01 (0.02) | -0.00 (0.02)
  Absolute Monocytes Day 1,989 (n=121,56) | 0.03 (0.02) | 0.03 (0.03)
  White Blood Cells Day 2,073 (n=81,38) | -1.00 (0.33) | -1.54 (0.44)
  Absolute Neutrophils Day 2,073 (n=81,38) | -1.57 (0.35) | -2.17 (0.47)
  Absolute Eosinophils Day 2,073 (n=81,38) | 0.02 (0.01) | 0.04 (0.02)
  Absolute Monocytes Day 2,073 (n=81,38) | 0.13 (0.03) | 0.11 (0.04)
  White Blood Cells Day 2,185 (n=82,37) | -1.41 (0.33) | -1.96 (0.39)
  Absolute Neutrophils Day 2,185 (n=82,37) | -1.78 (0.33) | -2.39 (0.43)
  Absolute Eosinophils Day 2,185 (n=82,37) | 0.03 (0.02) | -0.01 (0.02)
  Absolute Monocytes Day 2,185 (n=82,37) | 0.08 (0.04) | 0.08 (0.04)

102. Primary Outcome: Mean BL Liver Function Parameters in the OL Period
Description: Mean baseline values are those that are reported for each cohort at each time point on Day 365 to Day 2,185.
Time Frame: BL (Day 0), Day 365, Day 729, Day 1,093, Day 1,457, Day 1,821, Day 1,905, Day 1,989, Day 2,073, Day 2,185
Population: as for outcome 73
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 378 | 161
U/L
  Alkaline Phosphatase Day 365 (n=365, 157) | 99.56 (37.11) | 98.73 (41.23)
  Alanine Aminotransferase Day 365 (n=365, 157) | 22.35 (22.07) | 23.40 (27.35)
  Aspartate Aminotransferase Day 365 (n=365, 157) | 21.53 (12.00) | 22.87 (15.14)
  G-Glutamyl Transferase Day 365 (n=365, 157) | 34.89 (32.59) | 30.73 (26.54)
  Alkaline Phosphatase Day 729 (n=328, 143) | 98.30 (35.22) | 99.49 (41.24)
  Alanine Aminotransferase Day 729 (n=328, 143) | 22.74 (22.91) | 23.21 (28.38)
  Aspartate Aminotransferase Day 729 (n=328, 143) | 21.62 (12.35) | 22.87 (15.50)
  G-Glutamyl Transferase Day 729 (n=328, 143) | 35.37 (33.62) | 28.73 (19.92)
  Alkaline Phosphatase Day 1,093 (n=312, 138) | 99.18 (34.95) | 99.43 (40.80)
  Alanine Aminotransferase Day 1,093 (n=312, 138) | 22.75 (23.38) | 23.01 (28.87)
  Aspartate Aminotransferase Day 1,093 (n=312, 138) | 21.60 (12.55) | 22.91 (15.69)
  G-Glutamyl Transferase Day 1,093 (n=312, 138) | 34.34 (29.93) | 28.43 (20.15)
  Alkaline Phosphatase Day 1,457 (n=292, 130) | 100.8 (36.04) | 99.75 (41.90)
  Alanine Aminotransferase Day 1,457 (n=292, 130) | 23.05 (23.95) | 23.43 (29.67)
  Aspartate Aminotransferase Day 1,457 (n=292, 130) | 21.88 (12.84) | 23.29 (16.08)
  G-Glutamyl Transferase Day 1,457 (n=292, 130) | 35.80 (34.83) | 28.34 (20.35)
  Alkaline Phosphatase Day 1,821 (n=262,124) | 99.80 (34.22) | 97.68 (33.66)
  Alanine Aminotransferase Day 1,821 (n=262,124) | 23.22 (24.74) | 23.55 (30.34)
  Aspartate Aminotransferase Day 1,821 (n=262,124) | 21.63 (12.98) | 23.50 (16.37)
  G-Glutamyl Transferase Day 1,821 (n=262,124) | 35.50 (34.74) | 27.76 (19.77)
  Alkaline Phosphatase Day 1,905 (n=134, 68) | 97.33 (35.95) | 92.19 (35.33)
  Alanine Aminotransferase Day 1,905 (n=134, 68) | 22.57 (22.33) | 25.65 (39.19)
  Aspartate Aminotransferase Day 1,905 (n=134, 68) | 21.43 (12.21) | 24.60 (20.64)
  G-Glutamyl Transferase Day 1,905 (n=134, 68) | 35.08 (31.28) | 30.01 (22.38)
  Alkaline Phosphatase Day 1,989 (n=121,56) | 97.46 (35.63) | 95.18 (36.81)
  Alanine Aminotransferase Day 1,989 (n=121,56) | 23.15 (23.24) | 27.80 (42.76)
  Aspartate Aminotransferase Day 1,989 (n=121,56) | 21.55 (12.72) | 25.82 (22.44)
  G-Glutamyl Transferase Day 1,989 (n=121,56) | 35.27 (32.43) | 31.39 (23.44)
  Alkaline Phosphatase Day 2,073 (n=81,38) | 86.87 (30.05) | 78.53 (22.77)
  Alanine Aminotransferase Day 2,073 (n=81,38) | 22.34 (24.62) | 27.50 (50.75)
  Aspartate Aminotransferase Day 2,073 (n=81,38) | 20.93 (12.70) | 25.37 (26.59)
  G-Glutamyl Transferase Day 2,073 (n=81,38) | 35.62 (37.07) | 30.47 (21.40)
  Alkaline Phosphatase Day 2,185 (n=82,37) | 87.33 (30.52) | 78.97 (22.92)
  Alanine Aminotransferase Day 2,185 (n=82,37) | 22.51 (24.78) | 27.82 (51.41)
  Alanine Aminotransferase Day 2,185 (n=82,37) | 20.80 (12.29) | 25.81 (26.81)
  G-Glutamyl Transferase Day 2,185 (n=82,37) | 36.23 (37.42) | 30.46 (21.69)

103. Primary Outcome: Mean Change From BL in Liver Function Parameters in the OL Period
Description: All changes in participant laboratory parameters were monitored on each day of study drug administration.
Time Frame: BL (Day 0), Day 365, Day 729, Day 1,093, Day 1,457, Day 1,821, Day 1,905, Day 1,989, Day 2,073, Day 2,185
Population: as for outcome 73
Measure: Mean (Standard Error); unit: U/L
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 378 | 161
U/L
  Alkaline Phosphatase Day 365 (n=365, 157) | -7.27 (1.60) | -10.8 (2.30)
  Alanine Aminotransferase Day 365 (n=365, 157) | 1.10 (1.25) | -2.64 (2.18)
  Aspartate Aminotransferase Day 365 (n=365, 157) | 1.50 (0.76) | -1.42 (1.20)
  G-Glutamyl Transferase Day 365 (n=365, 157) | -4.42 (1.48) | -2.83 (1.79)
  Alkaline Phosphatase Day 729 (n=328, 143) | -13.3 (1.70) | -18.8 (2.85)
  Alanine Aminotransferase Day 729 (n=328, 143) | 0.39 (1.39) | -1.69 (2.38)
  Aspartate Aminotransferase Day 729 (n=328, 143) | 1.30 (0.83) | 0.47 (1.43)
  G-Glutamyl Transferase Day 729 (n=328, 143) | -4.96 (1.62) | -3.98 (1.68)
  Alkaline Phosphatase Day 1,093 (n=312, 138) | -10.0 (1.69) | -13.0 (2.74)
  Alanine Aminotransferase Day 1,093 (n=312, 138) | 0.81 (1.40) | -0.17 (2.52)
  Aspartate Aminotransferase Day 1,093 (n=312, 138) | 1.11 (0.85) | 0.07 (1.39)
  G-Glutamyl Transferase Day 1,093 (n=312, 138) | -6.81 (1.55) | -4.51 (1.54)
  Alkaline Phosphatase Day 1,457 (n=292, 130) | -12.4 (1.73) | -12.0 (3.02)
  Alanine Aminotransferase Day 1,457 (n=292, 130) | 1.43 (2.66) | -3.11 (2.57)
  Aspartate Aminotransferase Day 1,457 (n=292, 130) | 1.40 (1.73) | -1.82 (1.40)
  G-Glutamyl Transferase Day 1,457 (n=292, 130) | -5.15 (2.35) | -3.66 (1.54)
  Alkaline Phosphatase Day 1,821 (n=262,124) | -14.6 (1.70) | -14.7 (1.99)
  Alanine Aminotransferase Day 1,821 (n=262,124) | -0.95 (1.49) | -0.75 (2.65)
  Aspartate Aminotransferase Day 1,821 (n=262,124) | 0.14 (0.85) | -0.52 (1.52)
  G-Glutamyl Transferase Day 1,821 (n=262,124) | -5.63 (2.04) | -4.65 (1.55)
  Alkaline Phosphatase Day 1,905 (n=134, 68) | -14.9 (2.82) | -10.6 (3.19)
  Alanine Aminotransferase Day 1,905 (n=134, 68) | -2.35 (2.03) | -5.74 (4.66)
  Aspartate Aminotransferase Day 1,905 (n=134, 68) | -0.49 (1.18) | -3.00 (2.46)
  G-Glutamyl Transferase Day 1,905 (n=134, 68) | -6.76 (3.16) | -3.09 (2.91)
  Alkaline Phosphatase Day 1,989 (n=121,56) | -12.4 (2.80) | -13.0 (3.80)
  Alanine Aminotransferase Day 1,989 (n=121,56) | -1.41 (2.04) | -4.98 (5.60)
  Aspartate Aminotransferase Day 1,989 (n=121,56) | 0.20 (1.24) | -1.71 (2.98)
  G-Glutamyl Transferase Day 1,989 (n=121,56) | -3.66 (3.58) | -4.00 (2.95)
  Alkaline Phosphatase Day 2,073 (n=81,38) | -10.6 (3.40) | -4.24 (3.57)
  Alanine Aminotransferase Day 2,073 (n=81,38) | -0.56 (2.82) | -8.08 (7.91)
  Aspartate Aminotransferase Day 2,073 (n=81,38) | 0.95 (1.68) | -2.37 (4.26)
  G-Glutamyl Transferase Day 2,073 (n=81,38) | -10.2 (4.23) | -4.92 (3.49)
  Alkaline Phosphatase Day 2,185 (n=82,37) | -14.2 (2.79) | -7.76 (3.40)
  Alanine Aminotransferase Day 2,185 (n=82,37) | -2.56 (2.84) | -7.43 (8.65)
  Alanine Aminotransferase Day 2,185 (n=82,37) | 0.60 (1.60) | -1.43 (4.64)
  G-Glutamyl Transferase Day 2,185 (n=82,37) | -13.9 (3.81) | -4.51 (2.95)

104. Primary Outcome: Mean BL Select Laboratory Parameters in the OL Period
Description: Mean baseline values are those that are reported for each cohort at each time point on Day 365 to Day 2,185.
Time Frame: BL (Day 0), Day 365, Day 729, Day 1,093, Day 1,457, Day 1,821, Day 1,905, Day 1,989, Day 2,073, Day 2,185
Population: as for outcome 73
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 378 | 161
mg/dL
  Total Bilirubin Day 365 (n=365, 157) | 0.42 (0.18) | 0.48 (0.23)
  Blood Urea Nitrogen (BUN) Day 365 (n=365, 157) | 16.05 (5.19) | 15.09 (4.41)
  Creatinine Day 365 (n=365, 157) | 0.74 (0.17) | 0.74 (0.17)
  Serum Calcium Day 365 (n=365, 157) | 9.26 (0.44) | 9.26 (0.50)
  Inorganic Phosphorous Day 365 (n=365, 157) | 3.48 (0.57) | 3.56 (0.54)
  Serum Glucose Day 365 (n=365, 157) | 96.63 (29.30) | 98.78 (58.76)
  Uric Acid Day 365 (n=365, 157) | 4.80 (1.45) | 4.83 (1.50)
  Total Bilirubin Day 729 (n=328, 143) | 0.42 (0.18) | 0.48 (0.23)
  BUN Day 729 (n=328, 143) | 16.02 (5.23) | 15.03 (4.40)
  Creatinine Day 729 (n=328, 143) | 0.74 (0.18) | 0.73 (0.17)
  Serum Calcium Day 729 (n=328, 143) | 9.26 (0.44) | 9.24 (0.50)
  Inorganic Phosphorous Day 729 (n=328, 143) | 3.50 (0.57) | 3.55 (0.50)
  Serum Glucose Day 729 (n=328, 143) | 97.36 (30.59) | 98.56 (60.79)
  Uric Acid Day 729 (n=328, 143) | 4.79 (1.41) | 4.75 (1.34)
  Total Bilirubin Day 1,093 (n=312, 138) | 0.42 (0.18) | 0.48 (0.22)
  BUN Day 1,093 (n=312, 138) | -0.36 (0.26) | 0.00 (0.40)
  Creatinine Day 1,093 (n=312, 138) | 0.73 (0.17) | 0.74 (0.17)
  Serum Calcium Day 1,093 (n=312, 138) | 0.04 (0.03) | 0.02 (0.04)
  Inorganic Phosphorous Day 1,093 (n=312, 138) | 0.02 (0.04) | 0.10 (0.05)
  Serum Glucose Day 1,093 (n=312, 138) | 96.49 (29.70) | 97.65 (61.54)
  Uric Acid Day 1,093 (n=312, 138) | -0.15 (0.06) | -0.32 (0.09)
  Total Bilirubin Day 1,457 (n=292, 130) | 0.42 (0.18) | 0.49 (0.23)
  BUN Day 1,457 (n=292, 130) | 15.86 (5.28) | 15.02 (4.36)
  Creatinine Day 1,457 (n=292, 130) | 0.73 (0.17) | 0.74 (0.18)
  Serum Calcium Day 1,457 (n=292, 130) | 9.26 (0.45) | 9.25 (0.46)
  Inorganic Phosphorous Day 1,457 (n=292, 130) | 3.49 (0.54) | 3.54 (0.50)
  Serum Glucose Day 1,457 (n=292, 130) | 95.81 (28.90) | 95.35 (55.47)
  Uric Acid Day 1,457 (n=292, 130) | 4.73 (1.40) | 4.75 (1.32)
  Total Bilirubin Day Day 1,821 (n=262,124) | 0.42 (0.18) | 0.50 (0.23)
  BUN Day 1,821 (n=262,124) | 15.93 (5.29) | 14.88 (3.96)
  Creatinine Day 1,821 (n=262,124) | 0.73 (0.16) | 0.74 (0.18)
  Serum Calcium Day 1,821 (n=262,124) | 9.25 (0.45) | 9.25 (0.46)
  Inorganic Phosphorous Day 1,821 (n=262,124) | 3.49 (0.53) | 3.54 (0.51)
  Serum Glucose Day 1,821 (n=262,124) | 96.81 (30.21) | 98.59 (64.79)
  Uric Acid Day 1,821 (n=262,124) | 4.66 (1.29) | 4.68 (1.31)
  Total Bilirubin Day 1,905 (n=134, 68) | 0.43 (0.18) | 0.50 (0.25)
  BUN Day 1,905 (n=134, 68) | 16.15 (5.74) | 14.77 (3.78)
  Creatinine Day 1,905 (n=134, 68) | 0.72 (0.16) | 0.75 (0.16)
  Serum Calcium Day 1,905 (n=134, 68) | 9.30 (0.45) | 9.30 (0.40)
  Inorganic Phosphorous Day 1,905 (n=134, 68) | 3.50 (0.56) | 3.44 (0.52)
  Serum Glucose Day 1,905 (n=134, 68) | 96.82 (31.18) | 101.1 (74.67)
  Uric Acid Day 1,905 (n=134, 68) | 4.70 (1.25) | 4.93 (1.30)
  Total Bilirubin Day 1,989 (n=121,56) | 0.43 (0.18) | 0.52 (0.27)
  BUN Day 1,989 (n=121,56) | 16.26 (5.68) | 15.18 (3.88)
  Creatinine Day 1,989 (n=121,56) | 0.71 (0.14) | 0.72 (0.15)
  Serum Calcium Day 1,989 (n=121,56) | 9.31 (0.44) | 9.33 (0.42)
  Inorganic Phosphorous Day 1,989 (n=121,56) | 3.51 (0.57) | 3.45 (0.53)
  Serum Glucose Day 1,989 (n=121,56) | 98.59 (33.41) | 104.80 (81.64)
  Uric Acid Day 1,989 (n=121,56) | 4.72 (1.25) | 4.99 (1.36)
  Total Bilirubin Day 2,073 (n=81,38) | 0.42 (0.19) | 0.52 (0.30)
  BUN Day 2,073 (n=81,38) | 16.36 (5.83) | 15.27 (3.91)
  Creatinine Day 2,073 (n=81,38) | 0.68 (0.13) | 0.69 (0.13)
  Serum Calcium Day 2,073 (n=81,38) | 9.41 (0.36) | 9.48 (0.38)
  Inorganic Phosphorous Day 2,073 (n=81,38) | 3.61 (0.58) | 3.52 (0.60)
  Serum Glucose Day 2,073 (n=81,38) | 100.4 (31.96) | 111.1 (97.97)
  Uric Acid Day 2,073 (n=81,38) | 4.58 (1.19) | 4.60 (1.37)
  Total Bilirubin Day 2,185 (n=82,37) | 0.42 (0.18) | 0.52 (0.30)
  BUN Day 2,185 (n=82,37) | 16.40 (5.86) | 15.22 (3.95)
  Creatinine Day 2,185 (n=82,37) | 0.68 (0.13) | 0.69 (0.13)
  Serum Calcium Day 2,185 (n=82,37) | 9.43 (0.41) | 9.48 (0.38)
  Inorganic Phosphorous Day 2,185 (n=82,37) | 3.58 (0.58) | 3.54 (0.61)
  Serum Glucose Day 2,185 (n=82,37) | 99.29 (30.71) | 111.4 (99.31)
  Uric Acid Day 2,185 (n=82,37) | 4.61 (1.22) | 4.60 (1.39)

105. Primary Outcome: Mean Change From BL in Select Laboratory Parameters in the OL Period
Description: All changes in participant laboratory parameters were monitored on each day of study drug administration.
Time Frame: BL (Day 0), Day 365, Day 729, Day 1,093, Day 1,457, Day 1,821, Day 1,905, Day 1,989, Day 2,073, Day 2,185
Population: as for outcome 73
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 378 | 161
mg/dL
  Total Bilirubin Day 365 (n=365, 157) | 0.06 (0.01) | 0.00 (0.01)
  Blood Urea Nitrogen (BUN) Day 365 (n=365, 157) | 16.05 (5.19) | 15.09 (4.41)
  Creatinine Day 365 (n=365, 157) | 0.74 (0.17) | 0.74 (0.17)
  Serum Calcium Day 365 (n=365, 157) | 0.25 (0.02) | 0.22 (0.04)
  Inorganic Phosphorous Day 365 (n=365, 157) | -0.02 (0.03) | -0.12 (0.04)
  Serum Glucose Day 365 (n=365, 157) | -1.65 (1.26) | -4.06 (4.29)
  Uric Acid Day 365 (n=365, 157) | 0.04 (0.05) | -0.06 (0.07)
  Total Bilirubin Day 729 (n=328, 143) | 0.09 (0.01) | 0.05 (0.02)
  BUN Day 729 (n=328, 143) | -0.38 (0.31) | -0.06 (0.35)
  Creatinine Day 729 (n=328, 143) | 0.08 (0.01) | 0.08 (0.01)
  Serum Calcium Day 729 (n=328, 143) | 0.14 (0.03) | 0.18 (0.05)
  Inorganic Phosphorous Day 729 (n=328, 143) | -0.06 (0.03) | -0.10 (0.05)
  Serum Glucose Day 729 (n=328, 143) | -1.77 (1.67) | -4.74 (5.18)
  Uric Acid Day 729 (n=328, 143) | 0.11 (0.06) | 0.00 (0.09)
  Total Bilirubin Day 1,093 (n=312, 138) | 0.05 (0.01) | 0.01 (0.02)
  BUN Day 1,093 (n=312, 138) | -0.36 (0.26) | 0.00 (0.40)
  Creatinine Day 1,093 (n=312, 138) | -0.00 (0.01) | -0.03 (0.01)
  Serum Calcium Day 1,093 (n=312, 138) | 0.04 (0.03) | 0.02 (0.04)
  Inorganic Phosphorous Day 1,093 (n=312, 138) | 0.02 (0.04) | 0.10 (0.05)
  Serum Glucose Day 1,093 (n=312, 138) | 0.36 (1.63) | -4.95 (4.84)
  Uric Acid Day 1,093 (n=312, 138) | -0.15 (0.06) | -0.32 (0.09)
  Total Bilirubin Day 1,457 (n=292, 130) | 0.01 (0.01) | -0.04 (0.02)
  BUN Day 1,457 (n=292, 130) | -0.48 (0.27) | -0.47 (0.42)
  Creatinine Day 1,457 (n=292, 130) | 0.02 (0.01) | -0.03 (0.01)
  Serum Calcium Day 1,457 (n=292, 130) | -0.08 (0.03) | -0.08 (0.04)
  Inorganic Phosphorous Day 1,457 (n=292, 130) | -0.00 (0.04) | 0.02 (0.05)
  Serum Glucose Day 1,457 (n=292, 130) | 0.43 (1.53) | -0.12 (5.09)
  Uric Acid Day 1,457 (n=292, 130) | -0.19 (0.06) | -0.43 (0.09)
  Total Bilirubin Day Day 1,821 (n=262,124) | 0.01 (0.01) | -0.01 (0.04)
  BUN Day 1,821 (n=262,124) | -0.54 (0.28) | 0.30 (0.44)
  Creatinine Day 1,821 (n=262,124) | -0.01 (0.01) | -0.04 (0.02)
  Serum Calcium Day 1,821 (n=262,124) | -0.07 (0.03) | -0.04 (0.04)
  Inorganic Phosphorous Day 1,821 (n=262,124) | 0.02 (0.04) | 0.01 (0.05)
  Serum Glucose Day 1,821 (n=262,124) | 3.27 (1.86) | -0.02 (5.51)
  Uric Acid Day 1,821 (n=262,124) | -0.13 (0.06) | -0.30 (0.09)
  Total Bilirubin Day 1,905 (n=134, 68) | 0.01 (0.02) | -0.05 (0.04)
  BUN Day 1,905 (n=134, 68) | -0.36 (0.39) | 0.56 (0.57)
  Creatinine Day 1,905 (n=134, 68) | -0.04 (0.01) | -0.03 (0.02)
  Serum Calcium Day 1,905 (n=134, 68) | -0.12 (0.04) | -0.11 (0.05)
  Inorganic Phosphorous Day 1,905 (n=134, 68) | -0.03 (0.06) | 0.11 (0.08)
  Serum Glucose Day 1,905 (n=134, 68) | 3.00 (2.96) | -0.50 (9.71)
  Uric Acid Day 1,905 (n=134, 68) | -0.29 (0.09) | -0.29 (0.12)
  Total Bilirubin Day 1,989 (n=121,56) | 0.01 (0.02) | -0.03 (0.03)
  BUN Day 1,989 (n=121,56) | -0.31 (0.45) | 0.09 (0.64)
  Creatinine Day 1,989 (n=121,56) | -0.01 (0.01) | -0.02 (0.02)
  Serum Calcium Day 1,989 (n=121,56) | -0.10 (0.04) | -0.08 (0.05)
  Inorganic Phosphorous Day 1,989 (n=121,56) | -0.07 (0.06) | 0.08 (0.08)
  Serum Glucose Day 1,989 (n=121,56) | -1.58 (2.85) | -2.70 (11.88)
  Uric Acid Day 1,989 (n=121,56) | -0.29 (0.09) | -0.38 (0.14)
  Total Bilirubin Day 2,073 (n=81,38) | 0.04 (0.02) | -0.100 (0.04)
  BUN Day 2,073 (n=81,38) | 0.33 (0.47) | 0.84 (0.72)
  Creatinine Day 2,073 (n=81,38) | 0.05 (0.01) | 0.04 (0.03)
  Serum Calcium Day 2,073 (n=81,38) | -0.10 (0.04) | -0.20 (0.08)
  Inorganic Phosphorous Day 2,073 (n=81,38) | -0.11 (0.07) | -0.11 (0.12)
  Serum Glucose Day 2,073 (n=81,38) | -0.74 (3.13) | -18.2 (16.92)
  Uric Acid Day 2,073 (n=81,38) | -0.08 (0.11) | -0.15 (0.16)
  Total Bilirubin Day 2,185 (n=82,37) | 0.05 (0.02) | 0.00 (0.04)
  BUN Day 2,185 (n=82,37) | 0.51 (0.53) | 0.18 (0.56)
  Creatinine Day 2,185 (n=82,37) | 0.03 (0.01) | 0.04 (0.02)
  Serum Calcium Day 2,185 (n=82,37) | -0.27 (0.04) | -0.19 (0.07)
  Inorganic Phosphorous Day 2,185 (n=82,37) | -0.14 (0.07) | -0.13 (0.13)
  Serum Glucose Day 2,185 (n=82,37) | 6.85 (3.81) | -8.86 (17.98)
  Uric Acid Day 2,185 (n=82,37) | -0.12 (0.10) | -0.17 (0.14)

106. Primary Outcome: Mean BL Serum Electrolytes in the OL Period
Description: Mean baseline values are those that are reported for each cohort at each time point on Day 365 to Day 2,185.
Time Frame: BL (Day 0), Day 365, Day 729, Day 1,093, Day 1,457, Day 1,821, Day 1,905, Day 1,989, Day 2,073, Day 2,185
Population: as for outcome 73
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 378 | 161
mEq/L
  Serum Sodium Day 365 (n=365, 157) | 139.9 (2.89) | 140.7 (3.03)
  Serum Potassium Day 365 (n=365, 157) | 4.27 (0.37) | 4.29 (0.43)
  Serum Chloride Day 365 (n=365, 157) | 104.1 (3.17) | 105.0 (3.63)
  Serum Sodium Day 729 (n=328, 143) | 139.8 (2.97) | 140.7 (3.06)
  Serum Potassium Day 729 (n=328, 143) | 4.27 (0.36) | 4.30 (0.42)
  Serum Chloride Day 729 (n=328, 143) | 103.9 (3.13) | 104.9 (3.65)
  Serum Sodium Day 1,093 (n=312, 138) | 139.9 (2.88) | 140.7 (3.11)
  Serum Potassium Day 1,093 (n=312, 138) | 4.27 (0.36) | 4.27 (0.39)
  Serum Chloride Day 1,093 (n=312, 138) | 104.0 (3.08) | 104.9 (3.64)
  Serum Sodium Day 1,457 (n=292, 130) | 139.9 (2.83) | 140.7 (3.16)
  Serum Potassium Day 1,457 (n=292, 130) | 4.27 (0.35) | 4.27 (0.38)
  Serum Chloride Day 1,457 (n=292, 130) | 104.0 (3.06) | 105.0 (3.64)
  Serum Sodium Day 1,821 (n=262,124) | 140.0 (2.84) | 140.7 (3.11)
  Serum Potassium Day 1,821 (n=262,124) | 4.26 (0.36) | 4.28 (0.40)
  Serum Chloride Day 1,821 (n=262,124) | 104.1 (3.08) | 104.8 (3.60)
  Serum Sodium Day 1,905 (n=134, 68) | 139.6 (3.13) | 140.5 (3.56)
  Serum Potassium Day 1,905 (n=134, 68) | 4.25 (0.37) | 4.25 (0.42)
  Serum Chloride Day 1,905 (n=134, 68) | 103.9 (3.44) | 104.9 (4.03)
  Serum Sodium Day 1,989 (n=121,56) | 139.5 (3.14) | 140.1 (3.72)
  Serum Potassium Day 1,989 (n=121,56) | 4.27 (0.41) | 4.24 (0.43)
  Serum Chloride Day 1,989 (n=121,56) | 103.8 (3.61) | 104.8 (4.33)
  Serum Sodium Day 2,073 (n=81,38) | 138.2 (2.33) | 139.0 (3.91)
  Serum Potassium Day 2,073 (n=81,38) | 4.31 (0.44) | 4.27 (0.48)
  Serum Chloride Day 2,073 (n=81,38) | 102.3 (2.57) | 103.0 (4.23)
  Serum Sodium Day 2,185 (n=82,37) | 138.2 (2.31) | 138.9 (3.93)
  Serum Potassium Day 2,185 (n=82,37) | 4.30 (0.43) | 4.28 (0.49)
  Serum Chloride Day 2,185 (n=82,37) | 102.3 (2.51) | 102.9 (4.24)

107. Primary Outcome: Mean Change From BL in Serum Electrolytes in the OL Period
Description: All changes in participant laboratory parameters were monitored on each day of study drug administration.
Time Frame: BL (Day 0), Day 365, Day 729, Day 1,093, Day 1,457, Day 1,821, Day 1,905, Day 1,989, Day 2,073, Day 2,185
Population: as for outcome 73
Measure: Mean (Standard Error); unit: mEq/L
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 378 | 161
mEq/L
  Serum Sodium Day 365 (n=365, 157) | -0.42 (0.17) | -1.37 (0.27)
  Serum Potassium Day 365 (n=365, 157) | -0.01 (0.02) | -0.06 (0.03)
  Serum Chloride Day 365 (n=365, 157) | 0.43 (0.14) | -0.21 (0.25)
  Serum Sodium Day 729 (n=328, 143) | 0.71 (0.19) | -0.29 (0.29)
  Serum Potassium Day 729 (n=328, 143) | -0.03 (0.02) | -0.12 (0.04)
  Serum Chloride Day 729 (n=328, 143) | 0.63 (0.17) | 0.15 (0.27)
  Serum Sodium Day 1,093 (n=312, 138) | -0.29 (0.21) | -1.34 (0.34)
  Serum Potassium Day 1,093 (n=312, 138) | -0.05 (0.02) | -0.08 (0.04)
  Serum Chloride Day 1,093 (n=312, 138) | -0.35 (0.18) | -1.17 (0.31)
  Serum Sodium Day 1,457 (n=292, 130) | -0.18 (0.25) | -0.88 (0.40)
  Serum Potassium Day 1,457 (n=292, 130) | -0.03 (0.03) | -0.08 (0.04)
  Serum Chloride Day 1,457 (n=292, 130) | 104.0 (3.06) | 105.0 (3.64)
  Serum Sodium Day 1,821 (n=262,124) | -0.68 (0.24) | -1.29 (0.38)
  Serum Potassium Day 1,821 (n=262,124) | -0.08 (0.02) | -0.15 (0.04)
  Serum Chloride Day 1,821 (n=262,124) | -0.19 (0.22) | -0.69 (0.34)
  Serum Sodium Day 1,905 (n=134, 68) | -0.27 (0.36) | -0.75 (0.54)
  Serum Potassium Day 1,905 (n=134, 68) | -0.06 (0.04) | -0.06 (0.05)
  Serum Chloride Day 1,905 (n=134, 68) | 0.31 (0.33) | -0.15 (0.53)
  Serum Sodium Day 1,989 (n=121,56) | -0.02 (0.40) | -0.25 (0.66)
  Serum Potassium Day 1,989 (n=121,56) | -0.05 (0.04) | -0.12 (0.06)
  Serum Chloride Day 1,989 (n=121,56) | 0.40 (0.38) | -0.52 (0.60)
  Serum Sodium Day 2,073 (n=81,38) | 2.56 (0.32) | 2.05 (0.71)
  Serum Potassium Day 2,073 (n=81,38) | -0.10 (0.05) | -0.14 (0.08)
  Serum Chloride Day 2,073 (n=81,38) | 2.27 (0.40) | 1.89 (0.72)
  Serum Sodium Day 2,185 (n=82,37) | 2.76 (0.34) | 2.24 (0.68)
  Serum Potassium Day 2,185 (n=82,37) | -0.11 (0.05) | -0.20 (0.08)
  Serum Chloride Day 2,185 (n=82,37) | 2.95 (0.40) | 1.81 (0.72)

108. Secondary Outcome: Mean BL Interleukin-6 (IL-6), SIL-2R, and Tumor Necrosis Alpha (TNF-Alpha) in the DB Period
Description: as for outcome 59
Time Frame: BL (Day 0), Day 169, Day 365
Population: All treated participants in the DB period. N = number of participants analyzed and n = the number of participants with measurements for that time point.
Measure: Mean (Standard Deviation); unit: pg / mL
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
pg / mL
  BL (Day 0) IL-6 for Day 169 Cohort (n=357, 175) | 36.35 (43.53) | 39.90 (54.43)
  BL (Day 0) SIL-2R for Day 169 Cohort (n=370, 171) | 1776 (946.5) | 1603 (933.1)
  BL (Day 0) TNF-Alpha for D169 Cohort (n=354,172) | 5.94 (7.90) | 7.86 (29.41)
  BL (Day 0) IL-6 for Day 365 Cohort (n=247, 121) | 35.27 (49.06) | 37.89 (49.61)
  BL (Day 0) SIL-2R for Day 365 Cohort (n=235, 106) | 1674 (835.1) | 1601 (1076)
  BL (Day 0) TNF-Alpha for D365 Cohort (n=246, 119) | 5.55 (7.84) | 5.46 (8.63)

109. Secondary Outcome: Mean Change From BL in Interleukin-6 (IL-6), SIL-2R, and Tumor Necrosis Alpha (TNF-Alpha) in the DB Period
Description: The mean change from baseline in potential biomarkers of disease (IL-6, SIL-3R, and TNF-Alpha were determined for all participants.
Time Frame: BL (Day 0), Day 169, Day 365
Population: as for outcome 108
Measure: Mean (Standard Error); unit: pg / mL
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 424 | 214
pg / mL
  IL-6 Day 169 (n=357, 175) | -21.0 (2.24) | -5.81 (3.00)
  SIL-2R Day 169 (n=370, 171) | -519.0 (32.72) | -85.5 (32.78)
  TNF-Alpha Day 169 (n=354, 172) | -0.82 (0.72) | 2.27 (2.49)
  IL-6 Day 365 (n=247, 121) | -23.4 (3.08) | -1.82 (5.23)
  SIL-2R Day 365(n=235, 106) | -562 (40.82) | -290 (87.97)
  TNF-Alpha Day 365 (n=246, 119) | -0.22 (1.04) | 1.22 (2.42)

110. Secondary Outcome: Mean Change From BL in RF in the DB Period
Description: The mean change from baseline in participant rheumatoid factor was determined after 6 months and 1 year of treatment relative to baseline. Time-matched BL(Day 0) values and post-BL vales were presented for each post-BL visit and represent only that cohort of participants with measurements available at that post-BL assessment.
Time Frame: BL (Day 0), Day 169, Day 365
Population: as for outcome 108
Measure: Mean (Standard Error); unit: IU / mL
Arm/Group | ABA + MTX DB | Placebo + MTX DB
Number analyzed (Participants) | 424 | 214
IU / mL
  BL (Day 0) for Day 169 Cohort (n=308, 126) | -49.8 (10.90) | -18.6 (10.28)
  BL (Day 0) for Day 365 Cohort (n=281, 104) | -46.5 (11.44) | -5.83 (22.38)

111. Secondary Outcome: Mean BL E-Selectin, SICAM-1, and MMP3 in the DB Period
Description: as for outcome 59
Time Frame: BL (Day 0), Day 169, Day 365
Population: as for outcome 108
Measure: Mean (Standard Error); unit: ng / mL
Arm/Group | ABA + MTX DB | Placebo + MTX DB
Number analyzed (Participants) | 424 | 214
ng / mL
  BL (Day 0) E-Selectin for D169 Cohort (n= 256,126) | 85.89 (72.62) | 85.53 (68.42)
  BL (Day 0) SICAM-1 for D169 Cohort (n=264, 130) | 444.0 (398.1) | 426.8 (323.5)
  BL (Day 0) MMP3 for D169 Cohort (n=362, 183) | 83.37 (81.53) | 77.22 (73.72)
  BL (Day 0) E-Selectin fpr D365 Cohort (n=162, 74) | 85.91 (71.66) | 88.39 (75.09)
  BL (Day 0) SICAM-1 for D365 Cohort (n=235, 114) | 467.2 (578.5) | 449.5 (356.0)
  BL (Day 0) MMP3 for D365 Cohort (n=232, 112) | 79.56 (78.35) | 64.02 (59.05)

112. Secondary Outcome: Mean Change From BL in E-Selectin, SICAM-1, and MMP3 in the DB Period
Description: The mean change from basline in particpant biomarkers of RA disease (E-Selectin, SICAM-1, and MMP3) after 6 months and 1 year of treatment, relative to baseline, were evaluated.
Time Frame: BL (Day 0), Day 169, Day 365
Population: as for outcome 108
Measure: Mean (Standard Error); unit: ng / mL
Arm/Group | ABA + MTX DB | Placebo + MTX DB
Number analyzed (Participants) | 424 | 214
ng / mL
  E-Selectin Day 169 (n= 256, 126) | -13.8 (3.28) | -6.52 (4.44)
  SICAM-1 Day 169 (n=264, 130) | -65.0 (9.87) | -42.0 (17.02)
  MMP3 Day 169 (n=362, 183) | -37.2 (2.85) | -8.03 (3.88)
  E-Selectin Day 365 (n=162, 74) | -15.4 (4.37) | -9.94 (5.73)
  SICAM-1 Day 365 (n=235, 114) | -80.0 (27.20) | -43.7 (16.25)
  MMP3 Day 365 (n=232, 112) | -41.0 (4.09) | -12.1 (5.01)

113. Secondary Outcome: Mean BL HAQ-DI Score and HAQ-DI Individual Component Scores at BL (Day 0) for the Day 365 Cohort of Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 365
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=369, 160) | 1.68 (0.63) | 1.70 (0.58)
  Dressing and Grooming (n=372, 160) | 1.47 (0.75) | 1.49 (0.73)
  Arising (n=372, 160) | 1.42 (0.82) | 1.46 (0.78)
  Eating (n=372, 160) | 1.63 (0.97) | 1.68 (0.84)
  Walking (n=372, 158) | 1.40 (0.83) | 1.37 (0.78)
  Hygiene (n=370, 160) | 1.93 (0.90) | 1.91 (0.89)
  Reaching (n=370, 160) | 1.94 (0.86) | 1.97 (0.80)
  Gripping (n=371, 160) | 1.80 (0.76) | 1.90 (0.67)
  Activities (n=369, 160) | 1.87 (0.79) | 1.86 (0.82)

114. Secondary Outcome: Mean Change From BL in HAQ-DI Score and HAQ-DI Individual Component Scores at Day 365 for Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 365
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=369, 160) | -0.68 (0.03) | -0.51 (0.05)
  Dressing and Grooming (n=372, 160) | -0.77 (0.04) | -0.62 (0.06)
  Arising (n=372, 160) | -0.75 (0.05) | -0.59 (0.07)
  Eating (n=372, 160) | -0.80 (0.05) | -0.46 (0.07)
  Walking (n=372, 158) | -0.62 (0.04) | -0.48 (0.06)
  Hygiene (n=370, 160) | -0.54 (0.05) | -0.36 (0.08)
  Reaching (n=370, 160) | -0.71 (0.05) | -0.60 (0.07)
  Gripping (n=371, 160) | -0.63 (0.05) | -0.49 (0.07)
  Activities (n=369, 160) | -0.66 (0.05) | -0.47 (0.07)

115. Secondary Outcome: Mean BL HAQ-DI Score and HAQ-DI Individual Component Scores at BL (Day 0) for the Day 449 Cohort of Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 449
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=366, 157) | 1.69 (0.64) | 1.71 (0.59)
  Dressing and Grooming (n=367, 157) | 1.48 (0.75) | 1.49 (0.73)
  Arising (n=367, 157) | 1.42 (0.83) | 1.46 (0.79)
  Eating (n=367, 157) | 1.64 (0.97) | 1.67 (0.84)
  Walking (n=367, 155) | 1.40 (0.83) | 1.37 (0.76)
  Hygiene (n=367, 157) | 1.93 (0.90) | 1.92 (0.89)
  Reaching (n= 367, 157) | 1.94 (0.86) | 1.97 (0.80)
  Gripping (n=368, 157) | 1.81 (0.75) | 1.90 (0.67)
  Activities (n=367, 157) | 1.87 (0.79) | 1.87 (0.82)

116. Secondary Outcome: Mean Change From BL in HAQ-DI Score and HAQ-DI Individual Component Scores at Day 449 for Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 449
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=366, 157) | -0.70 (0.03) | -0.71 (0.05)
  Dressing and Grooming (n=367, 157) | -0.78 (0.04) | -0.85 (0.06)
  Arising (n=367, 157) | -0.72 (0.05) | -0.86 (0.07)
  Eating (n=367, 157) | -0.82 (0.05) | -0.63 (0.07)
  Walking (n=367, 155) | -0.60 (0.05) | -0.61 (0.06)
  Hygiene (n=367, 157) | -0.57 (0.05) | -0.59 (0.08)
  Reaching (n= 367, 157) | -0.75 (0.05) | -0.76 (0.07)
  Gripping (n=368, 157) | -0.67 (0.05) | -0.73 (0.08)
  Activities (n=367, 157) | -0.70 (0.05) | -0.65 (0.08)

117. Secondary Outcome: Mean BL HAQ-DI Score and HAQ-DI Individual Component Scores at BL (Day 0) for the Day 533 Cohort of Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 533
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=354, 157) | 1.69 (0.64) | 1.71 (0.58)
  Dressing and Grooming (n=355, 156) | 1.47 (0.75) | 1.49 (0.73)
  Arising (n=355, 157) | 1.42 (0.84) | 1.45 (.078)
  Eating (n=355, 156) | 1.64 (0.98) | 1.67 (0.84)
  Walking (n=351, 156) | 1.40 (0.84) | 1.37 (0.78)
  Hygiene (n=354, 157) | 1.94 (0.91) | 1.92 (0.88)
  Reaching (n=354, 157) | 1.95 (0.86) | 1.97 (0.80)
  Gripping (n=354, 157) | 1.81 (0.76) | 1.91 (0.66)
  Activities (n=354, 157) | 1.88 (0.79) | 1.87 (0.82)

118. Secondary Outcome: Mean Change From BL in HAQ-DI Score and HAQ-DI Individual Component Scores at Day 533 for Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 533
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=354, 157) | -0.73 (0.04) | -0.73 (0.05)
  Dressing and Grooming (n=355, 156) | -0.81 (0.05) | -0.85 (0.06)
  Arising (n=355, 157) | -0.76 (0.05) | -0.86 (0.07)
  Eating (n=355, 156) | -0.83 (0.05) | -0.74 (0.07)
  Walking (n=351, 156) | -0.64 (0.05) | -0.69 (0.07)
  Hygiene (n=354, 157) | -0.64 (0.05) | -0.57 (0.08)
  Reaching (n=354, 157) | -0.77 (0.05) | -0.57 (0.08)
  Gripping (n=354, 157) | -0.68 (0.05) | -0.74 (0.08)
  Activities (n=354, 157) | -0.70 (0.05) | -0.68 (0.08)

119. Secondary Outcome: Mean BL HAQ-DI Score and HAQ-DI Individual Component Scores at BL (Day 0) of the Day 617 Cohort of Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 617
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=348, 154) | 1.69 (0.64) | 1.71 (0.59)
  Dressing and Grooming (n=348, 155) | 1.47 (0.75) | 1.50 (0.73)
  Arising (n=348, 155) | 1.42 (0.84) | 1.46 (0.79)
  Eating (n=348, 155) | 1.64 (0.97) | 1.68 (0.84)
  Walking (n=348, 154) | 1.40 (0.83) | 1.37 (0.78)
  Hygiene (n=348, 155) | 1.93 (0.90) | 1.92 (0.89)
  Reaching (n=348, 155) | 1.96 (0.86) | 1.97 (0.81)
  Gripping (n=348, 154) | 1.82 (0.75) | 1.91 (0.67)
  Activities (n=348, 155) | 1.88 (0.79) | 1.87 (0.83)

120. Secondary Outcome: Mean Change From BL in HAQ-DI Score and HAQ-DI Individual Component Scores at Day 617 for Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 617
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=348, 154) | -0.73 (0.04) | -0.74 (0.06)
  Dressing and Grooming (n=348, 155) | -0.76 (0.05) | -0.82 (0.07)
  Arising (n=348, 155) | -0.84 (0.05) | -0.81 (0.07)
  Eating (n=348, 155) | -0.80 (0.05) | -0.75 (0.07)
  Walking (n=348, 154) | -0.66 (0.05) | -0.67 (0.07)
  Hygiene (n=348, 155) | -0.56 (0.05) | -0.66 (0.08)
  Reaching (n=348, 155) | -0.81 (0.05) | -0.80 (0.08)
  Gripping (n=348, 154) | -0.75 (0.05) | -0.68 (0.08)
  Activities (n=348, 155) | -0.71 (0.05) | -0.76 (0.09)

121. Secondary Outcome: Mean BL HAQ-DI Score and HAQ-DI Individual Component Scores at BL (Day 0) of the Day 729 Cohort of Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 729
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=337, 148) | 1.69 (0.64) | 1.72 (0.60)
  Dressing and Grooming (n=337, 148) | 1.48 (0.76) | 1.51 (0.74)
  Arising (n=338, 148) | 1.41 (0.83) | 1.45 (0.79)
  Eating (n= 337, 148) | 1.63 (0.98) | 1.72 (0.83)
  Walking (n=338, 147) | 1.41 (0.84) | 1.37 (0.78)
  Hygiene (n=338, 148) | 1.93 (0.89) | 1.93 (0.89)
  Reaching (n=336, 148) | 1.95 (0.87) | 1.97 (0.81)
  Gripping (n=338, 148) | 1.81 (0.77) | 1.92 (0.65)
  Activities (n=338, 148) | 1.86 (0.79) | 1.89 (0.83)

122. Secondary Outcome: Mean Change From BL in HAQ-DI Score and HAQ-DI Individual Component Scores at Day 729 for Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 729
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=337, 148) | -0.74 (0.04) | -0.72 (0.06)
  Dressing and Grooming (n=337, 148) | -0.82 (0.05) | -0.91 (0.07)
  Arising (n=338, 148) | -0.80 (0.05) | -0.82 (0.08)
  Eating (n= 337, 148) | -0.81 (0.05) | -0.72 (0.08)
  Walking (n=338, 147) | -0.68 (0.05) | -0.63 (0.07)
  Hygiene (n=338, 148) | -0.53 (0.05) | -0.62 (0.09)
  Reaching (n=336, 148) | -0.79 (0.05) | -0.73 (0.08)
  Gripping (n=338, 148) | -0.75 (0.05) | -0.62 (0.08)
  Activities (n=338, 148) | -0.72 (0.05) | -0.72 (0.09)

123. Secondary Outcome: Mean BL HAQ-DI Score and HAQ-DI Individual Component Scores at BL (Day 0) of the Day 813 Cohort of Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 813
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=325, 146) | 1.70 (0.64) | 1.72 (0.60)
  Dressing and Grooming (n=325, 147) | 1.48 (0.75) | 1.51 (0.74)
  Arising (n=325, 147) | 1.42 (0.83) | 1.46 (0.80)
  Eating (n=325, 147) | 1.65 (0.98) | 1.70 (0.83)
  Walking (n=324, 146) | 1.42 (0.83) | 1.38 (0.78)
  Hygiene (n=325, 146) | 1.95 (0.89) | 1.94 (0.90)
  Reaching (n=324, 146) | 1.97 (0.87) | 1.97 (0.82)
  Gripping (n=325, 146) | 1.81 (0.77) | 1.92 (0.66)
  Activities (n=324, 146) | 1.87 (0.79) | 1.87 (0.84)

124. Secondary Outcome: Mean Change From BL in HAQ-DI Score and HAQ-DI Individual Component Scores at Day 813 for Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 813
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=325, 146) | -0.77 (0.04) | -0.71 (0.06)
  Dressing and Grooming (n=325, 147) | -0.82 (0.06) | -0.87 (0.07)
  Arising (n=325, 147) | -0.80 (0.05) | -0.78 (0.08)
  Eating (n=325, 147) | -0.88 (0.06) | -0.72 (0.08)
  Walking (n=324, 146) | -0.69 (0.05) | -0.66 (0.07)
  Hygiene (n=325, 146) | -0.58 (0.06) | -0.53 (0.09)
  Reaching (n=324, 146) | -0.85 (0.05) | -0.72 (0.08)
  Gripping (n=325, 146) | -0.76 (0.05) | -0.77 (0.08)
  Activities (n=324, 146) | -0.76 (0.05) | -0.71 (0.08)

125. Secondary Outcome: Mean BL HAQ-DI Score and HAQ-DI Individual Component Scores at BL (Day 0) of the Day 897 Cohort of Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 897
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=318, 140) | 1.69 (0.64) | 1.72 (0.60)
  Dressing and Grooming (n=319, 140) | 1.47 (0.76) | 1.52 (0.75)
  Arising (n=319, 140) | 1.43 (0.84) | 1.46 (0.80)
  Eating (n=319, 140) | 1.63 (0.99) | 1.71 (0.84)
  Walking (n=319, 138) | 1.41 (0.84) | 1.38 (0.79)
  Hygiene (n=319, 140) | 1.95 (0.90) | 1.94 (0.90)
  Reaching (n=319, 140) | 1.96 (0.87) | 2.01 (0.80)
  Gripping (n=319, 140) | 1.80 (0.76) | 1.92 (0.67)
  Activities (n=319, 140) | 1.87 (0.79) | 1.87 (0.85)

126. Secondary Outcome: Mean Change From BL in HAQ-DI Score and HAQ-DI Individual Component Scores at Day 897 for Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 897
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=318, 140) | -0.76 (0.04) | -0.74 (0.06)
  Dressing and Grooming (n=319, 140) | -0.86 (0.05) | -0.90 (0.08)
  Arising (n=319, 140) | -0.81 (0.05) | -0.87 (0.07)
  Eating (n=319, 140) | -0.88 (0.05) | -0.78 (0.08)
  Walking (n=319, 138) | -0.69 (0.05) | -0.67 (0.07)
  Hygiene (n=319, 140) | -0.60 (0.06) | -0.54 (0.09)
  Reaching (n=319, 140) | -0.82 (0.06) | -0.74 (0.08)
  Gripping (n=319, 140) | -0.74 (0.06) | -0.74 (0.08)
  Activities (n=319, 140) | -0.69 (0.05) | -0.71 (0.09)

127. Secondary Outcome: Mean BL HAQ-DI Score and HAQ-DI Individual Component Scores at BL (Day 0) of the Day 981 Cohort of Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 981
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=312, 137) | 1.69 (0.65) | 1.72 (0.60)
  Dressing and Grooming (n=312, 137) | 1.47 (0.76) | 1.52 (0.75)
  Arising (n=312, 137) | 1.42 (0.84) | 1.45 (0.79)
  Eating (n=312, 137) | 1.63 (0.99) | 1.70 (0.83)
  Walking (n=308, 136) | 1.41 (0.84) | 1.37 (0.79)
  Hygiene (n=312, 137) | 1.94 (0.89) | 1.93 (0.90)
  Reaching (n=312, 137) | 1.97 (0.86) | 1.99 (0.80)
  Gripping (n=312, 137) | 1.80 (0.78) | 1.92 (0.68)
  Activities (n=312, 137) | 1.87 (0.79) | 1.85 (0.84)

128. Secondary Outcome: Mean Change From BL in HAQ-DI Score and HAQ-DI Individual Component Scores at Day 981 for Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 981
Population: All treated participants in the OL period (Treatment groups represent treatment received in the DB period). Due to the non-compliance of a single site, 3 participants were not included in this analysis.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=312, 137) | -0.74 (0.04) | -0.69 (0.06)
  Dressing and Grooming (n=312, 137) | -0.80 (0.05) | -0.86 (0.08)
  Arising (n=312, 137) | -0.82 (0.05) | -0.77 (0.08)
  Eating (n=312, 137) | -0.84 (0.06) | -0.64 (0.08)
  Walking (n=308, 136) | -0.66 (0.05) | -0.63 (0.08)
  Hygiene (n=312, 137) | -0.54 (0.06) | -0.49 (0.09)
  Reaching (n=312, 137) | -0.82 (0.05) | -0.75 (0.09)
  Gripping (n=312, 137) | -0.68 (0.06) | -0.74 (0.08)
  Activities (n=312, 137) | -0.74 (0.05) | -0.64 (0.09)

129. Secondary Outcome: Mean BL HAQ-DI Score and HAQ-DI Individual Component Scores at BL (Day 0) of the Day 1,093 Cohort of Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 1,093
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=308, 137) | 1.69 (0.64) | 1.72 (0.60)
  Dressing and Grooming (n=310, 138) | 1.47 (0.75) | 1.51 (0.75)
  Arising (n=309, 138) | 1.41 (0.84) | 1.45 (0.79)
  Eating (n=309, 138) | 1.62 (0.98) | 1.69 (0.84)
  Walking (n=308, 137) | 1.41 (0.83) | 1.36 (0.78)
  Hygiene (n=310, 137) | 1.94 (0.89) | 1.92 (0.90)
  Reaching (n=310, 137) | 1.96 (0.87) | 1.99 (0.80)
  Gripping (n=310, 137) | 1.79 (0.77) | 1.92 (0.68)
  Activities (n=310, 137) | 1.87 (0.79) | 1.85 (0.84)

130. Secondary Outcome: Mean Change From BL in HAQ-DI Score and HAQ-DI Individual Component Scores at Day 1,093 for Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 1,093
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=308, 137) | -0.74 (0.04) | -0.76 (0.06)
  Dressing and Grooming (n=310, 138) | -0.80 (0.05) | -0.91 (0.07)
  Arising (n=309, 138) | -0.82 (0.05) | -0.87 (0.08)
  Eating (n=309, 138) | -0.81 (0.06) | -0.70 (0.08)
  Walking (n=308, 137) | -0.70 (0.05) | -0.69 (0.08)
  Hygiene (n=310, 137) | -0.58 (0.05) | -0.59 (0.09)
  Reaching (n=310, 137) | -0.79 (0.05) | -0.81 (0.08)
  Gripping (n=310, 137) | -0.71 (0.06) | -0.74 (0.08)
  Activities (n=310, 137) | -0.71 (0.05) | -0.73 (0.09)

131. Secondary Outcome: Mean BL HAQ-DI Score and HAQ-DI Individual Component Scores at BL (Day 0) of the Day 1,177 Cohort of Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 1,177
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=274, 125) | 1.69 (0.63) | 1.71 (0.61)
  Dressing and Grooming (n=274, 125) | 1.47 (0.76) | 1.53 (0.77)
  Arising (n=274, 125) | 1.39 (0.81) | 1.45 (0.80)
  Eating (n=274, 125) | 1.68 (0.97) | 1.70 (0.85)
  Walking (n=272, 122) | 1.37 (0.83) | 1.37 (0.78)
  Hygiene (n=275, 124) | 1.94 (0.89) | 1.90 (0.91)
  Reaching (n=275, 125) | 1.96 (0.85) | 1.99 (0.80)
  Gripping (n=275, 125) | 1.83 (0.75) | 1.91 (0.68)
  Activities (n=275, 125) | 1.87 (0.80) | 1.85 (0.86)

132. Secondary Outcome: Mean Change From BL in HAQ-DI Score and HAQ-DI Individual Component Scores at Day 1,177 for Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 1,177
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=274, 125) | -0.76 (0.04) | -0.74 (0.07)
  Dressing and Grooming (n=274, 125) | -0.82 (0.05) | -0.86 (0.09)
  Arising (n=274, 125) | -0.74 (0.06) | -0.79 (0.09)
  Eating (n=274, 125) | -0.92 (0.06) | -0.74 (0.09)
  Walking (n=272, 122) | -0.63 (0.06) | -0.66 (0.08)
  Hygiene (n=275, 124) | -0.57 (0.06) | -0.48 (0.10)
  Reaching (n=275, 125) | -0.82 (0.06) | -0.84 (0.09)
  Gripping (n=275, 125) | -0.80 (0.06) | -0.80 (0.09)
  Activities (n=275, 125) | -0.75 (0.06) | -0.76 (0.10)

133. Secondary Outcome: Mean BL HAQ-DI Score and HAQ-DI Individual Component Scores at BL (Day 0) of the Day 1,261 Cohort of Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 1,261
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=292, 134) | 1.69 (0.65) | 1.70 (0.60)
  Dressing and Grooming (n=292, 135) | 1.47 (0.77) | 1.51 (0.75)
  Arising (n=292, 135) | 1.42 (0.85) | 1.44 (0.79)
  Eating (n=292, 135) | 1.64 (1.00) | 1.69 (0.83)
  Walking (n=290, 134) | 1.40 (0.83) | 1.36 (0.79)
  Hygiene (n=292, 134) | 1.96 (0.90) | 1.92 (0.90)
  Reaching (n=292, 134) | 1.97 (0.87) | 1.97 (0.79)
  Gripping (n=292, 134) | 1.79 (0.77) | 1.91 (0.68)
  Activities (n=292, 133) | 1.87 (0.81) | 1.83 (0.85)

134. Secondary Outcome: Mean Change From BL in HAQ-DI Score and HAQ-DI Individual Component Scores at Day 1,261 for Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 1,261
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=292, 134) | -0.74 (0.04) | -0.73 (0.06)
  Dressing and Grooming (n=292, 135) | -0.81 (0.05) | -0.91 (0.08)
  Arising (n=292, 135) | -0.82 (0.05) | -0.82 (0.08)
  Eating (n=292, 135) | -0.85 (0.06) | -0.73 (0.08)
  Walking (n=290, 134) | -0.66 (0.06) | -0.63 (0.08)
  Hygiene (n=292, 134) | -0.52 (0.06) | -0.54 (0.09)
  Reaching (n=292, 134) | -0.83 (0.06) | -0.80 (0.09)
  Gripping (n=292, 134) | -0.68 (0.06) | -0.70 (0.09)
  Activities (n=292, 133) | -0.75 (0.05) | -0.68 (0.10)

135. Secondary Outcome: Mean BL HAQ-DI Score and HAQ-DI Individual Component Scores at BL (Day 0) of the Day 1,345 Cohort of Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 1,345
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=152, 62) | 1.65 (0.63) | 1.73 (0.58)
  Dressing and Grooming (n=152, 62) | 1.45 (0.73) | 1.50 (0.70)
  Arising (n=152, 62) | 1.34 (0.79) | 1.44 (0.74)
  Eating (n=152, 62) | 1.63 (0.97) | 1.69 (0.84)
  Walking (n=151, 62) | 1.32 (0.80) | 1.35 (0.79)
  Hygiene (n=152, 62) | 1.82 (0.89) | 2.05 (0.86)
  Reaching (n=152, 62) | 1.98 (0.82) | 2.06 (0.74)
  Gripping (n=152, 62) | 1.77 (0.74) | 1.94 (0.60)
  Activities (n=152, 62) | 1.88 (0.79) | 1.79 (0.77)

136. Secondary Outcome: Mean Change From BL in HAQ-DI Score and HAQ-DI Individual Component Scores at Day 1,345 for Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 1,345
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=152, 62) | -0.69 (0.06) | -0.73 (0.09)
  Dressing and Grooming (n=152, 62) | -0.74 (0.07) | -0.81 (0.11)
  Arising (n=152, 62) | -0.68 (0.08) | -0.84 (0.12)
  Eating (n=152, 62) | -0.84 (0.08) | -0.68 (0.13)
  Walking (n=151, 62) | -0.61 (0.07) | -0.60 (0.13)
  Hygiene (n=152, 62) | -0.46 (0.09) | -0.71 (0.13)
  Reaching (n=152, 62) | -0.84 (0.08) | -0.76 (0.13)
  Gripping (n=152, 62) | -0.63 (0.08) | -0.82 (0.11)
  Activities (n=152, 62) | -0.73 (0.08) | -0.60 (0.12)

137. Secondary Outcome: Mean BL HAQ-DI Score and HAQ-DI Individual Component Scores at BL (Day 0) of the Day 1,457 Cohort of Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 1,457
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=289, 129) | 1.70 (0.65) | 1.71 (0.60)
  Dressing and Grooming (n=289, 129) | 1.48 (0.76) | 1.51 (0.74)
  Arising (n=289, 129) | 1.43 (0.85) | 1.44 (0.78)
  Eating (n=289, 129) | 1.64 (1.00) | 1.70 (0.83)
  Walking (n=287, 126) | 1.42 (0.83) | 1.37 (0.78)
  Hygiene (n=289, 129) | 1.95 (0.89) | 1.91 (0.91)
  Reaching (n=289, 129) | 1.97 (0.86) | 1.99 (0.79)
  Gripping (n=289, 129) | 1.80 (0.77) | 1.91 (0.69)
  Activities (n=289, 129) | 1.88 (0.80) | 1.84 (0.84)

138. Secondary Outcome: Mean Change From BL in HAQ-DI Score and HAQ-DI Individual Component Scores at Day 1,457 for Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 1,457
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=289, 129) | -0.77 (0.04) | -0.74 (0.06)
  Dressing and Grooming (n=289, 129) | -0.85 (0.06) | -0.91 (0.08)
  Arising (n=289, 129) | -0.80 (0.05) | -0.82 (0.08)
  Eating (n=289, 129) | -0.89 (0.06) | -0.81 (0.08)
  Walking (n=287, 126) | -0.68 (0.05) | -0.63 (0.08)
  Hygiene (n=289, 129) | -0.57 (0.06) | -0.59 (0.10)
  Reaching (n=289, 129) | -0.84 (0.06) | -0.76 (0.09)
  Gripping (n=289, 129) | -0.77 (0.06) | -0.71 (0.09)
  Activities (n=289, 129) | -0.77 (0.06) | -0.74 (0.09)

139. Secondary Outcome: Mean BL HAQ-DI Score and HAQ-DI Individual Component Scores at BL (Day 0) of the Day 1,625 Cohort of Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 1,625
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=280, 126) | 1.69 (0.65) | 1.72 (0.59)
  Dressing and Grooming (n=280, 126) | 1.46 (0.77) | 1.52 (0.73)
  Arising (n=280, 126) | 1.42 (0.85) | 1.45 (0.75)
  Eating (n=280, 126) | 1.63 (0.99) | 1.69 (0.83)
  Walking (n=279, 125) | 1.43 (0.84) | 1.37 (0.78)
  Hygiene (n=280, 126) | 1.94 (0.90) | 1.93 (0.89)
  Reaching (n=280, 126) | 1.96 (0.85) | 2.00 (0.78)
  Gripping (n=280, 126) | 1.80 (0.77) | 1.93 (0.67)
  Activities (n=280, 126) | 1.88 (0.80) | 1.87 (0.83)

140. Secondary Outcome: Mean Change From BL in HAQ-DI Score and HAQ-DI Individual Component Scores at Day 1,625 for Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 1,625
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=280, 126) | -0.76 (0.04) | -0.78 (0.06)
  Dressing and Grooming (n=280, 126) | -0.84 (0.06) | -0.98 (0.08)
  Arising (n=280, 126) | -0.79 (0.06) | -0.84 (0.08)
  Eating (n=280, 126) | -0.83 (0.06) | -0.79 (0.09)
  Walking (n=279, 125) | -0.70 (0.06) | -0.74 (0.08)
  Hygiene (n=280, 126) | -0.56 (0.06) | -0.57 (0.10)
  Reaching (n=280, 126) | -0.83 (0.06) | -0.81 (0.09)
  Gripping (n=280, 126) | -0.80 (0.06) | -0.76 (0.09)
  Activities (n=280, 126) | -0.78 (0.06) | -0.76 (0.09)

141. Secondary Outcome: Mean BL HAQ-DI Score and HAQ-DI Individual Component Scores at BL (Day 0) of the Day 1,821 Cohort of Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 1,821
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=273, 125) | 1.69 (0.65) | 1.69 (0.60)
  Dressing and Grooming (n=273, 125) | 1.47 (0.77) | 1.49 (0.74)
  Arising (n=273, 125) | 1.41 (0.83) | 1.42 (0.76)
  Eating (n=273, 124) | 1.63 (1.00) | 1.67 (0.83)
  Walking (n=271, 122) | 1.43 (0.84) | 1.34 (0.78)
  Hygiene (n=273, 125) | 1.93 (0.90) | 1.88 (0.91)
  Reaching (n=273, 125) | 1.97 (0.86) | 1.97 (0.78)
  Gripping (n=273, 125) | 1.79 (0.78) | 1.90 (0.70)
  Activities (n=273, 125) | 1.88 (0.81) | 1.82 (0.85)

142. Secondary Outcome: Mean Change From BL in HAQ-DI Score and HAQ-DI Individual Component Scores at Day 1,821 for Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 1,821
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=273, 125) | -0.77 (0.44) | -0.72 (0.06)
  Dressing and Grooming (n=273, 125) | -0.82 (0.06) | -0.86 (0.08)
  Arising (n=273, 125) | -0.83 (0.06) | -0.90 (0.08)
  Eating (n=273, 124) | -0.86 (0.07) | -0.78 (0.09)
  Walking (n=271, 122) | -0.68 (0.06) | -0.61 (0.08)
  Hygiene (n=273, 125) | -0.56 (0.07) | -0.53 (0.10)
  Reaching (n=273, 125) | -0.83 (0.06) | -0.74 (0.09)
  Gripping (n=273, 125) | -0.79 (0.06) | -0.80 (0.09)
  Activities (n=273, 125) | -0.76 (0.06) | -0.61 (0.09)

143. Secondary Outcome: Mean BL HAQ-DI Score and HAQ-DI Individual Component Scores at BL (Day 0) of the Day 1,989 Cohort of Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 1,989
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=119, 55) | 1.72 (0.61) | 1.67 (0.62)
  Dressing and Grooming (n=119, 55) | 1.51 (0.72) | 1.49 (0.69)
  Arising (n=119, 55) | 1.36 (0.78) | 1.38 (0.78)
  Eating (n=119, 55) | 1.66 (0.99) | 1.62 (0.85)
  Walking (n=117, 54) | 1.45 (0.79) | 1.30 (0.84)
  Hygiene (n=119, 55) | 1.87 (0.94) | 1.89 (0.92)
  Reaching (n=119, 55) | 2.08 (0.81) | 1.98 (0.76)
  Gripping (n=119, 55) | 1.85 (0.74) | 1.87 (0.67)
  Activities (n=119, 55) | 1.97 (0.81) | 1.84 (0.74)

144. Secondary Outcome: Mean Change From BL in HAQ-DI Score and HAQ-DI Individual Component Scores at Day 1,989 for Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 1,989
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=119, 55) | -0.81 (0.07) | -0.70 (0.10)
  Dressing and Grooming (n=119, 55) | -0.84 (0.09) | -0.76 (0.11)
  Arising (n=119, 55) | -0.86 (0.08) | -0.84 (0.12)
  Eating (n=119, 55) | -0.83 (0.10) | -0.62 (0.14)
  Walking (n=117, 54) | -0.77 (0.09) | -0.67 (0.12)
  Hygiene (n=119, 55) | -0.56 (0.11) | -0.58 (0.13)
  Reaching (n=119, 55) | -0.89 (0.10) | -0.75 (0.14)
  Gripping (n=119, 55) | -0.88 (0.10) | -0.67 (0.12)
  Activities (n=119, 55) | -0.84 (0.10) | -0.71 (0.13)

145. Secondary Outcome: Mean BL HAQ-DI Score and HAQ-DI Individual Component Scores at BL (Day 0) of the Day 2,185 Cohort of Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 2,185
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=85, 38) | 1.73 (0.55) | 1.69 (0.49)
  Dressing and Grooming (n=85, 37) | 1.54 (0.70) | 1.54 (0.65)
  Arising (n=85, 38) | 1.36 (0.72) | 1.37 (0.59)
  Eating (n=85, 38) | 1.64 (0.96) | 1.58 (0.79)
  Walking (n=84, 38) | 1.39 (0.73) | 1.37 (0.71)
  Hygiene (n=85, 38) | 1.86 (0.91) | 1.97 (0.82)
  Reaching (n=85, 38) | 2.11 (0.79) | 2.03 (0.68)
  Gripping (n=85, 38) | 1.86 (0.73) | 1.84 (0.55)
  Activities (n=85, 38) | 2.04 (0.70) | 1.84 (0.59)

146. Secondary Outcome: Mean Change From BL in HAQ-DI Score and HAQ-DI Individual Component Scores at Day 2,185 for Participants Continuing in the OL Period
Description: as for outcome 2
Time Frame: BL (Day 0), Day 2,185
Population: as for outcome 53
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | ABA + MTX DB | MTX + Placebo DB
Number analyzed (Participants) | 376 | 160
Units on a Scale
  HAQ DI (n=85, 38) | -0.70 (0.08) | -0.68 (0.10)
  Dressing and Grooming (n=85, 37) | -0.68 (0.10) | -0.78 (0.13)
  Arising (n=85, 38) | -0.66 (0.11) | -0.82 (0.12)
  Eating (n=85, 38) | -0.82 (0.11) | -0.74 (0.16)
  Walking (n=84, 38) | -0.67 (0.11) | -0.58 (0.14)
  Hygiene (n=85, 38) | -0.55 (0.13) | -0.68 (0.15)
  Reaching (n=85, 38) | -0.88 (0.12) | -0.66 (0.17)
  Gripping (n=85, 38) | -0.64 (0.11) | -0.47 (0.12)
  Activities (n=85, 38) | -0.68 (0.10) | -0.68 (0.13)

ADVERSE EVENTS:
Arm/Group | ABA + MTX OL | ABA + MTX DB | MTX + Placebo DB
Serious Adverse Events (participants affected / at risk) | 215/539 | 68/433 | 27/219
Other Adverse Events (participants affected / at risk) | 466/539 | 320/433 | 144/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABA + MTX OL (N=539) | ABA + MTX DB (N=433) | MTX + Placebo DB (N=219)
CATARACT (Eye disorders) | 3 | 0 | 1
STRABISMUS (Eye disorders) | 1 | 0 | 0
VITREOUS DETACHMENT (Eye disorders) | 1 | 0 | 0
ARTERIOGRAM (Investigations) | 1 | 0 | 0
WEIGHT DECREASED (Investigations) | 1 | 0 | 0
LABORATORY TEST ABNORMAL (Investigations) | 1 | 0 | 0
ELECTROCARDIOGRAM ST SEGMENT ABNORMAL (Investigations) | 1 | 0 | 0
ARRHYTHMIA (Cardiac disorders) | 1 | 0 | 0
BRADYCARDIA (Cardiac disorders) | 1 | 0 | 0
CARDIAC ARREST (Cardiac disorders) | 3 | 0 | 0
ANGINA UNSTABLE (Cardiac disorders) | 2 | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 1 | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 1 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 1
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 2 | 0 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 4 | 1 | 0
TACHYCARDIA PAROXYSMAL (Cardiac disorders) | 0 | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 2 | 1 | 0
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1 | 0 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 | 0 | 0
HYPERTENSION (Vascular disorders) | 1 | 0 | 0
VARICOSE VEIN (Vascular disorders) | 1 | 0 | 0
AORTIC ANEURYSM (Vascular disorders) | 1 | 0 | 0
THROMBOPHLEBITIS (Vascular disorders) | 1 | 0 | 0
ARTERIAL DISORDER (Vascular disorders) | 0 | 0 | 1
VENOUS THROMBOSIS (Vascular disorders) | 1 | 0 | 0
HYPOVOLAEMIC SHOCK (Vascular disorders) | 1 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 0
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 | 1 | 0
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 1 | 0 | 0
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 0 | 1 | 0
DELIRIUM (Psychiatric disorders) | 1 | 0 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 6 | 1 | 0
BILE DUCT STONE (Hepatobiliary disorders) | 3 | 0 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0 | 0
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 2 | 0 | 0
APHASIA (Nervous system disorders) | 1 | 0 | 0
SYNCOPE (Nervous system disorders) | 1 | 0 | 0
MIGRAINE (Nervous system disorders) | 1 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 0 | 1
HYPOAESTHESIA (Nervous system disorders) | 1 | 0 | 0
OPTIC NEURITIS (Nervous system disorders) | 1 | 0 | 0
POLYNEUROPATHY (Nervous system disorders) | 2 | 0 | 0
TENSION HEADACHE (Nervous system disorders) | 1 | 0 | 0
NERVE COMPRESSION (Nervous system disorders) | 1 | 0 | 0
CEREBRAL INFARCTION (Nervous system disorders) | 0 | 0 | 1
CERVICAL MYELOPATHY (Nervous system disorders) | 1 | 0 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1 | 1
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 | 1 | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 4 | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 2 | 1 | 0
COMPLEX REGIONAL PAIN SYNDROME (Nervous system disorders) | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 0 | 1
PERITONITIS (Gastrointestinal disorders) | 1 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 0 | 1
OESOPHAGITIS (Gastrointestinal disorders) | 1 | 0 | 0
PEPTIC ULCER (Gastrointestinal disorders) | 1 | 0 | 0
RECTAL POLYP (Gastrointestinal disorders) | 1 | 0 | 0
ENTEROCOLITIS (Gastrointestinal disorders) | 1 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 0 | 1
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1 | 0 | 0
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0
GASTRODUODENITIS (Gastrointestinal disorders) | 1 | 0 | 0
UMBILICAL HERNIA (Gastrointestinal disorders) | 3 | 2 | 0
COLITIS ULCERATIVE (Gastrointestinal disorders) | 2 | 0 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0 | 0
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0
ABDOMINAL HERNIA OBSTRUCTIVE (Gastrointestinal disorders) | 1 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 | 0 | 0
ABDOMINAL STRANGULATED HERNIA (Gastrointestinal disorders) | 1 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0 | 0
MESENTERIC VASCULAR INSUFFICIENCY (Gastrointestinal disorders) | 1 | 0 | 0
SEPSIS (Infections and infestations) | 1 | 1 | 1
ABSCESS (Infections and infestations) | 0 | 1 | 0
CYSTITIS (Infections and infestations) | 1 | 0 | 0
RHINITIS (Infections and infestations) | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 7 | 4 | 1
SINUSITIS (Infections and infestations) | 2 | 0 | 0
BRONCHITIS (Infections and infestations) | 4 | 0 | 0
CELLULITIS (Infections and infestations) | 5 | 1 | 1
ERYSIPELAS (Infections and infestations) | 2 | 0 | 0
PARONYCHIA (Infections and infestations) | 0 | 1 | 0
ABSCESS JAW (Infections and infestations) | 1 | 0 | 0
BACTERAEMIA (Infections and infestations) | 1 | 0 | 0
PHARYNGITIS (Infections and infestations) | 1 | 0 | 0
ABSCESS LIMB (Infections and infestations) | 1 | 0 | 1
APPENDICITIS (Infections and infestations) | 1 | 0 | 1
SEPTIC SHOCK (Infections and infestations) | 2 | 0 | 0
TUBERCULOSIS (Infections and infestations) | 0 | 1 | 0
DACRYOCYSTITIS (Infections and infestations) | 1 | 0 | 0
DIVERTICULITIS (Infections and infestations) | 1 | 2 | 0
LUNG INFECTION (Infections and infestations) | 1 | 0 | 0
PYELONEPHRITIS (Infections and infestations) | 2 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 2 | 1 | 0
LOBAR PNEUMONIA (Infections and infestations) | 2 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 1 | 0 | 0
WOUND INFECTION (Infections and infestations) | 1 | 0 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 2 | 0
DOUGLAS' ABSCESS (Infections and infestations) | 0 | 0 | 1
HERPES DERMATITIS (Infections and infestations) | 1 | 0 | 0
ESCHERICHIA SEPSIS (Infections and infestations) | 1 | 0 | 0
PERIRECTAL ABSCESS (Infections and infestations) | 1 | 0 | 0
ARTHRITIS BACTERIAL (Infections and infestations) | 1 | 1 | 0
LOCALISED INFECTION (Infections and infestations) | 1 | 0 | 0
OSTEOMYELITIS ACUTE (Infections and infestations) | 1 | 0 | 0
PERINEPHRIC ABSCESS (Infections and infestations) | 1 | 0 | 0
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 | 1 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 2 | 0 | 0
TUBERCULOUS PLEURISY (Infections and infestations) | 1 | 0 | 0
SOFT TISSUE INFECTION (Infections and infestations) | 1 | 0 | 0
ABDOMINAL WALL ABSCESS (Infections and infestations) | 1 | 0 | 0
ENDOCARDITIS BACTERIAL (Infections and infestations) | 1 | 0 | 0
HERPES VIRUS INFECTION (Infections and infestations) | 1 | 0 | 0
PULMONARY TUBERCULOSIS (Infections and infestations) | 2 | 0 | 0
INCISION SITE INFECTION (Infections and infestations) | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 5 | 2 | 0
POST PROCEDURAL INFECTION (Infections and infestations) | 1 | 0 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 | 0 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 2 | 0 | 0
STAPHYLOCOCCAL SKIN INFECTION (Infections and infestations) | 1 | 0 | 0
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
RENAL COLIC (Renal and urinary disorders) | 1 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 2 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 2 | 1 | 0
CALCULUS BLADDER (Renal and urinary disorders) | 1 | 0 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 0 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 1 | 0 | 0
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 1 | 0 | 0
OBESITY (Metabolism and nutrition disorders) | 2 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 2 | 2 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 4 | 1 | 0
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 | 1 | 0
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
DERMATOMYOSITIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
CYSTOCELE (Reproductive system and breast disorders) | 1 | 0 | 0
RECTOCELE (Reproductive system and breast disorders) | 1 | 0 | 0
METRORRHAGIA (Reproductive system and breast disorders) | 1 | 0 | 0
OVARIAN CYST (Reproductive system and breast disorders) | 0 | 1 | 0
ENDOMETRIOSIS (Reproductive system and breast disorders) | 1 | 0 | 0
UTERINE POLYP (Reproductive system and breast disorders) | 1 | 0 | 0
UTERINE PROLAPSE (Reproductive system and breast disorders) | 1 | 0 | 0
BREAST CALCIFICATIONS (Reproductive system and breast disorders) | 0 | 1 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 3 | 0 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0 | 0
EYE INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 3 | 0 | 0
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
ULNA FRACTURE (Injury, poisoning and procedural complications) | 2 | 0 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
GUN SHOT WOUND (Injury, poisoning and procedural complications) | 1 | 0 | 0
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
MENISCUS LESION (Injury, poisoning and procedural complications) | 0 | 1 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 | 0 | 0
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 | 0 | 0
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 | 0 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 4 | 0 | 0
FAILURE OF IMPLANT (Injury, poisoning and procedural complications) | 0 | 1 | 0
TRAUMATIC FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 2 | 0 | 0
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
PROCEDURAL VOMITING (Injury, poisoning and procedural complications) | 0 | 1 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 0 | 2 | 0
INCORRECT DOSE ADMINISTERED (Injury, poisoning and procedural complications) | 1 | 0 | 0
MEDICAL DEVICE COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0 | 0
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 2 | 0 | 0
DISLOCATION OF JOINT PROSTHESIS (Injury, poisoning and procedural complications) | 2 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 7 | 3 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
BONE CYST (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
MONARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
METATARSALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 20 | 2 | 2
RHEUMATOID NODULE (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
MUSCLE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 36 | 13 | 6
SOFT TISSUE NECROSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
TONSILLAR INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
PYREXIA (General disorders) | 2 | 0 | 0
CHEST PAIN (General disorders) | 5 | 1 | 0
IMPAIRED HEALING (General disorders) | 3 | 1 | 0
HERNIA OBSTRUCTIVE (General disorders) | 1 | 0 | 0
MULTI-ORGAN FAILURE (General disorders) | 0 | 0 | 1
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
CARDIAC MYXOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 4 | 1
BENIGN BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
FIBROADENOMA OF BREAST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
NEUROENDOCRINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
GASTROINTESTINAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
MALIGNANT MELANOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
ACUTE LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
BRONCHIOLOALVEOLAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
LYMPHOPROLIFERATIVE DISORDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 1
EXTRANODAL MARGINAL ZONE B-CELL LYMPHOMA (MALT TYPE) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABA + MTX OL (N=539) | ABA + MTX DB (N=433) | MTX + Placebo DB (N=219)
CONJUNCTIVITIS (Eye disorders) | 37 | 4 | 2
HYPERTENSION (Vascular disorders) | 86 | 26 | 4
ANXIETY (Psychiatric disorders) | 27 | 15 | 6
INSOMNIA (Psychiatric disorders) | 51 | 12 | 6
DEPRESSION (Psychiatric disorders) | 41 | 15 | 7
HEADACHE (Nervous system disorders) | 99 | 77 | 26
DIZZINESS (Nervous system disorders) | 54 | 41 | 16
NAUSEA (Gastrointestinal disorders) | 53 | 53 | 25
VOMITING (Gastrointestinal disorders) | 30 | 17 | 8
DIARRHOEA (Gastrointestinal disorders) | 83 | 48 | 22
DYSPEPSIA (Gastrointestinal disorders) | 72 | 28 | 10
GASTRITIS (Gastrointestinal disorders) | 29 | 9 | 6
ABDOMINAL PAIN (Gastrointestinal disorders) | 33 | 12 | 7
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 50 | 19 | 13
RHINITIS (Infections and infestations) | 42 | 15 | 7
INFLUENZA (Infections and infestations) | 76 | 30 | 12
SINUSITIS (Infections and infestations) | 64 | 19 | 15
BRONCHITIS (Infections and infestations) | 95 | 37 | 16
PHARYNGITIS (Infections and infestations) | 70 | 27 | 10
GASTROENTERITIS (Infections and infestations) | 42 | 10 | 9
NASOPHARYNGITIS (Infections and infestations) | 137 | 66 | 25
URINARY TRACT INFECTION (Infections and infestations) | 118 | 21 | 11
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 131 | 47 | 21
ANAEMIA (Blood and lymphatic system disorders) | 35 | 9 | 8
RASH (Skin and subcutaneous tissue disorders) | 30 | 19 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 110 | 40 | 13
TENDONITIS (Musculoskeletal and connective tissue disorders) | 29 | 1 | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 83 | 31 | 15
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 29 | 3 | 4
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 31 | 11 | 7
FATIGUE (General disorders) | 32 | 24 | 15
CHEST PAIN (General disorders) | 38 | 7 | 5
OEDEMA PERIPHERAL (General disorders) | 38 | 13 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.